# CLINICAL STUDY PROTOCOL

A Phase 1, Partially-Blinded, Placebo-Controlled, Randomized Single Ascending Dose (SAD) with a Food Effect Cohort Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBI-223 in Healthy Adult Participants

PROTOCOL NUMBER

TBI-223-CL-001

Version: 3.0

21 Jan 2020

#### **CONFIDENTIALITY STATEMENT**

The confidential information in this document is provided to you as an Investigator or consultant for review by you, your staff, and the applicable Institutional Review Board/Independent Ethics Committee. Your acceptance of this document constitutes agreement that you will not disclose the information herein to others without written authorization from Worldwide Clinical Trials Early Phase Services, LLC, except to the extent necessary to obtain informed consent from persons who participate as subjects in this study.

# PROTOCOL APPROVAL PAGE

A Phase 1, Partially-Blinded, Placebo-Controlled, Randomized, Single Ascending Dose (SAD)with a Food Effect Cohort Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBI-223 in Healthy Adult Participants

Protocol Number: TBI-223-CL-001

Sponsor: Global Alliance for TB Drug Development

Sponsor Contact and

Medical Monitor: Paul Bruinenberg MD, MBA

Global Alliance for TB Drug Development

40 Wall Street, 24th Floor

New York, NY 10005, United States of America

Telephone: +1 646 616 8629 Mobile: +1-201-312-0988 Facsimile: +1 212 227 7541

Email: Paul.Bruinenberg@tballiance.org

DocuSigned by:

full Environment
Signing Reason: I approve his document
Signing Time: 21-Jan-2020 | 10:51:10 EST
38496C383A5A4B0AAE3273125587116B

21-Jan-2020 | 10:51:14 EST

(Signature)

Principal Investigator: Cynthia A. Zamora, MD

Worldwide Clinical Trials Early Phase Services, LLC

(Date)

2455 N.E. Loop 410, Suite 150 San Antonio, Texas 78217 Telephone: 210.635.1500

Fax: 210.635.1646

DocuSigned by:

Upulluia Lanera

Signer Name: Cynthia Zamora
Signing Reason: Lapprove this document
Signing Time: 2-1-Jan-2020 | 16:11:56 GMT
FA8D8484FD8647B3A4A33071357CA7F7

21-Jan-2020 | 16:12:01 GMT

(Signature) (Date)

# **SUMMARY OF CHANGES**

The primary reasons for this amendment are to incorporate the changes from the protocol clarification letter dated 18 Oct 2019 regarding subject replacement of subjects who experience emesis, how replacement subjects will be numbered, and that replacement subjects will receive the same dose allocation of study drug.

This amendment also includes clarifying Part 1 and Part 2 and updates whereby Part 1 captures adding a capsule cohort (3b, TBI-223, 300 mg), updating the dose of cohort 7 (TBI-223, 2600 mg) and whereby Part 2 consists of 2 additional cohorts (Cohort 8 and 9) that will be added to the study in relation to evaluating tablet formulations of TBI-223.

Part 1: (TBI-223 oral suspension)

Cohort 3b: Is a cohort that was added to evaluate a capsule formulation of TBI-223 150 mg in oral enteric capsules, dosed at 300 mg

Cohort 7: Is the final TBI-223 oral suspension cohort at a dose of 2600 mg

Part 2: (TBI-223 tablet formulation)

**Cohort 8:** Is a single dose cohort that investigates 3 different TBI-223 Sustained Release (SR) tablet formulations (Prototypes 1, 2, and 3) and one TBI-223 Immediate Release (IR) tablet formulation. The cohort includes 4 arms with 6 subjects per arm. The 3 SR tablet formulations (Prototypes 1, 2, and 3) will be evaluated under fed conditions (Arms 1-3) and the IR tablet formulation will be evaluated under fasting conditions (Arm 4).

**Cohort 9:** 6 subjects from Cohort 8, Arm 4, who received the IR tablet formulation will be brought back following a 7-day washout and receive the IR tablet formulation under fed conditions. If more than 2 subjects of these 6 subjects from Cohort 8 drop-out, they will be replaced by healthy volunteers (a minimum of 4 subjects are needed to complete Cohort 9).

Additional minor changes to format, grammar, and spelling have been applied.

The sections of protocol version 2.0 dated 12 Jul 2019 affected by these changes are indicated below.

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) |
|---|---|---|
| Synopsis | Study period<br>(maximum<br>duration, from<br>screening to<br>study exit): | From: Single ascending dose (SAD) cohort (fasting): 40 days Food-effect cohort: 50 days The maximum duration of the study will depend upon the final number and timing of each cohort. |

| Section | | |
|---|---|---|
| Number (s) | Section Title(s) | Description of Change (s) |
| | | To: |
| | | Part 1: |
| | | Single ascending dose (SAD) cohort (fasting): 40 days |
| | | Food-effect cohort: 50 days |
| | | Part 2: |
| | | Cohort 8: Single dose cohort of the 4 TBI-223 tablet formulations (Prototypes 1, 2, and 3 SR tablet formulations under fed conditions and one IR tablet formulation under fasting conditions): Duration 40 days. |
| | | Cohort 9: The IR tablet formulation will be evaluated under fed conditions |
| | | Single dose: 40 days |
| | | The maximum duration of the study will depend upon the final number and timing of each cohort. |
| Synopsis | Duration of treatment | From: |
| | | <u>Fasting cohorts</u> : One single dose of TBI-223 oral suspension or placebo for TBI-223 oral suspension |
| | | Food-effect cohort: Two single doses of TBI-223 oral suspension or placebo for TBI-223 oral suspension separated by a washout period of at least 7 days |
| | | To: |
| | | Part 1: |
| | | <u>Fasting cohorts</u> : One single dose of TBI-223 oral suspension or placebo for TBI-223 oral suspension |
| | | Food-effect cohort: Two single doses of TBI-223 oral suspension or placebo for TBI-223 oral suspension separated by a washout period of at least 7 days |
| | | Part 2: |
| | | Cohort 8: Single dose cohort of 4 TBI-223 tablet formulations (three SR tablet formulations as prototypes 1, 2, and3 and one IR tablet formulation). The SR tablet formulations will be evaluated under fed conditions and the IR tablet formulation will be evaluated under fasting conditions |
| | | Cohort 9: The IR tablet formulation will be evaluated under fed conditions |
| Synopsis | Number of | From: |
| | subjects<br>(planned) | Fasting Cohorts: Planned to enroll up to 48 subjects in a total of 6 single ascending dose (SAD) cohorts of 8 subjects each (6 to receive active drug |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) |
|---|---|---|
| (5) | Section Title(s) | and 2 to receive placebo). |
| | | Food-effect Cohort: 1 cohort with 10 subjects (8 active and 2 placebo) who will receive TBI-223 or placebo under both fasting and fed conditions. |
| | | Additional cohorts may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level. These decisions on additional cohorts will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort have been demonstrated to permit proceeding to the next cohort. The Institutional Review Board (IRB) should be immediately notified of this revised approach. |
| | | To: |
| | | Part 1: |
| | | <u>Fasting Cohorts</u> : Planned to enroll up to 48 subjects in a total of 6 single ascending dose (SAD) cohorts of 8 subjects each (6 to receive active drug and 2 to receive placebo). |
| | | Food-effect Cohort: 1 cohort with 10 subjects (8 active and 2 placebo) who will receive TBI-223 or placebo under both fasting and fed conditions. |
| | | Part 2: |
| | | Cohort 8: Planned to enroll 24 subjects in a total of 4 arms with 6 subjects in each. Subjects will receive a single dose of 1 of the 3 prototypes of TBI-223 SR tablets under fed conditions (Arms 1-3) or a single dose of TBI-223 IR tablets under fasted conditions (Arm 4). |
| | | Cohort 9: Plan to bring back the 6 subjects from Cohort 8, Arm 4, who received the IR tablet formulation, following a 7-day washout to receive the IR tablet formulation under fed conditions. |
| | | If more than 2 subjects of these 6 subjects from Cohort 8 drop-out, they will be replaced by heathy volunteers (a minimum of 4 subjects are needed to complete Cohort 9). |
| | | Additional cohorts may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level. These decisions on additional cohorts will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort have been demonstrated to permit proceeding to the next cohort. The Institutional Review Board (IRB) should be immediately notified of this revised approach. |
| Synopsis | Objective | From: |
| and 2 | | The primary objective of the study is: |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) |
|---|---|---|
| | | • To evaluate the safety and tolerability of single ascending doses of TBI-<br>223 oral suspension in healthy adult subjects. |
| | | The secondary objectives of the study are: |
| | | • To determine the pharmacokinetics of TBI-223 and its metabolite M2 after single doses of TBI 223 oral suspension in healthy adult subjects; and |
| | | • To compare the rate and extent of absorption of a single dose of TBI-223 oral suspension when administered in healthy adult subjects either after a high-calorie, high-fat meal or in the fasting state. |
| | | To: |
| | | The primary objective of the study is: |
| | | • To evaluate the safety and tolerability of single ascending doses of TBI-223 oral suspension, TBI-223 oral enteric capsules, and TBI-223 tablet formulations in healthy adult subjects. |
| | | The secondary objectives of the study are: |
| | | <ul> <li>To determine the pharmacokinetics of TBI-223 and its metabolite M2 after single doses of TBI-223 oral suspension, TBI-223 oral enteric capsules, and TBI-223 tablet formulations in healthy adult subjects; and</li> </ul> |
| | | • To compare the rate and extent of absorption of a single dose of TBI-223 oral suspension, TBI-223 oral enteric capsules, and TBI-223 tablet formulations when administered in healthy adult subjects either after a high-calorie, high-fat meal or in the fasting state. |
| Synopsis | Section before | From: |
| | Test product,<br>dosage and<br>mode of | This is a partially-blinded, placebo-controlled, randomized SAD study with a food effect cohort. The study will be conducted at one study center in the United States. |
| | administration | This study will have up to 6 planned dose levels. Based on interim pharmacokinetic data obtained during the dose escalation, a dose cohort will be selected to return for additional dosing after a high-calorie, high-fat meal (food-effect cohort). |
| | | Sentinel Cohort: The first cohort will be separated into 2 groups. A sentinel group of 3 subjects (2 active and 1 placebo) will be dosed at least 24 hours before the remaining 5 subjects (4 active and 1 placebo). The remaining cohorts will be dosed in 2 groups of 4 subjects each (3 active and 1 placebo), at least 24 hours apart. |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) |
|---|---|---|
| | | Food-effect Cohort: Based on exposure levels, subjects in one of the dose levels will return after a 7-day minimum washout or 5 half-lives of the drug (whichever is longer) to receive the same dose under fed conditions. |
| | | Safety will be assessed throughout the study for all subjects. |
| | | Blood will be collected for pharmacokinetic analysis. Plasma samples will be analyzed for TBI-223 and TBI-223 metabolite (M2). |
| | | Dose escalation to the next cohort (i.e., dose level) will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort has been demonstrated to permit proceeding to the next cohort. |
| | | Additional cohorts may be enrolled if deemed appropriate (e.g. if bioavailability is lower than expected) by the Sponsor to repeat a dose level, to study other dose levels, change proposed cohorts, or to study a different dosage formulation. These decisions regarding changed or additional cohorts will not take place until the Sponsor, in conjunction with the Principal Investigator and dose escalating committee, has determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort have been demonstrated to permit proceeding to the next cohort. The Institutional Review Board (IRB) should be immediately notified of this revised approach for review and approval. |
| | | To: |
| | | This is a partially-blinded, placebo-controlled, randomized SAD study with a food effect cohort. The study will be conducted at one study center in the United States. |
| | | Safety will be assessed throughout the study for all subjects. |
| | | Blood will be collected for pharmacokinetic analysis. Plasma samples will be analyzed for TBI-223 and TBI-223 metabolite (M2). |
| | | Part 1: |
| | | There will be up to 6 planned dose levels. Based on interim pharmacokinetic data obtained during the dose escalation, a dose cohort will be selected to return for additional dosing after a high-calorie, high-fat meal (food-effect cohort). |
| | | Sentinel Cohort: The first cohort will be separated into 2 groups. A sentinel group of 3 subjects (2 active and 1 placebo) will be dosed at least 24 hours before the remaining 5 subjects (4 active and 1 placebo). The remaining cohorts will be dosed in 2 groups of 4 subjects each (3 active and 1 placebo), at least 24 hours apart. |
| | | Food-effect Cohort: Based on exposure levels, subjects in one of the dose |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) |
|---|---|---|
| | | levels will return after a 7-day minimum washout or 5 half-lives of the drug (whichever is longer) to receive the same dose under fed conditions. |
| | | Dose escalation to the next cohort (i.e., dose level) will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort has been demonstrated to permit proceeding to the next cohort. |
| | | Cohort 8: |
| | | There will be 4 arms each consisting of 6 subjects. Subjects will be assigned to one of the following arms and dose: |
| | | • Arm 1 – TBI-223 SR Tablets (Prototype 1) - 1800 mg dose (3 x 600 mg tablets), under fed conditions |
| | | • Arm 2 – TBI-223 SR Tablets (Prototype 2) - 1800 mg dose (3 x 600 mg tablets), under fed conditions |
| | | • Arm 3 – TBI-223 SR Tablets (Prototype 3) - 1800 mg dose (2 x 900 mg tablets), under fed conditions |
| | | <ul> <li>Arm 4 – TBI-223 IR Tablets - 2000 mg dose (2 x 1000 mg tablets),<br/>under fasting conditions</li> </ul> |
| | | Cohort 9: |
| | | The 6 subjects from Cohort 8, Arm 4, who were received IR tablet formulation will be brought back following a 7-day washout – TBI-223 IR Tablets – 2000 mg (2 x 1000 mg tablets), under fed conditions. |
| | | If more than 2 subjects of these 6 subjects from Cohort 8 drop-out, they will be replaced by heathy volunteers (a minimum of 4 subjects are needed to complete Cohort 9). |
| | | Additional cohorts may be enrolled if deemed appropriate (e.g. if bioavailability is lower than expected) by the Sponsor to repeat a dose level, to study other dose levels, change proposed cohorts, or to study a different dosage formulation. These decisions regarding changed or additional cohorts will not take place until the Sponsor, in conjunction with the Principal Investigator and dose escalating committee, has determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort have been demonstrated to permit proceeding to the next cohort. The Institutional Review Board (IRB) should be immediately notified of this revised approach for review and approval. |
| Synopsis | Test product, | From: |
| | dosage and mode of | TBI-223 oral suspension, orally administered |
| | 111040 01 | Dose level 1 = single dose of 50 mg TBI-223 |

| Section | | |
|---|---|---|
| Number | | |
| (s) | Section Title(s) | Description of Change (s) |
| | administration | Dose level 2 = single dose of 100 mg TBI-223 |
| | | Dose level 3 = single dose of 300 mg TBI-223 |
| | | Dose level 4 = single dose of 600 mg TBI-223 |
| | | Dose level 5 = single dose of 1200 mg TBI-223 |
| | | Dose level 6 = single dose of 2000 mg TBI-223 |
| | | Additional cohorts may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level or a different dosage formulation. |
| | | To: |
| | | Part 1: |
| | | TBI-223 oral suspension, orally administered |
| | | Dose level 1 = single dose of 50 mg TBI-223 |
| | | Dose level 2 = single dose of 100 mg TBI-223 |
| | | Dose level 3 = single dose of 300 mg TBI-223 |
| | | Dose level 3 includes a Cohort 3a with TBI-223 (oral suspension) and the same subjects participated in Cohort 3b with TBI-223 within oral enteric capsules |
| | | Dose level 4 = single dose of 600 mg TBI-223 |
| | | Dose level 5 = single dose of 1200 mg TBI-223 |
| | | Dose level 6 = single dose of 2000 mg TBI-223 |
| | | Dose level 7= Single dose of 2600 mg TBI-223 |
| | | Additional cohorts may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level or a different dosage formulation. |
| | | Part 2: |
| | | Cohort 8: |
| | | Arm 1 - TBI-223 SR Tablets 600 mg (Prototype 1). Dose of 1800 mg (3 tablets of 600 mg), under fed conditions |
| | | Arm 2 - TBI-223 SR Tablets 600 mg (Prototype 2). Dose of 1800 mg (3 tablets of 600 mg), under fed conditions |
| | | Arm 3 - TBI-223 SR Tablets 900 mg (Prototype 3). Dose of 1800 mg (2 tablets of 900 mg), under fed conditions Arm 4 - TBI-223 IR Tablets 1000 mg. Dose of 2000 mg (2 tablets of |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) 1000 mg), under fasting conditions Cohort 9: TBI-223 IR Tablets 1000 mg. Dose of 2000 mg (2 tablets of 1000 mg), under fed conditions. Additional cohorts may be enrolled if deemed appropriate by the |
|---|---|---|
| | | Sponsor to repeat a dose level or to study another dose level or a different dosage formulation. |
| Synopsis | Control product,<br>dosage and<br>mode of | Add the following to the beginning of the section: |
| | administration: | Part 1 only: |
| Synopsis | Criteria of evaluation | <ul> <li>Second paragraph. Delete the following pharmacokinetic parameters and definitions:</li> <li>AUC<sub>tau</sub> – area under the concentration time curve during the dosing interval</li> <li>C<sub>avg</sub> – average stead state concentration</li> <li>CLss/F - apparent total clearance at steady state</li> <li>C<sub>min</sub> minimum concentration</li> <li>C<sub>trough</sub>- trough plasma concentration</li> <li>R<sub>AUC</sub> accumulation ration for AUC</li> <li>R<sub>Cmax</sub>- accumulation ratio for C<sub>max</sub></li> </ul> Add the following to the definitions of CL/F and Vz/F |
| | | Delete the third paragraph: Noncompartmental pharmacokinetic parameters of AUC <sub>last</sub> , AUC <sub>inf</sub> , C <sub>max</sub> , T <sub>max</sub> , CL/F, Vz/F, λ <sub>z</sub> , and T <sub>1/2</sub> will be calculated from plasma concentrations of TBI-223 and M2. Additional pharmacokinetic parameters may be calculated if deemed appropriate. Add the following to the fourth paragraph from: Food Effect: The effect of food will be assessed comparing pharmacokinetic parameters under fed versus fasting conditions using an analysis of variance (ANOVA) approach. |

| Section | | |
|---|---|---|
| Number | | |
| (s) | Section Title(s) | Description of Change (s) |
| | | To: |
| | | Food Effect: The effect of food will be assessed comparing pharmacokinetic parameters (C <sub>max</sub> , AUCs) under fed versus fasting conditions using an analysis of variance (ANOVA) approach. |
| 3 | Study Design | Add the following before the first paragraph of the section |
| | Summary | Part 1: |
| | | Add the following to the end of the section, after Table 2 |
| | | Part 2: |
| | | Cohort 8: A minimum of 24 subjects in 4 dosing arms are planned to be enrolled; within each arm, 6 subjects will be assigned to receive a single dose treatment. Subjects will be assigned to one of the following arms and dose: |
| | | • Arm 1 – TBI-223 SR Tablets (Prototype 1) - 1800 mg dose (3 x 600 mg tablets), under fed conditions |
| | | • Arm 2 – TBI-223 SR Tablets (Prototype 2) -1800 mg dose (3 x 600 mg tablets), under fed conditions |
| | | • Arm 3 – TBI-223 SR Tablets (Prototype 3) - 1800 mg dose (2 x 900 mg tablets), under fed conditions |
| | | • Arm 4 – TBI-223 IR Tablets - 2000 mg dose (2 x 1000 mg tablets), under fasting conditions |
| | | Procedures and analyses will be conducted as outlined in Appendix 6. |
| | | Cohort 9: |
| | | The 6 subjects from Cohort 8, Arm 4, who received the IR tablet formulation fasted will return after a 7-day washout and receive a single dose of TBI-223 IR Tablets, 2000 mg dose (2 x 1000 mg tablets), under fed conditions. |
| | | If more than 2 subjects of these 6 subjects from Cohort 8 drop-out, they will be replaced by heathy volunteers (a minimum of 4 subjects are needed to complete Cohort 9). |
| | | Procedures and analyses will be conducted as outlined in Appendix 6. |
| 3.1 | Dose Escalation | Change the title of the section from: |

| Section<br>Number<br>(s) | Section Title(s) | | Description of Change (s) | |
|---|---|---|---|---|
| | | Dose Escalation | | |
| | | To: | | |
| | | Part 1 Dose Escalation | | |
| 3 (pg 12 | Table 2 | Update Table 2 | | |
| 5 (98 12 | 10010 2 | From: | | |
| | | | e planned dose cohorts for the study. | |
| | | Table 2 Planned I | • | |
| | | Cohort <sup>a</sup><br>(Group <sup>b</sup> ) | Dose <sup>c</sup> | |
| | | 1 (sentinel group) | Single dose of 50 mg TBI-223 (n=2) | Placebo (n=1) |
| | | 1 (remainder of cohort) | Single dose of 50 mg TBI-223 (n=4) | Placebo (n=1) |
| | | 2 (Group 1) | Single dose of 100 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 2 (Group 2) | Single dose of 100 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 3 (Group 1) | Single dose of 300 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 3 (Group 2) | Single dose of 300 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 4 (Group 1) | Single dose of 600 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 4 (Group 2) | Single dose of 600 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 5 (Group 1) | Single dose of 1200 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 5 (Group 2) | Single dose of 1200 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 6 (Group 1) | Single dose of 2000 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 6 (Group 2) | Single dose of 2000 mg TBI-223 (n=3) | Placebo (n=1) |
| | | To: | | |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) | | |
|---|---|---|---|---|
| | | Table 2 presents th | tudy. | |
| | | <b>Table 2 Actual Dose Cohorts for Part 1</b> | | |
| | | Cohort <sup>a</sup><br>(Group <sup>b</sup> ) | Dose <sup>c</sup> | |
| | | 1 (sentinel group) | Single dose of 50 mg TBI-223 (n=2) | Placebo (n=1) |
| | | 1 (remainder of cohort) | Single dose of 50 mg TBI-223 (n=4) | Placebo (n=1) |
| | | 2 (Group 1) | Single dose of 100 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 2 (Group 2) | Single dose of 100 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 3a (Group 1) | Single dose of 300 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 3a (Group 2) | Single dose of 300 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 3b (Capsule cohort) | Single dose of 300 mg (TBI oral in oral enteric) (n=4) | N/A |
| | | 4 (Group 1) | Single dose of 600 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 4 (Group 2) | Single dose of 600 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 5 (Group 1) | Single dose of 1200 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 5 (Group 2) | Single dose of 1200 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 6 (Group 1) | Single dose of 2000 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 6 (Group 2) | Single dose of 2000 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 7 (Group 1) | Single dose of 2600 mg TBI-223 (n=3) | Placebo (n=1) |
| | | 7 (Group 2) | Single dose of 2600 mg TBI-223 (n=3) | Placebo (n=1) |
| 4 | Identity of<br>Investigational | Add the following t | to Table 3, Identify of Investigational Pro | oduct |

| Section<br>Number<br>(s) | Section Title(s) | | Description of Change (s) |
|---|---|---|---|
| | Product | From: | |
| | | Test Product: | TBI-223 oral suspension 25 mg/mL Manufactured for Global Alliance for TB Drug Development |
| | | Control<br>Product: | Placebo for TBI-223 oral suspension Manufactured for Global Alliance for TB Drug Development |
| | | To: | 2148201010 |
| | | Part 1 | |
| | | Test Product: | TBI-223 oral suspension 25 mg/mL Manufactured for Global Alliance for TB Drug Development |
| | | Control<br>Product: | Placebo for TBI-223 oral suspension Manufactured for Global Alliance for TB |
| | | Togs Duo du os | Drug Development |
| | | Test Product:<br>Cohort 3b | TBI-223 Oral Enteric Capsules, 150 mg Manufactured for Global Alliance for TB Drug Development |
| | | Part 2 | Drug Development |
| | | Test Products: | TBI-223 SR Tablets 600 mg (Prototype 1) |
| | | Cohort 8<br>(Arms 1-4) | Manufactured for Global Alliance for TB<br>Drug Development by Piramal Enterprise<br>Limited |
| | | | TBI-223 SR Tablets 600 mg (Prototype 2) |
| | | | Manufactured for Global Alliance for TB Drug Development by Piramal Enterprise Limited |
| | | | TBI-223 SR Tablets 900 mg (Prototype 3) Manufactured for Global Alliance for TB Drug Development by Piramal Enterprise Limited |
| | | | TBI-223 IR Tablets 1000 mg Manufactured for Global Alliance for TB Drug Development by Piramal Enterprise |
| | | Test | Limited TBI-223 IR Tablets 1000 mg |
| | | Products:<br>Cohort 9 | Manufactured for Global Alliance for TB Drug Development by Piramal Enterprise Limited |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) |
|---|---|---|
| 6.1 | Subjects | From: |
| | Assignment | Up to 50 subjects are planned to be enrolled in the study. Additional subjects may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level. The number of subjects selected for the study was based on the adequate number considered to provide sufficient safety data. This study has not been formally powered. |
| | | Each subject will receive an assigned treatment (active or placebo) based on the randomization schedule prepared by the unblinded statistician. The unblinded pharmacy staff will ensure compliance with the randomization schedule. |
| | | Note: the repeat cohort using a different dosage formulation will be non-randomized and unblinded; see Appendix 5. |
| | | To: |
| | | For Part 1, up to 50 subjects are planned to be enrolled in the study. Additional subjects may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level. For Part 2, Cohort 8, 24 subjects will be enrolled. For Part 2, Cohort 9, the 6 subjects from Cohort 8 who received the IR tablet formulation fasted will return after a 7-day washout and receive the IR tablet formulation under fed conditions. If more than 2 subjects of these 6 subjects from Cohort 8 drop-out, they will be replaced by heathy volunteers (a minimum |
| | | of 4 subjects are needed to complete Cohort 9). |
| | | The number of subjects selected for the study was based on the adequate number considered to provide sufficient safety data. This study has not been formally powered. |
| | | For Part 1, each subject will receive an assigned treatment (active or placebo) based on the randomization schedule prepared by the unblinded statistician. The unblinded pharmacy staff will ensure compliance with the randomization schedule. |
| | | Note: the repeat cohort using a different dosage formulation in Part 1 and subjects in Part 2 will be non-randomized and unblinded; see Appendix 5 and Appendix 6. |
| 6.3 | Check-in | Update the first sentence from: |
| | Procedures | Subjects will check into the clinic on Day -2. |
| | | To: |
| | | Subjects will check into the clinic on Day -2 for Part 1 and Day -1 for Part 2. |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) |
|---|---|---|
| | | Add the following to the last bullet point: |
| | | (Part 1 only) |
| 6.4 | Confinement | First paragraph, change from: |
| | | Fasting cohorts: Subjects will be admitted to the research center on Day -2 and remain confined until after completion of the 48-hour procedures on Day 3. Subjects will return for a follow-up visit approximately 72 hours after dosing (Day 4) and receive a follow up phone call on Day 11 (+1 day). <i>To:</i> |
| | | Part 1 fasting cohorts and Part 2, Cohort 8, Arm 4 only: Subjects will be admitted to the research center on Day -2 (Part 1) or Day -1 (Part 2) and remain confined until after completion of the 48-hour procedures on Day 3. Subjects will return for a follow-up visit approximately 72 hours after dosing (Day 4) and receive a follow up phone call on Day 11 (+1 day). |
| İ | | Second paragraph, change from: |
| | | Food-effect cohort: Subjects will be admitted to the research center on Day -2 of Period 1 and Period 2 and remain confined until after completion of the 48-hour procedures on Day 3 of each study period. Subjects will return for a follow-up visit approximately 72 hours after dosing (Day 4) in each study period. Subjects will receive a follow up phone call on Day 11 (+1 day) of Period 2. |
| | | To: |
| | | Part 1 food-effect cohort, Part 2, Cohort 8, Arms 1-3 and Cohort 9: Subjects will be admitted to the research center on Day -2 of Period 1 and Period 2 (Part 1) or Day -1 (Part 2) and remain confined until after completion of the 48-hour procedures on Day 3 of each study period. Subjects will return for a follow-up visit approximately 72 hours after dosing (Day 4) in each study period. Subjects will receive a follow up phone call on Day 11 (+1 day) of Period 2. |
| | | Please note that Cohort 9 is the same 6 subjects that were in Cohort 8, Arm 4 (IR tablet formulation) under fed conditions. In Cohort 8, Arm 4, subjects fasted. |
| 6.5.1 | Fasting/Meals | First paragraph, change from: |
| | | <u>Fasted cohorts</u> : Optional meals (lunch, snack, and dinner) may be served the day of check-in. All subjects will then be required to fast for at least 10 hours before dosing. The subjects will fast for 4 hours after dosing. Standard meals will be provided at appropriate times after dosing. |
| | | To: |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) |
|---|---|---|
| | | Part 1 fasted cohorts and Part 2, Cohort 8, Arm 4 only: Optional meals (lunch, snack, and dinner) may be served the day of check-in. All subjects will then be required to fast for at least 10 hours before dosing. The subjects will fast for 4 hours after dosing. Standard meals will be provided at appropriate times after dosing. |
| | | Second paragraph, change from: |
| | | Food-effect cohort: Optional meals (lunch, snack, and dinner) may be served the day of check-in. |
| | | To: |
| | | Part 1 food-effect cohort, Part 2, Cohort 8, Arms 1-3 and Cohort 9: Optional meals (lunch, snack, and dinner) may be served the day of check-in. |
| | | Fourth paragraph, first sentence, change from: |
| | | In the fed study period. Subjects will be required to fast for at least 10 hours overnight before consuming a required FDA standard high-fat, high-calorie breakfast. |
| | | To: |
| | | In the fed study period of Part 1 and Part 2 (Cohort 8, Arms 1-3 and Cohort 9), subjects will be required to fast for at least 10 hours overnight before consuming a required FDA standard high-fat, high-calorie breakfast. |
| | | Add the following to the end of the section: |
| | | Please note that Part 2, Cohort 9 is the same 6 subjects that were in Cohort 8 Arm 4 (IR tablet formulation) under fed conditions. In Cohort 8 Arm 4, subjects fasted. |
| 6.6 | Drug | Add the following subsection: |
| | administration | 6.6.3 Administration of TBI-223 SR and IR Tablets |
| | | Add the following to the new section: |
| | | For Part 2, Cohort 8 and Cohort 9, each subject will receive the oral dose of the assigned study treatment (TBI-223 SR tablet formulations [Prototypes 1, 2, or 3] or TBI-223 IR tablet formulation) with approximately 240 mL (8 fl. oz.) of room temperature water. Subjects must swallow the study medication intact. The medication should NOT be crushed or chewed. A hand and mouth check will be performed immediately after dose to ensure that the medication has been appropriately swallowed. The subjects will remain seated, except as otherwise required for study procedures or personal needs, for the first 4 hours after dosing. Should the need to move about occur during the first 4 hours after each dose, |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) |
|---|---|---|
| | | subjects may be escorted to such procedures or activities by research personnel as deemed medically necessary. Subjects will not be allowed to lie down, except as directed by clinical staff secondary to AEs, for the first 4 hours after dosing. |
| 6.7.1 | Fasting cohort | Change title of section from: Fasting cohort To: Part 1 fasting cohorts, Part 2, Cohort 8, Arm 4 only |
| 6.7.2 | Food-effect<br>cohort | Change title of section from: Food-effect cohort To: Part 1 food-effect cohort, Part 2, Cohort 8, Arms 1-3 only, and Cohort 9 Add the following after the first paragraph: Please note that Part 2, Cohort 9 is the same 6 subjects that were in Cohort 8 Arm 4 (IR tablet formulation) under fed conditions. In Cohort 8 Arm 4, subjects fasted. |
| 6.9.7 | Cardiac Holter<br>Monitoring, and<br>Cardiodynamic<br>Assessment | Add the following sentence to the end of the section: Part 2 of the study will not have cardiac Holter monitoring. |
| 8.4 | Indications for<br>Subject<br>Withdrawal | Add the following paragraphs to the end of the section: Subjects who experience emesis may be replaced if the emesis could potentially impact drug absorption and therefore the pharmacokinetic data. Cases of emesis will be evaluated by the Sponsor and Principal Investigator to determine if subject replacement is needed. For Part 1, replacement subjects will be numbered 17XX where XX is 10 plus the original subject's last 2 assigned numbers (e.g. if subject 1702 needs to be replaced due to emesis, the replacement subject number would be 1712). Replacement subjects will receive the same dose allocation of study drug. |
| 9.2 | Pharmacokinetic<br>Analysis | Add the following to the definitions of CL/F and Vz/F: (TBI-223 only) Deleted the first sentence from third paragraph, from: Noncompartmental pharmacokinetic parameters of AUC <sub>last</sub> , AUC <sub>inf</sub> , C <sub>max</sub> , T <sub>max</sub> , CL/F, Vz/F, λ <sub>z</sub> , and T <sub>1/2</sub> will be calculated from plasma concentrations of TBI-223 and M2. Additional pharmacokinetic parameters may be |

| Section<br>Number | | |
|---|---|---|
| (s) | Section Title(s) | Description of Change (s) |
| | | calculated if deemed appropriate. |
| | | To: |
| | | Additional pharmacokinetic parameters may be calculated if deemed appropriate. |
| | | Add the following to last paragraph, from: |
| | | Food Effect: The effect of food will be assessed comparing pharmacokinetic parameters under fed versus fasting conditions using an analysis of variance (ANOVA) approach. |
| | | To: |
| | | Food Effect: The effect of food will be assessed comparing pharmacokinetic parameters (C <sub>max</sub> , AUCs) under fed versus fasting conditions using an analysis of variance (ANOVA) approach. |
| 9.3 | Statistical | Second and third paragraph, change from: |
| | Analysis | Pharmacokinetic parameters will be summarized by cohort using descriptive statistics. Summary statistics will also be presented by gender within each cohort. Dose proportionality will be assessed using a power model approach. |
| | | Food-effect cohort: The effect of food will be assessed comparing pharmacokinetic parameters under fed versus fasting conditions using an analysis of variance (ANOVA) approach. |
| | | To: |
| | | Pharmacokinetic parameters will be summarized by cohort using descriptive statistics. Summary statistics will also be presented by gender within each cohort. Dose proportionality <b>for exposure parameters</b> (C <sub>max</sub> , AUCs) will be assessed using a power model approach. |
| | | Food-effect cohort: The effect of food will be assessed comparing pharmacokinetic parameters ( $C_{max}$ , AUCs) under fed versus fasting conditions using an analysis of variance (ANOVA) approach. |
| 11 | Drug Supplies | Add the following to the end of the section: |
| | | Global Alliance for TB Drug Development will supply sufficient quantity of the study drug, TBI 223 SR tablet formulations (Prototypes 1, 2, and 3) and TBI-223 IR tablet formulation for Part 2 of the study. |
| | | Study drug formulations will be shipped to Worldwide Clinical Trials Early Phase Services, LLC pursuant to site standard operating procedures. Upon receipt of the study drug products, the supplies will be inventoried and stored in an environmentally controlled and secure, limited access area. The lot numbers of the drugs along with the |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) expiration dates (where available) will be recorded and copies of the Certificate of Analysis (where available) will be maintained on file. Records will be maintained of the receipt and dispensation of the drugs supplied. At the conclusion of the study, any unused study drug will be returned to the sponsor or destroyed by the site pursuant to written authorization by the sponsor and applicable federal and state regulations. |
|---|---|---|
| Table 9 | Schedule of<br>Assessments | Change title of table from: Schedule of Assessments To: Schedule of Assessments, Part 1 |
| Appendix 2 | Description and Composition of Test Product | |

| Section<br>Number | Section Title(s) | | Dogavintian | of Change (s) | |
|---|---|---|---|---|---|
| (s) | Section Title(s) | Vcaps® Enteric<br>Capsules¹, Off-<br>white, Opaque, Size<br>00 | Capsule shell | of Change (s) Commerciall available | y 2 capsules |
| | | | <b>Total Quantity</b> | | 300 mg in 2 capsules |
| | | <sup>1</sup> Capsule shell composition: titanium dioxide 2% in Hypromellose-Hypromellos AS. Container and Closure System TBI-223 Oral Enteric Capsules are stored in white HDPE bottles with PP CRC with a liner. These bottles are used for storage prior to | | | |
| | | administration. Tablets Description of the Dosage Form | | | |
| | | | n of the tablets a | nd strengths are | R) or sustained release presented in Table 11. SBI-223 IR and SR |
| | | Tablet Strength | Tablet | Weight | Tablet Appearance |
| | | T | BI-223 Immediate | | |
| | | 600 mg | 75 | 0 mg | White to off-white, capsule shaped tablets, lebossed with "TBA" on one side and "22" on the other |
| | | 1000 mg | 125 | 50 mg | White to off-white, oval shaped tablets, debossed with "TBA" on one side and "23" on the other |
| | | TBI-223 Sustained Release (SR) Tablets | | | |
| | | 600 mg (Prototype | | 00 mg d | White to off-white, capsule shaped tablets, lebossed with "TBA" on one side and "11" on the other |
| | | 600 mg (Prototype | 2) 100 | | White to off-white, |

| Section<br>Number<br>(s) | Section Title(s) | | Descript | tion of Chan | ge (s) | | |
|---|---|---|---|---|---|---|---|
| | | | | | deb<br>one | sule shape<br>ossed with<br>side and '<br>other | "TBA" on |
| | | 900 mg (Prototyp | ne 3) | 1200 mg | sha <sub>l</sub><br>with | ped tablets | vhite, oval<br>s, debossed<br>on one side<br>the other |
| | | Composition of the | e Drug Produc | ct | | | _ |
| | | The composition of in Table 12. The composition of the composition of | composition of<br>ype 2) and 900<br>Table 15, respe<br>on of TBI-223 I | TBI-223 SR<br>O mg (prototy<br>ectively. | Tablets<br>ype 3) is | , 600 mg<br>presented | (Prototype d in Table |
| | | Component | Function | (% w/w) | mg/t | tablet | to<br>Standard |
| | | | | Intr | agranula | r | _ |
| | | TBI-223 a | Active | 80.00 | 600.00 | 1000.00 | In-House |
| | | Microcrystalline cellulose (Avicel PH 302) | Diluent | 10.00 | 75.00 | 125.00 | USP-NF,<br>Ph.Eur. |
| | | Hypromellose<br>(Methocel E5<br>Premium LV) | Binder | 3.00 | 22.50 | 37.50 | USP-NF,<br>Ph.Eur. |
| | | Crospovidone (Kollidon CL) | Disintegrant | 3.00 | 22.50 | 37.50 | USP-NF,<br>Ph.Eur. |
| | | Purified water <sup>c</sup> | Granulating solvent | q.s | q.s | q.s | USP,<br>Ph.Eur. |
| | | Extragranular | | | | _ | |
| | | Crospovidone<br>(Kollidon CL)<br>Colloidal silicon | Disintegrant | 2.00 | 15.00 | 25.00 | USP-NF,<br>Ph.Eur. |
| | | dioxide<br>(Aerosil 200<br>Pharma) | Glidant | 1.00 | 7.50 | 12.50 | USP-NF,<br>Ph.Eur. |
| | | Magnesium<br>stearate<br>(Ligamed MF-2-<br>V) | Lubricant | 1.00 | 7.50 | 12.50 | USP-NF,<br>Ph.Eur. |

| Section<br>Number<br>(s) | Section Title(s) | | Description | of Change | (s) | |
|---|---|---|---|---|---|---|
| | | Total unit dose | | 100.00 7 | 50.0 1250 | .0 |
| | | <ul> <li>The molecular weight of TBI-223 is 365.4 g/mol. The actual quant be adjusted based on the assay value (anhydrous basis) and water content of the drug substance lot used.</li> <li>The quantity of microcrystalline cellulose may be adjusted to compensate for the actual amount of TBI-223 and to maintain a ctablet weight.</li> <li>Removed during processing.</li> </ul> | | | | |
| | | Table 13 Composition of | of TBI-223 SR T | ablets, 600 m | ng (Prototype | |
| | | Component | Function | Percentage<br>(% w/w) | mg/tablet | Reference<br>to<br>Standard |
| | | | | Intragr | anular | |
| | | TBI-223 a | Active | 60.00 | 600.00 | In-House |
| | | Lactose<br>monohydrate <sup>b</sup><br>(Pharmatose<br>200M) | Diluent | 9.90 | 99.00 | USP-NF,<br>Ph.Eur. |
| | | Microcrystalline<br>cellulose<br>(Avicel PH 200) | Diluent | 6.60 | 66.00 | USP-NF,<br>Ph.Eur. |
| | | Hypromellose<br>(Methocel E5<br>Premium LV) | Binder | 5.00 | 50.00 | USP-NF,<br>Ph.Eur. |
| | | Purified water <sup>c</sup> | Granulating solvent | q.s | q.s | USP,<br>Ph.Eur. |
| | | | | Extragranular | | |
| | | Hypromellose<br>(Methocel K100M<br>Premium DC2) | Control<br>Release<br>Polymer | 16.00 | 160.00 | USP-NF,<br>Ph.Eur. |
| | | Colloidal silicon<br>dioxide<br>(Aerosil 200<br>Pharma) | Glidant | 1.50 | 15.00 | USP-NF,<br>Ph.Eur. |
| | | Magnesium<br>stearate<br>(Ligamed MF-2-<br>V) | Lubricant | 1.00 | 10.00 | USP-NF,<br>Ph.Eur. |
| | | Total unit dose | | 100.00 | 1000.0 | |

| Section<br>Number<br>(s) | Section Title(s) | | Description | of Change ( | s) | |
|---|---|---|---|---|---|---|
| (4) | | a The molecular way be adjusted water content of The quantity of for the actual an weight. | veight of TBI-22 l based on the a f the drug substa<br>lactose monohy nount of TBI-22 g processing. | 23 is 365.4 g/n<br>ssay value (an<br>ance lot used.<br>drate may be<br>23 and to main | nol. The actu<br>hydrous bas<br>adjusted to ontain a const | is) and<br>compensate<br>ant tablet |
| | | Component | Function | Percentage<br>(% w/w) | mg/tablet | Reference<br>to<br>Standard |
| | | | | Intragr | anular | |
| | | TBI-223 a | Active | 60.00 | 600.00 | In-House |
| | | Lactose<br>monohydrate <sup>b</sup><br>(Pharmatose<br>200M) | Diluent | 12.90 | 129.00 | USP-NF,<br>Ph.Eur. |
| | | Microcrystalline<br>cellulose<br>(Avicel PH 200) | Diluent | 8.60 | 86.00 | USP-NF,<br>Ph.Eur. |
| | | Hypromellose<br>(Methocel K4M<br>Premium CR) | Control<br>Release<br>Polymer | 5.00 | 50.00 | USP-NF,<br>Ph.Eur. |
| | | Purified water <sup>c</sup> | Granulating solvent | q.s | q.s | USP,<br>Ph.Eur. |
| | | | | Extragr | Extragranular | |
| | | Hypromellose<br>(Methocel K100<br>Premium LV)<br>Colloidal silicon | Control<br>Release<br>Polymer | 11.00 | 110.00 | USP-NF,<br>Ph.Eur. |
| | | dioxide<br>(Aerosil 200<br>Pharma) | Glidant | 1.50 | 15.00 | USP-NF,<br>Ph.Eur. |
| | | Magnesium<br>stearate<br>(Ligamed MF-2-V) | Lubricant | 1.00 | 10.00 | USP-NF,<br>Ph.Eur. |
| | | Total unit dose | | 100.00 | 1000.0 | |

| Section<br>Number<br>(s) | Section Title(s) | | Description | of Change (s | s) | |
|---|---|---|---|---|---|---|
| | | The molecular w may be adjusted water content of The quantity of l for the actual an weight. Removed during | based on the as<br>the drug substa<br>actose monohy-<br>nount of TBI-22<br>g processing. | ssay value (an<br>ance lot used.<br>drate may be<br>3 and to mair | hydrous bas<br>adjusted to c<br>ntain a const | is) and<br>compensate<br>ant tablet |
| | | Component | Function | ablets, 900 mg Percentage (% w/w) | g (Prototype<br>mg/tablet | Reference<br>to<br>Standard |
| | | | | Intragr | anular | |
| | | TBI-223 a | Active | 75.00 | 900.00 | In-House |
| | | Lactose<br>monohydrate b<br>(Pharmatose<br>200M) | Diluent | 3.90 | 46.80 | USP-NF,<br>Ph.Eur. |
| | | Microcrystalline<br>cellulose<br>(Avicel PH 200) | Diluent | 2.60 | 31.20 | USP-NF,<br>Ph.Eur. |
| | | Hypromellose<br>(Methocel E5<br>Premium LV) | Binder | 5.00 | 60.00 | USP-NF,<br>Ph.Eur. |
| | | Purified water <sup>c</sup> | Granulating solvent | q.s | q.s | USP.<br>Ph.Eur. |
| | | | | Extragr | anular | |
| | | Hypromellose<br>(Methocel K100M<br>Premium DC2) | Control<br>Release<br>Polymer | 11.00 | 132.00 | USP-NF,<br>Ph.Eur. |
| | | Colloidal silicon<br>dioxide<br>(Aerosil 200<br>Pharma) | Glidant | 1.50 | 18.00 | USP-NF,<br>Ph.Eur. |
| | | Magnesium<br>stearate<br>(Ligamed MF-2-V) | Lubricant | 1.00 | 12.00 | USP-NF,<br>Ph.Eur. |
| | | Total unit dose | | 100.00 | 1200.0 | |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) |
|---|---|---|
| | | <ul> <li>The molecular weight of TBI-223 is 365.4 g/mol. The actual quantity may be adjusted based on the assay value (anhydrous basis) and water content of the drug substance lot used.</li> <li>The quantity of lactose monohydrate may be adjusted to compensate for the actual amount of TBI-223 and to maintain a constant tablet weight.</li> <li>Removed during processing.</li> </ul> |
| | | Container and Closure System |
| | | TBI-223 IR and SR Tablets are packaged as 30-count in 100 cc round high-density polyethylene (HDPE) bottles and closed with aluminum foil lined heat induction seals and 38 mm polypropylene (PP) child resistant closures (CRC). |
| Appendix | Part 2 of the | Add the following: |
| 6 | study | Procedures and analyses as outlined in this protocol will be the same, with the following exceptions: |
| | | The dose of TBI-223 will be delivered as follows in Cohort 8: |
| | | <ul> <li>Arm 1 – TBI-223 SR Tablets (Prototype 1) - 1800 mg dose (3 x 600 mg tablets), under fed conditions</li> </ul> |
| | | <ul> <li>Arm 2 – TBI-223 SR Tablets (Prototype 2) - 1800 mg dose (3 x 600 mg tablets), under fed conditions</li> </ul> |
| | | <ul> <li>Arm 3 – TBI-223 SR Tablets (Prototype 3) - 1800 mg dose (2 x 900 mg tablets), under fed conditions</li> </ul> |
| | | <ul> <li>Arm 4 – TBI-223 IR Tablets - 2000 mg dose (2 x 1000 mg<br/>tablets), under fasting conditions</li> </ul> |
| | | In Cohort 9, the subjects from Cohort 8, Arm 4, who received the IR tablet formulation will be brought back following a 7-day washout and administered TBI-223 IR tablets, 2000 mg dose (2 x 1000 mg tablets), under fed conditions. |
| | | • A minimum of 6 subjects per treatment arm in Part 2 |
| | | <ul> <li>Part 2 will not be blinded (blinding is not necessary because all<br/>subjects will receive the same treatment).</li> </ul> |
| | | <ul> <li>Cardiac telemetry and Holter recording will not be performed<br/>during Part 2. Subjects will check-in on Day -1 instead of Day -2.<br/>With the exception of cardiac telemetry and Holter monitoring,<br/>the procedures that were previously scheduled for Day -2 will be<br/>performed on Day -1. The Day -1 results will be used to qualify<br/>repeat subjects for study participation. If additional subjects are</li> </ul> |

| Section<br>Number<br>(s) | Section Title(s) | Description of Change (s) |
|---|---|---|
| | | needed, they will undergo screening to qualify for the study. |
| | | <ul> <li>Neurological examinations will be performed at Screening, Day -<br/>1, and at 3 and 48 hours postdose.</li> </ul> |
| | | Add Table 16, Schedule of Assessments, Part 2 |

#### PROTOCOL SYNOPSIS

Name of Sponsor/Company: Global Alliance for TB Drug Development

Name of test product: TBI-223 oral suspension

Name of active ingredient: TBI-223

**Title of study:** A Phase 1, Partially-Blinded, Placebo-Controlled, Randomized, Single Ascending Dose (SAD) with a Food Effect Cohort Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBI-223 in Healthy Adult Participants

Principal Investigator: Cynthia A. Zamora, MD

## **Study Center**

Worldwide Clinical Trials Early Phase Services, LLC 2455 NE Loop 410, Suite 150 San Antonio, Texas 78217

**Study period** (maximum duration, from screening to study exit):

#### Part 1:

Single ascending dose (SAD) cohort (fasting): 40 days

Food-effect cohort: 50 days

#### Part 2:

**Cohort 8:** Single dose cohort of the 4 TBI-223 tablet formulations (Prototypes 1, 2, and 3 Sustained Release [SR] tablet formulations under fed conditions and one Immediate Release [IR] tablet formulation under fasting conditions): Duration 40 days.

**Cohort 9:** The IR tablet formulation will be evaluated under fed conditions

Single dose: 40 days

The maximum duration of the study will depend upon the final number and timing of each cohort.

# Number of sites enrolling subjects: 1

Phase of development: 1

#### **Duration of treatment:**

# Part 1:

<u>Fasting cohorts</u>: One single dose of TBI-223 oral suspension or placebo for TBI-223 oral suspension <u>Food-effect cohort</u>: Two single doses of TBI-223 oral suspension or placebo for TBI-223 oral suspension separated by a washout period of at least 7 days

# Part 2:

**Cohort 8:** Single dose cohort of 4 TBI-223 tablet formulations (Three SR tablet formulations as prototypes 1, 2, and 3 and one IR tablet formulation). The SR tablet formulations will be evaluated under fed conditions and the IR tablet formulation will be evaluated under fasting conditions

**Cohort 9:** The IR tablet formulation will be evaluated under fed conditions

# Number of subjects (planned):

#### Part 1:

<u>Fasting Cohorts</u>: Planned to enroll up to 48 subjects in a total of 6 single ascending dose (SAD) cohorts of 8 subjects each (6 to receive active drug and 2 to receive placebo).

<u>Food-effect Cohort</u>: 1 cohort with 10 subjects (8 active and 2 placebo) who will receive TBI-223 or placebo under both fasting and fed conditions.

#### Part 2:

**Cohort 8:** Planned to enroll 24 subjects in a total of 4 arms with 6 subjects in each. Subjects will receive a single dose of 1 of the 3 prototypes of TBI-223 SR tablets under fed conditions (Arms 1-3) or a single dose of TBI-223 IR tablets under fasted conditions (Arm 4).

**Cohort 9:** Plan to bring back the 6 subjects from Cohort 8, Arm 4, who received the IR tablet formulation, following a 7-day washout to receive the IR tablet formulation under fed conditions.

If more than 2 subjects of these 6 subjects from Cohort 8 drop-out, they will be replaced by heathy volunteers (a minimum of 4 subjects are needed to complete Cohort 9).

Additional cohorts may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level. These decisions on additional cohorts will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort have been demonstrated to permit proceeding to the next cohort. The Institutional Review Board (IRB) should be immediately notified of this revised approach.

# Diagnosis and main criteria for inclusion:

Volunteers will be healthy adult male or female, ages 19 to 50 years (inclusive) at screening, with a body mass index (BMI)  $\geq$ 18.5 and  $\leq$ 32.0 kg.m<sup>2</sup> and body weight of no less than 50.0 kg, who do not use tobacco or nicotine-containing products. Females must be of non-childbearing potential or must use an allowable method of birth control.

# **Objectives:**

The primary objective of the study is:

• To evaluate the safety and tolerability of single ascending doses of TBI-223 oral suspension, TBI-223 oral enteric capsules, and TBI-223 tablet formulations in healthy adult subjects.

The secondary objectives of the study are:

- To determine the pharmacokinetics of TBI-223 and its metabolite M2 after single doses of TBI-223 oral suspension, TBI-223 oral enteric capsules, and TBI-223 tablet formulations in healthy adult subjects; and
- To compare the rate and extent of absorption of a single dose of TBI-223 oral suspension, TBI-223 oral enteric capsules, and TBI-223 tablet formulations when administered in healthy adult subjects either after a high-calorie, high-fat meal or in the fasting state.

This is a partially-blinded, placebo-controlled, randomized SAD study with a food effect cohort. The study will be conducted at one study center in the United States.

Safety will be assessed throughout the study for all subjects.

Blood will be collected for pharmacokinetic analysis. Plasma samples will be analyzed for TBI-223 and TBI-223 metabolite (M2).

#### Part 1:

There will be up to 6 planned dose levels. Based on interim pharmacokinetic data obtained during the dose escalation, a dose cohort will be selected to return for additional dosing after a high-calorie, high-fat meal (food-effect cohort).

Sentinel Cohort: The first cohort will be separated into 2 groups. A sentinel group of 3 subjects (2 active and 1 placebo) will be dosed at least 24 hours before the remaining 5 subjects (4 active and 1 placebo). The remaining cohorts will be dosed in 2 groups of 4 subjects each (3 active and 1 placebo), at least 24 hours apart.

<u>Food-effect Cohort</u>: Based on exposure levels, subjects in one of the dose levels will return after a 7-day minimum washout or 5 half-lives of the drug (whichever is longer) to receive the same dose under fed conditions.

Dose escalation to the next cohort (i.e., dose level) will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort has been demonstrated to permit proceeding to the next cohort.

#### Part 2:

#### Cohort 8:

There will be 4 arms each consisting of 6 subjects. Subjects will be assigned to one of the following arms and dose:

- Arm 1 TBI-223 SR Tablets (Prototype 1) 1800 mg dose (3 x 600 mg tablets), under fed conditions
- Arm 2 TBI-223 SR Tablets (Prototype 2) 1800 mg dose (3 x 600 mg tablets), under fed conditions
- Arm 3 TBI-223 SR Tablets (Prototype 3) 1800 mg dose (2 x 900 mg tablets), under fed

# conditions

• Arm 4 – TBI-223 IR Tablets - 2000 mg dose (2 x 1000 mg tablets), under fasting conditions

# Cohort 9:

The 6 subjects from Cohort 8, Arm 4, who received the IR tablet formulation will be brought back following a 7-day washout – TBI-223 IR Tablets – 2000 mg (2 x 1000 mg tablets), under fed conditions.

If more than 2 subjects of these 6 subjects from Cohort 8 drop-out, they will be replaced by heathy volunteers (a minimum of 4 subjects are needed to complete Cohort 9).

Additional cohorts may be enrolled if deemed appropriate (e.g. if bioavailability is lower than expected) by the Sponsor to repeat a dose level, to study other dose levels, change proposed cohorts, or to study a different dosage formulation. These decisions regarding changed or additional cohorts will not take place until the Sponsor, in conjunction with the Principal Investigator and dose escalating committee, has determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort have been demonstrated to permit proceeding to the next cohort. The Institutional Review Board (IRB) should be immediately notified of this revised approach for review and approval.

Page xxxi

# Test product, dosage and mode of administration:

#### Part 1:

TBI-223 oral suspension, orally administered

Dose level 1 = single dose of 50 mg TBI- 223

Dose level 2 = single dose of 100 mg TBI- 223

Dose level 3 = single dose of 300 mg TBI- 223

Dose level 3 includes a Cohort 3a with TBI-223 (oral suspension) and the same subjects participated in Cohort 3b with TBI-223 within oral enteric capsules

Dose level 4 = single dose of 600 mg TBI- 223

Dose level 5 = single dose of 1200 mg TBI- 223

Dose level 6 = single dose of 2000 mg TBI-223

Dose level 7= Single dose of 2600 mg TBI-223

Additional cohorts may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level or a different dosage formulation.

#### Part 2:

#### Cohort 8:

**Arm 1 -** TBI-223 SR Tablets 600 mg (Prototype 1). Dose of 1800 mg (3 tablets of 600 mg), under fed conditions

**Arm 2 -** TBI-223 SR Tablets 600 mg (Prototype 2). Dose of 1800 mg (3 tablets of 600 mg), under fed conditions

**Arm 3 -** TBI-223 SR Tablets 900 mg (Prototype 3). Dose of 1800 mg (2 tablets of 900 mg), under fed conditions

**Arm 4 -** TBI-223 IR Tablets 1000 mg. Dose of 2000 mg (2 tablets of 1000 mg), under fasting conditions

#### Cohort 9:

TBI-223 IR Tablets 1000 mg. Dose of 2000 mg (2 tablets of 1000 mg), under fed conditions.

Additional cohorts may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level or a different dosage formulation.

# Control product, dosage and mode of administration:

#### Part 1 only:

Placebo for TBI-223 oral suspension; orally administered

All levels = Single dose of placebo for TBI-223 oral suspension

#### **Criteria for evaluation:**

Safety: Safety assessments will include physical and neurological examinations, vital signs including heart rate and respiratory rate, electrocardiograms (ECGs), cardiac monitoring, adverse events (AEs), and clinical laboratory tests (including hematology, serum chemistry, coagulation, and urinalysis). Female subjects will have blood collected for serum pregnancy testing. Females claiming postmenopausal status will have blood collected to measure follicle stimulating hormone (FSH) levels.

Pharmacokinetics: Final pharmacokinetic calculations will be performed using appropriate software, e.g. Phoenix™ WinNonlin® (Version 8.1 or higher, Certara, L.P. in conjunction with the internet-accessible implementation of Pharsight® Knowledgebase Server™ [PKSO; Version 4.0.4 or higher, Certara, L.P.]) and/or SAS® (Version 9.4 or higher, SAS Institute Inc.). Pharmacokinetic parameters will be calculated using non-compartmental analysis. The following pharmacokinetic parameters will be determined as appropriate for each study part.

| AUC <sub>Extrap</sub> (%) | The percentage of extrapolated AUC to AUC <sub>inf</sub> based on extrapolation |
|---|---|
| AUCinf | Area under the concentration-time curve from time-zero extrapolated to infinity; calculated as: $AUC_{\rm inf} = AUC_{\rm last} + \frac{C_{\rm last}}{\lambda_z}$ |
| AUC <sub>last</sub> | Area under the concentration-time curve from time-zero to the time of the last quantifiable concentration; calculated using the linear trapezoidal rule |
| C <sub>last</sub> | The last quantifiable concentration determined directly from individual concentration-time data |
| CL/F | Apparent total clearance after single administration (TBI-223 only) |
| C <sub>max</sub> | Maximum concentration, determined directly from individual concentration-time data |
| $T_{last}$ | Time of the last quantifiable concentration |
| $T_{\text{max}}$ | Time of the maximum concentration |
| T <sub>1/2</sub> | The observed terminal half-life, calculated as: $T_{1/2} = \frac{\ln(2)}{\lambda_z}$ |
| Vz/F | Apparent volume of distribution in the terminal phase (TBI-223 only) |
| $\lambda_{\rm z}$ | The observed terminal rate constant; estimated by linear regression through at least 3 data points in the terminal phase of the log concentration-time profile |

Pharmacokinetic parameters will be summarized by cohort using descriptive statistics. Dose proportionality will be assessed using the power model approach.

Food Effect: The effect of food will be assessed comparing pharmacokinetic parameters (C<sub>max</sub>, AUCs) under fed versus fasting conditions using an analysis of variance (ANOVA) approach.

Efficacy: No efficacy evaluations will be performed in this study.

# **TABLE OF CONTENTS**

| PROT | ГОСОL APPROVAL PAGE | i |
|-------|------------------------------------------------|----------|
| SUM | MARY OF CHANGES | ii |
| PROT | TOCOL SYNOPSIS | xxvii |
| TABI | LE OF CONTENTS | XXXV |
| | OF TABLES | |
| LIST | OF FIGURES | xxxvii |
| LIST | OF ABBREVIATIONS | xxxix |
| 1 | INTRODUCTION | 1 |
| 1.1 | Background Information | |
| 1.2 | Tuberculosis and Rationale for New Medications | 1 |
| 1.3 | Preclinical Studies and Toxicity Studies | |
| 1.4 | Adverse Effects, Warnings, and Precautions | |
| 1.5 | Overview and Dose Rationale | <i>.</i> |
| 2 | OBJECTIVE | g |
| 3 | STUDY DESIGN SUMMARY | 9 |
| 3.1 | Part 1 Dose Escalation | 13 |
| 3.2 | Stopping Rules for Cohorts | |
| 4 | IDENTITY OF INVESTIGATIONAL PRODUCT | 14 |
| 5 | SUBJECT SELECTION | 15 |
| 5.1 | Inclusion Criteria | 15 |
| 5.2 | Exclusion Criteria | 17 |
| 5.3 | Medication and Activity Restrictions | 20 |
| 5.4 | Screening | 21 |
| 6 | STUDY PROCEDURES | 21 |
| 6.1 | Subject Assignment | 21 |
| 6.2 | Blinding | 22 |
| 6.2.1 | Clinical Research Staff | 23 |
| 6.2.2 | Study Subjects | 23 |
| 6.2.3 | Bioanalytical Laboratory | |
| 6.2.4 | Pharmacokinetic Analysis | 23 |
| 6.2.5 | Cardiac Vendor | 23 |
| 6.2.6 | Unblinding Procedures | 23 |
| 6.3 | Check-In Procedures | 23 |
| 6.4 | Confinement | 24 |
| 6.5 | Fasting/Meals/Beverages | |
| 6.5.1 | Fasting/Meals <sup>3</sup> | 24 |
| 6.5.2 | Beverages | 25 |
| 6.6 | Drug Administration | |
| 6.6.1 | Administration of oral care strips | 25 |

| 6.6.2 | Administration of TBI-223 Oral Suspension or Placebo for TBI-223 Oral Suspension. | 26 |
|---|---|---|
| 6.6.3 | Administration of TBI-223 Sustained Release and Immediate Release Tablets | 26 |
| 6.7 | Blood Sampling, Processing and Shipment | 27 |
| 6.7.1 | Part 1 fasting cohorts, and Part 2, Cohort 8, Arm 4 only | 27 |
| 6.7.2 | Part 1 food-effect cohort, Part 2, Cohort 8, Arms 1-3 only, and Cohort 9 | 27 |
| 6.7.3 | Pharmacokinetic Sampling Time Windows | 28 |
| 6.8 | End-of-Study Procedures | 28 |
| 6.9 | Safety Monitoring and Procedures | 29 |
| 6.9.1 | Adverse Events | 29 |
| 6.9.2 | Clinical Laboratory Evaluations | 29 |
| 6.9.3 | Vital Signs | 30 |
| 6.9.4 | Physical Examinations | 30 |
| 6.9.5 | Neurological Examinations | 30 |
| 6.9.6 | 12-Lead Electrocardiograms | 31 |
| 6.9.7 | Cardiac Holter Monitoring, and Cardiodynamic Assessment | 31 |
| 6.9.8 | Other Safety Measures | 31 |
| 7 | ADVERSE EVENTS | 32 |
| 7.1 | Definitions | 32 |
| 7.1.1 | Adverse Event | 32 |
| 7.1.2 | Serious Adverse Event | 32 |
| 7.2 | Attribution/Causality | 33 |
| 7.3 | Reporting | 35 |
| 7.3.1 | Adverse Event | 35 |
| 7.4 | Serious Adverse Event Reporting | 35 |
| 7.5 | Follow up of Adverse Events | 36 |
| 7.6 | Post-Trial Serious Adverse Events | 37 |
| 7.7 | Clinical Laboratory Adverse Events | 37 |
| 7.8 | Drug Interaction | 38 |
| 7.9 | Pregnancy | 38 |
| 7.10 | Monitoring and Safety for Specific Toxicities | 38 |
| 8 | GENERAL CONSIDERATIONS | 38 |
| 8.1 | Basic Principles | 38 |
| 8.2 | Institutional Review Board | 39 |
| 8.3 | Informed Consent | 39 |
| 8.4 | Indications for Subject Withdrawal | 39 |
| 8.5 | Termination of the Study | 39 |
| 8.6 | Documentation | 40 |
| 8.7 | Trial Monitoring. | 40 |
| 8.8 | Reimbursement, Indemnity, and Insurance | 40 |
| 9 | PHARMACOKINETIC ANALYSIS | 40 |
| 9.1 | Analytical Methodology | 40 |
| 9.2 P | harmacokinetic Analysis | 40 |
|---|---|---|
| 9.3 S | tatistical Analysis | 42 |
| 10 F | ACILITIES | 42 |
| 11 I | DRUG SUPPLIES | 43 |
| 12 A | ADMINISTRATIVE ISSUES | 44 |
| 13 E | VENTS SCHEDULE | 45 |
| 14 F | EFERENCES | 48 |
| | DIX 1 PHARMACOKINETIC SAMPLE PROCESSING | |
| APPENI | DIX 2 DESCRIPTION AND COMPOSITION OF TEST PRODUCT | 51 |
| APPENI | DIX 3 DIVISION OF MICROBIOLOGY AND INFECTIOUS DISEASE TOXI | CITY |
| TABLE. | | 57 |
| APPENI | DIX 4 HOLTER RECORDING AND ANALYSIS | 65 |
| APPENI | DIX 5 REPEAT COHORT USING DIFFERENT DOSAGE FORMULATION | 67 |
| <b>APPENI</b> | DIX 6 PART 2 OF THE STUDY | 68 |
| Table 1 | Comparison of Projected TBI-223 Efficacious Exposure and T>MIC at 1200 in Efficacious Exposures in Mouse Efficacy Studies | ng to the |
| T 11 0 | Efficacious Exposures in Mouse Efficacy Studies | |
| Table 2 | Actual Dose Cohorts for Part 1 | |
| Table 3 | Identity of Investigational Product | |
| Table 4 | Total Volume of Blood to be Collected for Testing: Fasting Cohorts | |
| Table 5 | Total Volume of Blood to be Collected for Testing: Food-effect Cohorts | 28 |
| Table 6 | Adverse French Attribution/Councility Potings | |
| Table 7 | Adverse Event Attribution/Causality Ratings | |
| Table 8 | | |
| Table 9 Table 10 | Schedule of Assessments, Part 1 | 43 |
| Table 10 | mg | |
| Tabla 11 | Strength, Tablet Weight and Appearance of TBI-223 IR and SR Tablets | |
| | Composition of TBI-223 IR Tablets, 600 mg and 1000 mg | |
| | Composition of TBI-223 R Tablets, 600 mg (Prototype 1) | |
| | Composition of TBI-223 SR Tablets, 600 mg (Prototype 1) | |
| | Composition of TBI-223 SR Tablets, 900 mg (Prototype 3) | |
| | Schedule of Assessments. Part 2 | |

# LIST OF FIGURES

| Figure 1 | Dosing Groups | 10 |
|----------|---------------|----|
|----------|---------------|----|

#### LIST OF ABBREVIATIONS

AE adverse event

ALP alkaline phosphatase ALT alanine transaminase ANOVA analysis of variance AST aspartate transaminase

AUC area under the (plasma concentration vs. time) curve

AUC<sub>last</sub> area under the curve from time 0 hours to last quantifiable concentration

AUC<sub>inf</sub> area under the curve from time 0 hours to infinity

BID twice daily
BMI body mass index
BP blood pressure
BUN blood urea nitrogen
bpm beats per minute

Ca calcium

CFR Code of Federal Regulations

CFU colony-forming unit CI confidence interval

Cl<sup>-</sup> chloride

C<sub>last</sub> last quantifiable drug concentration

CLIA Clinical Laboratory Improvement Amendments

cm centimeter(s)

C<sub>max</sub> maximum concentration CNS central nervous system

CRF case report form CYP cytochrome P450

DMID Division of Microbiology and Infectious Disease

ECG electrocardiogram

FDA Food and Drug Administration FSH follicle-stimulating hormone

g gram(s)

GCP Good Clinical Practice GGT gamma-glutamyl transferase

HIPAA Health Insurance Portability and Accountability Act

GLP Good Laboratory Practice
HIV human immunodeficiency virus
ICD informed consent document

ICH International Council for Harmonisation of Technical Requirements for

Pharmaceuticals for Human Use

INDInvestigational New DrugIPInvestigational ProductIRBinstitutional review boardISFInvestigator Site FileIUDintrauterine device

K<sup>+</sup> potassium kg kilogram(s)

K<sub>3</sub>-EDTA ethylenediaminetetraacetic acid

L liter(s) lbs pounds

LDH lactate dehydrogenase

m meter(s)

MAO monoamine oxidase

max. maximum

MDR-TB multidrug resistant tuberculosis

mg milligram(s)

MICs minimum inhibitory concentrations

min. minute(s) mL milliliter(s)

mmHg millimeter of mercury

MPS mitochondrial protein synthesis

msec millisecond

Mtb Mycobacterium tuberculosis

Na<sup>+</sup> sodium

NOAEL no-observed-adverse-effect level

OTC over-the-counter

oz ounce(s)

PK pharmacokinetic PT prothrombin time rbc red blood cell

SAD Single Ascending Dose SAE serious adverse event SAP statistical analysis plan

T<sub>1/2</sub> or t<sub>1/2</sub> terminal elimination half-life

TB Tuberculosis

T<sub>last</sub> time of the last measurable concentration

 $T_{\text{max}}$  time to reach  $C_{\text{max}}$ 

Worldwide Worldwide Clinical Trials Early Phase Services, LLC

Worldwide Clinical Trials Early Phase Services/Bioanalytical Sciences, LLC

 $\lambda_z$  apparent elimination rate constant in terminal phase

°C degrees Celsius/Centigrade

#### 1 INTRODUCTION

## 1.1 Background Information

This study will be conducted in accordance with the protocol, International Good Clinical Practice (GCP) Guidelines, the ethical principles that have their origin in the Declaration of Helsinki and the applicable regulatory requirement(s).

A brief overview of available confidential information regarding TBI-223 follows below. Unless noted otherwise, the information in this introduction was provided by TB Alliance.

#### 1.2 Tuberculosis and Rationale for New Medications

Tuberculosis (TB) in humans is an infectious disease caused by the bacterium *Mycobacterium tuberculosis* (Mtb), which typically affects the lungs (pulmonary TB) but can affect other sites as well (extrapulmonary TB). While incidence rates and mortality for TB have been falling, it remains the ninth leading cause of death worldwide, the world's leading cause of death from a single infectious disease and is responsible for more deaths than human immunodeficiency virus (HIV). In 2016, 6.3 million new cases of TB were reported, with an overall estimated incidence of 10.4 million (World Health Organization [WHO] Global TB Report 2017).

The current TB treatment regimens and treatments for drug-sensitive TB are decades old and are relatively ineffective. The available treatments have a lengthy duration of treatment, can involve multi-drug therapy, many tolerability issues, and require large commitments of resources and infrastructure. High rates of noncompliance are common, which often results in increased mortality, chronic, infectious, and drug-resistant cases. The present TB epidemic and treatment conditions demonstrate the clear need in patients with drug-sensitive or drug-resistant TB for novel drugs and drug regimens that will shorten the current treatment duration and be safe and well tolerated. In addition, new TB drugs and regimens should also be affordable, easy to adopt and implement, suitable for pediatric use and for co-administration with antiretroviral therapy in individuals co-infected with Mtb and HIV. Following the declaration of TB as a global emergency by the WHO in 1993, there has been a resurgence of efforts to develop improved TB therapies and several promising new agents are presently in or approaching clinical evaluation.

TBI-223 like linezolid (Zyvox®), is a novel oxazolidinone antimicrobial that inhibits the growth of Mtb by blocking microbial translation and, thereby, protein synthesis. Linezolid, which is licensed for the treatment of complicated skin infections and hospital-acquired pneumonia (at an adult dose of 600 mg given twice daily [BID] for up to 28 days), has been used to treat difficult cases of multiple drug-resistant and extensively drug-resistant TB with apparent clinical benefit. Since bacterial protein

synthesis is not currently targeted by any of the drugs in the first-line standard of care for treatment of TB (isoniazid, rifampin, pyrazinamide, ethambutol), TBI-223, like linezolid, has no known pre-existing resistance. Therefore, TBI-223 should be effective against multi-drug resistant and extensively drug-resistant forms of TB (MDR-TB and XDR-TB) as well.

The standard dose of linezolid for a multitude of indications is 400 mg or 600 mg BID. Doses of linezolid varying from 300 mg to 1200 mg per day were used to treat pulmonary TB in combination with other TB drugs in novel regimes over periods of up to 20 months with impressive improved outcomes - e.g. in the Nix-TB trial (A Phase 3 Study Assessing the Safety and Efficacy of Bedaquiline Plus PA-824 (Pretomanid) Plus Linezolid in Subjects with Drug Resistant Pulmonary Tuberculosis: NCT02333799), but treatments can be impacted with periods of non-compliance and adverse events (AEs), especially neuropathic and myelosuppressive effects. These AEs are often ameliorated if the dose is reduced or if the drug is discontinued for several weeks and then resumed at a lower dose. Although manageable there is a clear need to develop effective and tolerable oxazolidinones with a better toxicology profile.

TBI-223 is a preclinical drug candidate from TB Alliance's efforts to develop a safer oxazolidinone with the potential to deliver efficacy similar to linezolid, without the characteristic bone marrow and neuropathic toxicities of the class. It emerged from a scaffold expansion effort based on the linezolid and sutezolid structures. Mammalian mitochondrial protein synthesis (MPS) inhibition is presumed to be the reason for the side effects associated with long-term administration of linezolid, such as anemia, thrombocytopenia, and peripheral neuropathy (Migliori et al., 2009). TBI-223 was tested in an MPS inhibition assay and found to have a half maximal inhibitory concentration (IC50) of 126  $\mu$ M (46  $\mu$ g/mL). This concentration exceeds the expected maximum clinical TBI-223 concentration by 2-fold and suggests a lower risk of MPS inhibition. In preclinical studies, TBI-223 showed low minimum inhibitory concentrations (MICs) against Mtb in vitro and efficacy against mouse models of TB as a single agent and in combination with bedaquiline and pretomanid. TBI-223 did not show significant myelosuppression in 28-day Good Laboratory Practice (GLP) toxicity studies in rats and dogs.

Current data suggest that TBI-223 could contribute to a new TB treatment, consistent with the high-priority target product profile for a novel and universal TB drug regimen. A comprehensive nonclinical pharmacology, pharmacokinetic, toxicology, and safety program have been completed to support the Investigational New Drug Application and clinical development of TBI-223. The first clinical trial will be a randomized, Single Ascending Dose Study with a Food Effect Cohort. The objectives are to evaluate the safety, tolerability, and pharmacokinetics, and to explore the potential maximum tolerable dose of TBI-223 in healthy men and women.

# 1.3 Preclinical Studies and Toxicity Studies

To support Investigational New Drug (IND) filing, a nonclinical development plan has been executed based upon the ICH M3(R2) guidance document, "Nonclinical Safety Studies for the Conduct of Human Clinical Trials and Marketing Authorization for Pharmaceuticals," January 2010.

A series of in vitro and in vivo studies to evaluate the efficacy of TBI-223 were carried out. TBI-223 was evaluated against a large, diverse panel of Mtb clinical isolates, consisting of 96 isolates representative of all identified genetic groups of Mtb, broad geography and diverse drug-susceptibility profiles. The panel included MDR-TB and XDR-TB strains. The MIC of TBI-223 was found to be 1.28 μg/mL for 90% of the strains tested with a range of 0.04 to 5. Like linezolid, TBI-223 demonstrated a mild bactericidal activity against acute mouse infections of TB as a single agent, good activity against chronic mouse infections, including additive activity within the Nix-like drug combination of bedaquiline, an ATP synthase inhibitor, and pretomanid, a nitroimidazole. This combination efficacy demonstrated a strong potential for TBI-223 to replace linezolid in the Nix trial regimen and deliver a universal treatment shortening regimen that is not confined to the XDR-TB population.

A comprehensive battery of in vitro and in vivo safety pharmacology assessments was conducted to characterize the effects of TBI-223 on the function of the nervous, respiratory, and cardiovascular systems. The battery included non-GLP studies of several cardiac ion channels with TBI-223, a GLP human Ether-à-go-go-Related Gene (hERG) assay with TBI-223, a standalone GLP single-dose cardiovascular study. Nervous system and respiratory assessments were conducted in rats administered as single doses of TBI-223.

The pharmacokinetics and oral bioavailability of TBI-223 were evaluated in mice, rats, dogs and monkeys given single or repeated daily doses of TBI-223.

In support of planned human studies, the following toxicology studies have been completed with TBI-223:

- Non-GLP, 4-week, repeat-dose, oral toxicity study in mice.
- Non-GLP, 2- and 4-week, repeat-dose, oral toxicity studies in rats.
- GLP-compliant, 4-week, repeat-dose, oral toxicity study with recovery in rats.
- Non-GLP, 5-day and 2-week, repeat-dose, oral toxicity studies in beagle dogs.
- GLP-compliant, 4-week, repeat-dose, oral toxicity study with recovery in beagle dogs.
- Standard battery of GLP-compliant in vitro and in vivo genetic toxicology studies.

Dogs tolerated doses up to 100 mg/kg/day (50 mg/kg BID) for 28 days but showed dose- and duration-related nervous system effects at repeated doses  $\geq$ 200 mg/kg/day. There were no correlating histopathology findings in the nervous system in these studies. It is unclear whether the nervous system effects are related to the maximum concentration ( $C_{max}$ ) or the area under the (plasma concentration vs. time) curve (AUC) of TBI-223.

- In a 5-day study, dogs developed prolonged tremors and 2 of 4 dogs were found dead after being given 400 mg/kg/day for 3 days. These dogs had previously been administered 200 mg/kg/day of TBI-223 without clinical signs.
- During the first 4 days of dosing of a 14-day DRF study, tremors and emesis were observed in dogs administered 200 mg/kg/day, and ataxia, prostration, and convulsions were observed in dogs administered 400 mg/kg/day. These dogs were given a 2-day washout period and then dosed at 75 mg/kg/day BID or 150 mg/kg daily (QD). Reversible tremors were observed after 8 to 10 days of dosing at 150 mg/kg/day (QD or 75 mg/kg BID). In the pivotal 28-day dog GLP study, 2 dogs given 200 mg/kg/day (100 mg/kg BID) had continuous tremors after 12 days of dosing.

In electrocardiogram (ECG) evaluation during the pivotal 28-day dog toxicity study, QT prolongation was observed. The findings are detailed below and correlated with similar findings in the GLP cardiovascular safety study in dogs, and likely related to inhibition of the hERG channel observed in the GLP hERG study.

• In dogs administered 200 mg/kg/day (100 mg/kg BID) doses of TBI-223, QT prolongation was observed in the GLP repeat dose toxicology study. The mean QTc interval at 2 to 4 hours post the first daily dose on Day 25 of the dosing phase was longer in males by 23 msec (10%) and in females by 27 msec (11%) administered 200 mg/kg/day compared with the respective controls. Mean uncorrected QT interval was also prolonged (up to 42 msec; 22%). The QT and QTc intervals returned to baseline during the recovery phase.

In addition to the above adverse effects, rats had nonadverse abdominal distension reported in repeat dose studies with TBI-223, which was associated with food-filled stomach in rats even though they were fasted overnight prior to necropsy.

# 1.4 Adverse Effects, Warnings, and Precautions

TBI-223 has not been tested in humans, therefore its potential adverse effects are unknown. The following adverse reactions were noted in more than 1% of adult subjects in a study of different drug in the oxazolidinone class, linezolid (marketed as Zyvox®): headache, diarrhea, nausea, vomiting, dizziness, rash, anemia, taste alteration, vaginal and oral candidiasis, abnormal liver functions tests, fungal infection, tongue discoloration, and abdominal pain.¹

The Zyvox<sup>®</sup> label carries warnings and precautions for myelosuppression, peripheral and optic neuropathy, serotonin syndrome, *Clostridium difficile* associated diarrhea, elevated blood pressure in patients with hypertension, lactic acidosis, convulsions, hypoglycemia, and development of drug-resistant bacteria. <sup>1</sup>

Given the key safety findings in the nonclinical safety studies for the cardiovascular system (prolonged QTc) and the nervous (CNS) system (tremors), we will implement the following monitoring procedures.

## **Cardiovascular Monitoring**

Cardiovascular monitoring will be conducted and include the following at both protocol-defined time points and whenever deemed necessary by the study investigator. Subjects treated with TBI-223 will have their ECGs evaluated prior to treatment and during treatment. During treatment, the timing of ECGs will be guided by pharmacokinetic (PK) data so that collection occurs around the estimated T<sub>max</sub>.

ECGs will be interpreted and signed and dated by the Principal Investigator or designee. The ECGs will be classified as normal, having a clinically insignificant abnormality, or having a clinically significant abnormality. All clinically significant abnormalities will be recorded as AEs. In addition, ECG parameters of ventricular rate, PQ or PR interval, QRS duration, and QT interval (corrected and uncorrected) will be noted on the case report form (CRF). If a patient's corrected QT interval (QTcF) exceeds 500 msec while on treatment or there is a change from baseline exceeding 60 msec, TBI-223 administration should be stopped, and the patient monitored with ECGs and/or telemetry until the QTcF returns to pre-treatment levels. Study subjects will also be monitored with Holter monitoring. Holter monitoring will begin approximately 24 hours prior to and continue until 48 hours after dosing.

### **Central Nervous System Monitoring**

A detailed neurological exam will be conducted and include the following at both protocol-defined time points and whenever deemed necessary by the study investigator:

- Mental status assessment of orientation, speech, and memory
- Cranial nerves assessment of cranial nerves II-XII, excluding fundoscopic examination
- Motor system brief assessment of tone and strength
- Sensory system brief survey for light touch and temperature of the face, neck, arms, trunk, and legs
- Reflexes assessment of deep tendon reflexes and plantar responses (Babinski sign)

- Coordination assessment of upper and lower extremities, including assessment for tremor
- Gait assessment of tandem gait

### 1.5 Overview and Dose Rationale

A two-compartment PK model with non-linear clearance was built to project TBI-223 human PK parameters from animal PK parameters.

The projected human efficacious doses range from 800 to 1200 mg, with a predicted  $C_{max}$  of 15.7-24.9  $\mu$ g/mL and predicted (AUC<sub>0-24hr</sub>) of 101 to 202  $\mu$ g.hr/mL.

TBI-223, as a single agent at 100 mg/kg, demonstrated moderate activity against acute murine TB in BALB/c mice, and in a C3HeB/FeJ mouse model of TB. When combined with the TB drug bedaquiline and the investigational TB drug pretomanid, TBI-223 at 100 mg/kg demonstrated bactericidal and sterilizing activity against murine TB in BALB/c mice that was similar to that of linezolid at the same dose (100 mg/kg). The PK exposure at 100 mg/kg was 179 μg•hr/mL, with T>MIC at 61% (or 14.6 hr/day) in the female BALB/c mice.

A dose fractionation study of TBI-223 in a BALB/c mouse model of TB showed that the efficacy drivers were AUC ( $R^2 = 0.92$ ) and T>MIC ( $R^2 = 0.83$ ). The study indicated that a 2 Log lung colony-forming unit (CFU) reduction can be achieved with total a weekly AUC of 868 µg.hr/mL, or daily AUC<sub>0-24hr</sub> of 124 µg.hr/mL, with T>MIC of 34% (T>MIC at 8.2 hours over 24 hours).

Comparing to the projected human exposure at 1200 mg based on nonlinear two-compartment model, the human AUC<sub>0-24hr</sub> (205.2  $\mu$ g.hr/mL) is 1.7-fold the mouse efficacious exposure (124  $\mu$ g.hr/mL) for a 2 Log CFU reduction (Table 1). The AUC<sub>0-24hr</sub> at 202  $\mu$ g.hr/mL could result in 2.8 Log CFU reduction. The predicted T>MIC at 1200 mg was 62.9% which is 1.8-fold the mouse efficacious T>MIC (34%) for 2 Log CFU reduction. At T>MIC of 62.9%, the calculated Log CFU reduction would be 3.4 based on the dose fraction study.

Comparing to linezolid clinical efficacious doses at 600 mg and 1200 mg daily dose, the projected TBI-223 exposure  $AUC_{0-24hr}$  at 1200 mg is 2-fold that of linezolid exposure at 600 mg daily dose and 0.7-fold of linezolid exposure at 1200 mg daily dose.

Table 1 Comparison of Projected TBI-223 Efficacious Exposure and T>MIC at 1200 mg

to the Efficacious Exposures in Mouse Efficacy Studies

| | Dose or Log CFU reduction | AUC <sub>0-24hr</sub><br>(μg.hr/mL) | T>MIC<br>(%) |
|---|---|---|---|
| TBI-223 Projected human efficacy dose | 1200 mg QD | 202 | 62.5 |
| TBI-223 Mouse efficacy studies | 100 mg/kg | 179 | 61 |
| EDI AAA D | 2 Log CFU reduction | 124 | 34 |
| TBI-223 Dose fraction study | AUC for 2.8 Log CFU reduction, or T>MIC for 3.7 Log CFU reduction | 202 | 62.5 |
| Linezolid efficacious | 600 mg, human | 104 | 91 |
| dose | 1200 mg, human | 300 | 100 |

## Starting dose for the SAD

A single dose of 50 mg appears to be an appropriate starting dose for the single ascending dose SAD study for the following reasons:

- The proposed 33-fold safety margin to the human equivalent dose (HED) derived from the no-observed-adverse-effect level (NOAEL, 100 mg/kg) in the 28-day dog toxicology study is based on twice daily dosing (50 mg/kg BID) compared to once daily dosing proposed in humans. The daily dosing frequency was changed from QD to BID in the animal studies to increase tolerability of TBI-223 when orally administered to dogs.
- The more relevant NOAEL at 50 mg/kg QD (HED 27 mg/kg) in the repeat-dose 28-day dog toxicology study provides a 17-fold safety margin to a first-in-human (FIH) starting dose of 100 mg QD. However, in the nonclinical safety pharmacology cardiovascular study in dogs, a trend of increasing QTc prolongation was observed in dogs after a single oral administration of TBI-223 at 50 and 100 mg/kg (max increase 11 to14 msec from baseline, 12 msec from control 2 hours post-dose) at 1 to 13 hours post-dose, and a statistically significant increase in QTc interval was detected at 200 mg/kg (mean increase 22 msec from baseline and control 2 to 5 hours post-dose, and 21 to 25 hours post-dose).
- Significant toxicity was observed in the 28-day dog toxicology study at a dose of 200 mg/kg/day (100 mg/kg BID) including intermittent and continuous tremors, ataxia, convulsions in several animals, QTc prolongation (10 to 11% baseline), decreased body weight, and vomitus. It should be noted that the dosing interval between twice daily dosing was not provided, and the clinical observations were

- performed at 1 and 12 hours post-dose, and not 2 to 4 hours at  $C_{max}/T_{max}$  when tremors may have a greatest chance of occurring and being detected.
- In the 14-day dog toxicology study with orally administered TBI-223, dose reduction from 200 mg/kg daily to 150 mg/kg (75 mg/kg BID) on Day 7 continued to cause tremors on Days 8 to 10 of dosing. This may be a result of drug accumulation noted with repeated dosing with TBI-223. Cage-side observations more appropriately timed at 3 to 4 hours post-dose and 6 to 9 hours post-dose in this 14-day study may have provided a greater opportunity of detecting tremors in animals. Had the clinical observations been performed at similar times in the 28-day dog toxicology study, perhaps tremors might have been observed at 100 mg/kg/day (50 mg/kg BID), reportedly the NOAEL in this study. No tremors were observed at 75 mg/kg/day QD in dogs in the 14-day study.

In the first cohort of this Phase 1 study, the proposed starting dose of 50 mg once daily (QD) is 66-fold lower than the HED of 3243 mg/day, derived from the lowest NOAEL, which was 50 mg/kg BID (100 mg/kg/day) in a 28-day dog GLP toxicity study. The proposed starting dose is 17-fold less than the HED of a single 50 mg/kg dose in dogs.

The predicted  $C_{max}$  and  $AUC_{0-24hr}$  at the proposed first in human dose of 50 mg once daily are 0.711 µg/mL and 2.5 µg.hr/mL, which are 20.4- and 86-fold less than the NOAEL in the dog toxicity study, respectively. The proposed starting doses for this first-in-human SAD study are well below the predicted NOAEL. The following dose escalations for each cohort receiving a single dose are proposed: 50 mg, 100 mg, 300 mg, 600 mg, 1200 mg, and 2000 mg. These proposed doses (cohorts) could change (e.g. if bioavailability is lower than expected or for potential emerging safety reasons).

For all the reasons noted above, a starting dose of 50 mg in the SAD would likely provide a reasonable margin of safety to any adverse -cardiovascular or CNS- effects observed with TBI-223 during administration to dogs.

Dose escalation will be guided by emerging safety and pharmacokinetic data so that predicted median  $C_{max}$  of a cohort can exceed 20.2  $\mu$ g/mL (the NOAEL plasma  $C_{max}$  in the 28-day GLP dog toxicity study) only if, after data review, the prior dose was considered safe and well tolerated. Human plasma M2 metabolite exposure will be measured at each dose level, and the M2 exposure for next dose level will be predicted for safety analysis by comparing to M2 exposures in dogs. However, the planned doses could change if the generated bioavailability is lower than expected. Therefore, additional cohorts may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study other dose levels or a different dosage formulation. These decisions regarding planned additional cohorts will not take place until the Sponsor, in conjunction with the Principal Investigator and dose-escalating committee, has

determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort have been demonstrated to permit proceeding to the next cohort. The Institutional Review Board (IRB) should be immediately notified of this revised approach for review and approval. The new approved dose for Cohort 6 will be 2000 mg.

#### 2 OBJECTIVE

The primary objective of the study is:

 To evaluate the safety and tolerability of single doses of TBI-223 oral suspension, TBI-223 oral enteric capsules, and TBI-223 tablet formulations in healthy adult subjects.

The secondary objectives of the study are:

- To determine the pharmacokinetics of TBI-223 and its metabolite M2 after single doses of TBI-223 oral suspension, TBI-223 oral enteric capsules, and TBI-223 tablet formulations in healthy adult subjects; and
- To compare the rate and extent of absorption of a single dose of TBI-223 oral suspension, TBI-223 oral enteric capsules, and TBI-223 tablet formulations when administered in healthy adult subjects either after a high-calorie, high-fat meal or in the fasting state.

#### 3 STUDY DESIGN SUMMARY

#### Part 1:

Up to 48 subjects in 6 dosing cohorts are planned to be enrolled; within each cohort, 6 subjects will be assigned to active treatment and 2 to placebo.

Each subject will participate in 1 dose level. Based on interim pharmacokinetic data obtained during the dose escalation, a dose cohort will be selected to return for additional dosing after a high-calorie, high-fat meal (food-effect cohort).

Each cohort will be dosed in 2 groups in order to monitor subjects for adverse experiences, in particular, convulsions (in the dog toxicity studies, tremors were observed at  $C_{max}$  or plasma concentration of  $\geq 82 \mu g/mL$ , and convulsions were observed at plasma concentration or  $C_{max}$  of  $\geq 158 \mu g/mL$ ).

In the first cohort, a sentinel group of 3 subjects (2 active and 1 placebo) will be dosed at least 24 hours before the remaining 5 subjects (4 active and 1 placebo).

The remaining cohorts will be dosed in 2 groups of 4 subjects each (3 active and 1 placebo), at least 24 hours apart.

Safety will be assessed throughout the study for all subjects. Safety assessments will include physical and neurological examinations, vital signs, ECGs, cardiac monitoring, AEs, and clinical laboratory tests (including hematology, serum chemistry, coagulation, and urinalysis).

Blood and urine will be collected for clinical laboratory evaluations.

Female subjects will have blood collected for serum pregnancy testing. Postmenopausal females will have blood collected to measure follicle-stimulating hormone (FSH) levels.

Blood will be collected for pharmacokinetic analysis.

Dose escalation to the next cohort (i.e., dose level) will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability and pharmacokinetic data from the previous cohorts have been demonstrated to permit proceeding to the next cohort.

The Principal Investigator, in conjunction with the Sponsor may collect additional blood if necessary, for repeat laboratory or safety evaluations including AE follow up.

An overview of the dosing groups in Part 1 is presented in Figure 1.

SAD (Single Ascending Dose) 24 h apart Day 1 Day 2 (group 1) (group 2) Cohort 1 (Sentinel group) n=5 n=3 Cohort 2 n=4 n=4 Cohort 3 n=4 n=4 Cohort 4 n=4n=4 Cohort 5 n=4n=4Cohort Etc. n=4n=4

Figure 1 Dosing Groups

Based on the interim pharmacokinetics for the dose escalation decisions, 10 subjects will be selected to participate in the **food-effect cohort**. These subjects will receive TBI-223 or placebo under fasting conditions in the first study period. They will return after a washout of at least 7 days or 5 half-lives (whichever is longer) of their fasting dose to receive the same dose under fed conditions.<sup>3</sup>

Additional cohorts (8 subjects per cohort) may be enrolled if it is deemed appropriate by the Sponsor to repeat a dose level or to study another dose level or dosage formulation. The IRB will notified of this revised approach.

Note: In the event that a dose level is repeated to study a different dosage formulation, procedures and analyses will be conducted as outlined in Appendix 5.

Interim pharmacokinetic analyses will be performed for the dose escalation decisions, to select the dose for the food-effect cohort, and to reconsider the timing, reducing, or adding of sampling time points as the study progresses.

Blood samples will be obtained prior to study drug administration on Day 1 and at serial timepoints through 72 hours after study drug administration. Plasma pharmacokinetic samples will be analyzed for TBI-223 and M2 using validated analytical methods. Appropriate pharmacokinetic parameters will be calculated for each formulation using non-compartmental methods.

An unblinded pharmacist will be responsible for dispensing the study treatment and to ensure that study personnel are blinded.

Except for during the fed period of the food-effect cohort, TBI-223 or matching placebo dose will be administered orally with 200 mL of water after a minimum 10-hour overnight fasting, and food will be given approximately 4 hours after each dose level.

Table 2 presents the actual dose cohorts for Part 1 of the study.

**Table 2** Actual Dose Cohorts for Part 1

| Cohort <sup>a</sup> (Group <sup>b</sup> ) | Dose <sup>c</sup> | |
|---|---|---|
| 1 (sentinel group) | Single dose of 50 mg TBI-223 (n=2) | Placebo (n=1) |
| 1 (remainder of cohort) | Single dose of 50 mg TBI-223 (n=4) | Placebo (n=1) |
| 2 (Group 1) | Single dose of 100 mg TBI-223 (n=3) | Placebo (n=1) |
| 2 (Group 2) | Single dose of 100 mg TBI-223 (n=3) | Placebo (n=1) |
| 3a (Group 1) | Single dose of 300 mg TBI-223 (n=3) | Placebo (n=1) |
| 3a(Group 2) | Single dose of 300 mg TBI-223 (n=3) | Placebo (n=1) |
| 3b (Capsule cohort) | Single dose of 300 mg (TBI-223 in oral enteric capsules) (n=4) | N/A |
| 4 (Group 1) | Single dose of 600 mg TBI-223 (n=3) | Placebo (n=1) |
| 4 (Group 2) | Single dose of 600 mg TBI-223 (n=3) | Placebo (n=1) |
| 5 (Group 1) | Single dose of 1200 mg TBI-223 (n=3) | Placebo (n=1) |
| 5 (Group 2) | Single dose of 1200 mg TBI-223 (n=3) | Placebo (n=1) |
| 6 (Group 1) | Single dose of 2000 mg TBI-223 (n=3) | Placebo (n=1) |
| 6 (Group 2) | Single dose of 2000 mg TBI-223 (n=3) | Placebo (n=1) |
| 7 (Group 1) | Single dose of 2600 mg TBI-223 (n=3) | Placebo (n=1) |
| 7 (Group 2) | Single dose of 2600 mg TBI-223 (n=3) | Placebo (n=1) |

mg = milligram; n = number of subjects.

- b) Dosing between Groups 1 and 2 to occur at least 24 hours apart.
- c) Subjects will be dosed under fasted conditions. One of the dose cohorts will be selected to return for an additional dose under fed conditions.

#### Part 2:

Cohort 8: A minimum of 24 subjects in 4 dosing arms are planned to be enrolled; within each arm, 6 subjects will be assigned to receive a single dose treatment. Subjects will be assigned to one of the following arms and dose:

- Arm 1 TBI-223 SR Tablets (Prototype 1) 1800 mg dose (3 x 600 mg tablets), under fed conditions
- Arm 2 TBI-223 SR Tablets (Prototype 2) -1800 mg dose (3 x 600 mg tablets), under fed conditions
- Arm 3 TBI-223 SR Tablets (Prototype 3) 1800 mg dose (2 x 900 mg tablets), under fed conditions
- Arm 4 TBI-223 IR Tablets 2000 mg dose (2 x 1000 mg tablets), under fasting conditions

a) Additional cohorts may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level or another dosage formulation.

Procedures and analyses will be conducted as outlined in Appendix 6.

Cohort 9: The 6 subjects from Cohort 8, Arm 4, who received the IR tablet formulation fasted will return after a 7-day washout and receive a single dose of TBI-223 IR Tablets, 2000 mg dose (2 x 1000 mg tablets), under fed conditions.

If more than 2 subjects of these 6 subjects from Cohort 8 drop-out, they will be replaced by heathy volunteers (a minimum of 4 subjects are needed to complete Cohort 9).

Procedures and analyses will be conducted as outlined in Appendix 6.

#### 3.1 Part 1 Dose Escalation

Each of the fasting cohorts will be dosed in 2 groups. The first cohort will start with a sentinel group. The decisions on continuing of dosing Group 2 (at least 24 hours after dosing of Group 1) will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined adequate safety and tolerability.

#### Dose Escalation Review

A review period will take place after the dosing of all subjects in each cohort in order to evaluate and interpret all pharmacokinetic and safety data collected.

The review of all pertinent safety/tolerability data will include physical and neurological examinations, ECGs, vital signs, clinical laboratory tests, cardiac monitoring, and AEs or serious adverse events (SAEs) through Day 4. Also, data from the current dose cohort and all previous cohorts will be considered.

The Sponsor and Investigator will determine if there are sufficient data available from all subjects to make a dose escalation decision. Any AEs of grade ≥2 toxicities (per Division of Microbiology and Infectious Disease [DMID] toxicity table; Appendix 3) must be considered in the decision to escalate to the next dose level. ECG data will be analyzed in a blinded fashion and unblinded by ECG vendor in order to be presented by treatment group in aggregate (reviewers will not be unblinded by subject). Pharmacokinetic analysis will be completed only on the active treatment subjects and will be blinded to subject. Blinding will also extend to others who are intimately involved with the study except for the designated unblinded pharmacy staff and in cases of medical emergencies.

Upon review of relevant cohort data, the Sponsor, in conjunction with the Investigator may decide to:

- 1: Escalate the dose as planned
- 2: If concerns arise from pharmacokinetic and safety data that do not warrant ceasing escalation:
  - a: evaluate an intermediate dose level prior to the next planned dose level;

OR

- b: repeat a given dose level in a new cohort of subjects
- c: Repeat a dose level using a different dosage formulation.
- 3. Add a cohort or increase the dose of the next cohort if the bioavailability is lower than expected in the previous cohort and there were no safety concerns.
- 4. Halt the study.

The next dose in the escalating phase of the SAD study will be guided by emerging safety and PK data. After each cohort, Bayesian linear models will be fitted to the data from all available cohorts with log-transformed  $C_{max}$  as the response variable and log-transformed dose as the predictor variable. Different prior distributions on the coefficient of log-transformed dose, representing different assumptions about dose proportionality, will be considered. Predictive distributions will be generated for  $C_{max}$  at doses to be considered for the next level of escalation. These predictive distributions, together with emerging safety data, will be assessed by the clinical team to reach a decision on the next dose. Key features of the predictive distributions to be evaluated are the median  $C_{max}$  and the number of subjects out of those receiving TBI-223 in the next cohort expected to have  $C_{max}$  exceed 20.2  $\mu g/mL$ . (the NOAEL plasma  $C_{max}$  in the 28-day GLP dog toxicity study).

## 3.2 Stopping Rules for Cohorts

If any of the cohort stopping rules are met, cohort dosing must be stopped until review of the data by the Sponsor and the Investigator.

Rules for stopping dosing of a cohort include the following:

- 1. Two or more subjects experience drug-related SAEs;
- 2. Two or more subjects experience grade 2 or higher (per DMID toxicity table; Appendix 3) central nervous system (CNS) AEs considered related to drug.
- 3. Two or more subjects develop drug-related QTcF prolongation greater than or equal to 500 msec or a change from baseline greater than 60 msec, after completing repeat testing.
- 4. Two or more subjects experience drug-related Grade 3 or Grade 4 cardiac rhythm cardiac disturbances.

#### 4 IDENTITY OF INVESTIGATIONAL PRODUCT

The Investigational Medicinal Product (IMP) will be supplied as TBI-223 25 mg/mL oral suspension or matching placebo.

Refer to Appendix 2 for details regarding the description and composition of TBI-223.

**Table 3 Identity of Investigational Product** 

| Part 1 | |
|---|---|
| Test Product: | TBI-223 oral suspension 25 mg/mL |
| | Manufactured for Global Alliance for TB Drug Development |
| Control Product: | Placebo for TBI-223 oral suspension |
| | Manufactured for Global Alliance for TB Drug Development |
| Test Product: | TBI-223 Oral Enteric Capsules, 150 mg |
| Cohort 3b | Manufactured for Global Alliance for TB Drug Development |
| Part 2 | |
| Test Products:<br>Cohort 8 | TBI-223 SR Tablets 600 mg (Prototype 1) |
| (Arms 1-4) | Manufactured for Global Alliance for TB Drug Development by Piramal Enterprise Limited |
| | TBI-223 SR Tablets 600 mg (Prototype 2) |
| | Manufactured for Global Alliance for TB Drug Development by Piramal Enterprise Limited |
| | TBI-223 SR Tablets 900 mg (Prototype 3) |
| | Manufactured for Global Alliance for TB Drug Development by Piramal Enterprise Limited |
| | TBI-223 IR Tablets 1000 mg |
| | Manufactured for Global Alliance for TB Drug Development by Piramal Enterprise Limited |
| Test Products:<br>Cohort 9 | TBI-223 IR Tablets 1000 mg |
| Colloit 9 | Manufactured for Global Alliance for TB Drug Development by Piramal Enterprise Limited |

### 5 SUBJECT SELECTION

## 5.1 Inclusion Criteria

All volunteers must satisfy the following criteria to be considered for study participation:

- 1. Understands study procedures and voluntarily provides written informed consent prior to the start of any study-specific procedures.
- 2. Is a healthy adult male or a healthy adult female, 19 to 50 years of age (inclusive) at the time of screening.

- 3. Has a body mass index (BMI)  $\geq$ 18.5 and  $\leq$ 32.0 (kg/m<sup>2</sup>) and a body weight of no less than 50.0 kg.
- 4. Is medically healthy with no clinically significant screening results, as determined by the Principal Investigator (e.g., laboratory profiles are normal up to and including Grade 1 per DMID toxicity tables; Appendix 3), medical history, vital signs, ECG, or physical/neurological examination findings. Note: If exclusionary lab criteria are met, values may be confirmed by repeat evaluation.
- 5. Has not used tobacco- or nicotine-containing products (including smoking cessation products), for a minimum of 6 months before dosing.
- 6. If female of non-childbearing potential, she has undergone one of the following sterilization procedures at least 6 months before dosing:
  - Hysteroscopic sterilization;
  - Bilateral tubal ligation or bilateral salpingectomy;
  - Hysterectomy; or
  - Bilateral oophorectomy;
  - Or is postmenopausal with amenorrhea for at least 1 year before the first dose with serum follicle-stimulating hormone (FSH) levels consistent with postmenopausal status (i.e., greater than 40 mIU/mL) at screening.

Or, if female of childbearing potential, must agree to use an allowable form of birth control from screening until 14 days after study completion. The following are allowed birth control methods for this study:

- Vasectomized partner (at least 6 months before dosing);
- Non-surgical permanent sterilization (e.g., Essure® procedure) at least 3 months before dosing;
- Double barrier method (e.g., diaphragm with spermicide; condoms with spermicide);
- Intrauterine device (IUD);
- Abstinence (and must agree to use a double barrier method if they become sexually active during the study);
- Implanted or intrauterine hormonal contraceptives in use for at least 6 consecutive months before study dosing; and/or
- Oral, patch, or injected contraceptives, or vaginal hormonal device (i.e. NuvaRing®), in use for at least 3 consecutive months before study dosing.

- 7. If a non-vasectomized male (or male vasectomized less than 120 days prior to study start) he must agree to the following during study participation and for 90 days after the last administration of study drug:
  - Use a condom with spermicide while engaging in sexual activity or be sexually abstinent
  - Not donate sperm during this time.

In the event the sexual partner is surgically sterile or postmenopausal, use of a condom with spermicide is not necessary. None of the birth control restrictions listed above are required for vasectomized males whose procedure was performed more than 120 days before study start.

- 8. Is willing to answer inclusion and exclusion criteria questionnaire at check-in.
- 9. Is able to comply with the protocol and the assessments therein, including all restrictions.
- 10. Is willing and able to remain in the study unit for the entire duration of the assigned confinement period(s), return for outpatient visit(s), and receive a phone call for follow-up questioning about AEs.
- 11. If enrolled in the food-effect cohort, is willing and able to consume the entire high-calorie, high-fat breakfast meal in the timeframe required.

### 5.2 Exclusion Criteria

Volunteers will be excluded from study participation for any of the following:

- 1. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological (including epilepsy), oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
- 2. Evidence on physical exam and targeted neurologic exam of specific findings such as resting or intention tremor, dysmetria, nystagmus or ataxia, or abnormal deep tendon reflexes (either zero or hyper-reflexia).
- 3. History of any illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk to the subject by their participation in the study.
- 4. Surgery within the past 90 days prior to dosing as determined by the Investigator to be clinically relevant, or any history of cholecystectomy.
- 5. History or presence of alcoholism or drug abuse within the past 2 years as determined by the Investigator to be clinically relevant.

- 6. History of sensitivity or contraindication to use of linezolid, sulfa drugs, or any study investigational products.
- 7. Participation in another clinical trial within 30 days prior to dosing.
- 8. Female subjects who are pregnant or lactating.
- 9. Positive result on a urine drug/alcohol/cotinine screen at Baseline or check-in.
- 10. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening. Out-of-range vital signs may be repeated once for confirmation.
- 11. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening. Out-of-range vital signs may be repeated once for confirmation.
- 12. Any clinically significant ECG abnormality at Screening (as deemed by decision of the Investigator and the Sponsor's Medical Monitor).

NOTE: The following may be considered not clinically significant without consulting the Sponsor's Medical Monitor:

- Mild first degree A-V block (P-R interval <0.23 sec)
- Right or left axis deviation
- Incomplete right bundle branch block
- Isolated left anterior fascicular block (left anterior hemiblock) in younger athletic subjects
- Early repolarization
- Tall T waves
- RSR in V1/V2 consistent with right ventricular conduction delay (with acceptable QRS)
- Sinus rhythm or sinus bradycardia with sinus arrhythmia
- Minimal or moderate voltage criteria for left ventricular hypertrophy (LVH).
- 13. QTcF interval >450 msec for males or >470 msec for females at screening, Day -1, or Day 1 (pre-dose), or history of prolonged QT syndrome. For the triplicate ECGs taken at screening and on Day -1, the average QTcF interval of the 3 ECG recordings will be used to determine qualification.
- 14. Family history of long-QT syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease, congestive heart failure, or terminal cancer).
- 15. History of 1 or any combination of, the following:

- Seizures or seizure disorders, other than childhood febrile seizures
- Brain surgery
- History of head injury in the last 5 years
- Any serious disorder of the CNS or related neurological system, particularly one that may lower the seizure threshold.
- 16. Lactose intolerant.
- 17. History or presence of allergic or adverse response to Listerine breath strips or aspartame.

### Specific Treatments

- 18. Use of any prescription medication within 14 days prior to dosing.
- 19. Use of any of the following medications within 30 days before the first dose of study drug or during the study drug treatment period: monoamine oxidase (MAO) inhibitors (phenelzine, tranylcypromine), tricyclic antidepressants (amitriptyline, nortriptyline, protriptyline, doxepin, amoxapine, etc.), antipsychotics such as chlorpromazine and buspirone, serotonin re-uptake inhibitors (fluoxetine, paroxetine, sertraline, etc.), bupropion, agents known to prolong the QTc interval (erythromycin, clarithromycin, astemizole, type Ia [quinidine, procainamide, disopyramide] and III [amiodarone, sotalol] anti-arrhythmics, carbamazepine, sulfonylureas, and meperidine).
- 20. Use of any over-the-counter (OTC) medication, including herbal products and vitamins, within 7 days prior to dosing, except acetaminophen. Up to 3 grams per day of acetaminophen is allowed at the discretion of the Investigator prior to dosing.
- 21. Use of any drugs or substances known to be significant inhibitors of cytochrome P450 (CYP) enzymes and/or significant inhibitors or substrates of P-glycoprotein (P-gp) and/or organic anion transporting polypeptides (OATP) within 14 days prior to the first dose of study drug.
- 22. Use of any drugs or substances known to be inducers of CYP enzymes and/or Pgp, including St. John's Wort, within 30 days prior to the first dose of study drug.
- 23. Use of any drugs or substance known to lower the seizure threshold.

## <u>Laboratory Abnormalities</u>

- 24. Serum magnesium, potassium, or calcium laboratory values outside of the normal range at screening. If exclusionary lab criteria are met, values may be confirmed by repeat evaluation.
- 25. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).

# 5.3 Medication and Activity Restrictions

- 1. Subject must not donate blood from 56 days or plasma from 7 days prior to the first dose of study medication until after the follow-up phone call. It is recommended that blood/plasma donations not be made for at least 30 days after discharge from the clinic.
- 2. Subject must not use tobacco- or nicotine-containing products (including smoking cessation products) from 6 months prior to the first dose of study medication until after the follow-up phone call.
- 3. Subjects must not consume alcohol from 72 hours prior to the first dose of study medication until after discharge from the clinic.
- 4. Subject must not consume beverages or foods that contain grapefruit or Mandarin oranges from 10 days before the first dose of study medication, or poppy seeds, broccoli, Brussels sprouts, pomegranate, star fruit, char-grilled meat, or caffeine/xanthine from 48 hours before the first dose of study medication, until after discharge from the clinic. Subjects will be instructed not to consume any of the above products; however, allowance for an isolated single incidental consumption may be evaluated and approved by the study Investigator based on the potential for interaction with the study drug.
- 5. Subject should avoid large quantities of foods or beverages with high tyramine content 48 hours prior to the first dose of study medication until discharge from the clinic. Quantities of tyramine consumed should be less than 100 mg per meal. Foods high in tyramine content include those that may have undergone protein changes by aging, fermentation, pickling, or smoking to improve flavor, such as aged cheeses (0 to 15 mg tyramine per ounce); fermented or air-dried meats (0.1 to 8 mg tyramine per ounce); sauerkraut (8 mg tyramine per 8 ounces); and soy sauce (5 mg tyramine per 1 teaspoon). The tyramine content of any protein-rich food may be increased if stored for long periods or improperly refrigerated.
- 6. Subject must not engage in strenuous exercise from 48 hours prior to the first dose of study medication until after discharge from the clinic.

- 7. Subject must be willing to remove any artificial nails (e.g., acrylic, gel) or fingernail polish and not use such products for the duration of the study.
- 8. Subject must not take any adrenergic/serotonergic agonists, such as pseudoephedrine and phenylpropanolamine (frequently found in cold and cough remedies), within 7 days before the first dose of study drug or during the study drug treatment period.

## 5.4 Screening

The informed consent documents (ICDs) will be discussed with each potential participant, and each individual will sign an ICD for the study prior to any study-specific procedures being performed.

Each potential study participant will have the following assessments by the Investigator or designee within 28 days prior to study start:

- Demographic data, including sex, age, race, ethnicity, body weight (kg), height (cm), BMI (kg/m²), and smoking habits.
- Medical history
- Serology tests for HIV, hepatitis B and C
- Clinical laboratory tests (hematology, coagulation, chemistry, and urinalysis)
- Serum pregnancy (all female subjects)
- FSH test (female subjects claiming post-menopausal status)
- Urine test for drugs of abuse, alcohol, and cotinine
- Physical and neurological examinations
- Triplicate 12-lead safety ECGs
- Vital signs (blood pressure, pulse rate, respiration rate, temperature, and pulse oximetry)
- Concomitant medication review

Only medically healthy subjects with clinically acceptable laboratory profiles and ECGs within the defined parameters who fulfill all other inclusion criteria and meet none of the exclusion criteria outlined in the previous sections will be enrolled in the study.

Subjects will be assigned numbers in an ascending order, based on successful completion of the screening process.

#### 6 STUDY PROCEDURES

#### 6.1 Subject Assignment

For Part 1, up to 50 subjects are planned to be enrolled in the study. Additional subjects may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level. For Part 2, Cohort 8, 24 subjects will be enrolled. For Part 2,

Cohort 9, the 6 subjects from Cohort 8 who received the IR tablet formulation fasted will return after a 7-day washout and receive the IR tablet formulation under fed conditions. If more than 2 subjects of these 6 subjects from Cohort 8 drop-out, they will be replaced by heathy volunteers (a minimum of 4 subjects are needed to complete Cohort 9).

The number of subjects selected for the study was based on the adequate number considered to provide sufficient safety data. This study has not been formally powered.

For Part 1, each subject will receive an assigned treatment (active or placebo) based on the randomization schedule prepared by the unblinded statistician. The unblinded pharmacy staff will ensure compliance with the randomization schedule.

Note: the repeat cohort using a different dosage formulation in Part 1 and subjects in Part 2 will be non-randomized and unblinded; see Appendix 5 and Appendix 6.

## 6.2 Blinding

All subjects and clinical staff (except for the unblinded pharmacy staff) will be blinded to treatment. An unblinded pharmacy staff will be required at the Clinical Site to comply with the study's randomization and blinding requirements. At the Clinical Site, prior to study initiation, the Principal Investigator will be responsible for designating a qualified pharmacy staff to serve as the unblinded pharmacy staff in the study. Unblinded pharmacy staff may dose subjects but may not participate in any subject assessments.

Throughout the study, the designated unblinded pharmacy staff will be responsible for all drug accountability issues, including preparing, labeling, dispensing, and dosing study drug according to the randomization code provided, yet remain independent of all subject assessments. The pharmacy staff will follow the Standard Operating Procedures and Work Instructions related to pharmacy services and protocol-specific requirements.

Randomization codes will be provided to the unblinded pharmacy staff. Confirmation of receipt of the randomization code will be required by the Sponsor. The unblinded pharmacy staff will be responsible for maintaining the blind, consistent with protocol design, throughout the study. All documentation is to be filed in the Pharmacy Manual. Access to this manual by study personnel will be restricted to the unblinded pharmacy staff.

The subjects, Principal Investigator, and all other study personnel involved with subject assessments will remain blinded to the actual treatment assignments of the subjects. The Principal Investigator will be ultimately responsible for ensuring that the integrity of the blind is maintained throughout the study and will be required to notify the Sponsor in the event of any breaking of the blind for any reason.

Note: The blinding rules and procedures described in the protocol do not apply to the unblinded repeat cohort using a different dosage formulation; see Appendix 5.

### 6.2.1 Clinical Research Staff

All observers who evaluate any reported AE, laboratory abnormalities, ECGs, and changes in the ECGs will be blinded as to what treatment sequence each subject is assigned.

## 6.2.2 Study Subjects

All subjects will be blinded as to which treatment they are receiving at any dose.

## 6.2.3 Bioanalytical Laboratory

All samples will be sent to the bioanalytical laboratory for analysis. The bioanalytical laboratory will be unblinded and only run the analysis on active treatment subjects.

### 6.2.4 Pharmacokinetic Analysis

Pharmacokinetic analysis will be completed only on the active treatment subjects and will be blinded by subject for interim assessments.

#### 6.2.5 Cardiac Vendor

Electrocardiogram data will be analyzed in a blinded fashion and then unblinded by the cardiac vendor in order to be presented by treatment group in aggregate (reviewers will remain blinded by subject).

#### 6.2.6 Unblinding Procedures

Unblinding of cohort data will occur after completion of the final subject study visit and follow-up telephone call for the cohort.

The treatment assignment should be unblinded at the clinic only in the case of an emergency, when knowledge of the study drug assignment is absolutely necessary for the clinical management or welfare of the subject. Breaking of the blind at the clinic under any other circumstances will be considered a protocol violation.

The Investigator is strongly encouraged to contact the Sponsor before unblinding the study drug assignment prior to the scheduled assessment of tolerance and safety data. If the blind is broken for any reason, the Investigator must notify the Sponsor within 1 day, and an SAE form must be completed, if appropriate. In addition, the Investigator will record the date and reason for revealing the blinded study drug assignment for that subject in the source documents and appropriate CRF page(s).

#### 6.3 Check-In Procedures

Subjects will check into the clinic on Day -2 for Part 1 and Day -1 for Part 2.

At check-in, all subjects will be evaluated to confirm they continue to meet all the inclusion criteria (Section 5.1) and none of the exclusion criteria (Section 5.2).

Subjects will undergo the following assessments during the confinement period prior to dosing:

- Physical and neurological examinations
- Weight
- Vital signs (temperature, respirations, blood pressure, pulse, and pulse oximetry)
- Triplicate 12-lead ECG
- Clinical laboratory tests
- Urine drug, alcohol, and cotinine screens results must be negative for the subject to continue study participation
- Serum pregnancy test (all female subjects) results must be negative for the subject to continue study participation
- Concomitant medication review
- AE review
- Cardiac telemetry (Part 1 only)

#### 6.4 Confinement

<u>Part 1 fasting cohorts, and Part 2, Cohort 8, Arm 4 only:</u> Subjects will be admitted to the research center on Day -2 (Part 1) or Day -1 (Part 2) and remain confined until after completion of the 48-hour procedures on Day 3. Subjects will return for a follow-up visit approximately 72 hours after dosing (Day 4) and receive a follow up phone call on Day 11 (+1 day).

Part 1 food-effect cohort, Part 2, Cohort 8, Arms 1-3 and Cohort 9: Subjects will be admitted to the research center on Day -2 of Period 1 and Period 2 (Part 1) or Day -1 (Part 2) and remain confined until after completion of the 48-hour procedures on Day 3 of each study period. Subjects will return for a follow-up visit approximately 72 hours after dosing (Day 4) in each study period. Subjects will receive a follow up phone call on Day 11 (+1 day) of Period 2.

Please note that Cohort 9 is the same 6 subjects that were in Cohort 8, Arm 4 (IR tablet formulation) under fed conditions. In Cohort 8, Arm 4, subjects fasted.

### 6.5 Fasting/Meals/Beverages

## 6.5.1 Fasting/Meals<sup>3</sup>

Part 1 fasted cohorts and Part 2, Cohort 8, Arm 4 only Optional meals (lunch, snack, and dinner) may be served the day of check-in. All subjects will then be required to fast for at least 10 hours before dosing. The subjects will fast for 4 hours after dosing. Standard meals will be provided at appropriate times after dosing.

<u>Part 1 food-effect cohort, Part 2, Cohort 8, Arms 1-3 and Cohort 9</u>: Optional meals (lunch, snack, and dinner) may be served the day of check-in.

In the fasting study period, all subjects will be required to fast overnight for at least 10 hours before dosing.

In the fed study period of Part 1 and Part 2 (Cohort 8, Arms 1-3 and Cohort 9) subjects will be required to fast for at least 10 hours overnight before consuming a required FDA standard high-fat, high-calorie breakfast. Subjects will receive the required FDA standard high-fat, high-calorie breakfast to begin 30 minutes prior to scheduled administration of the dose and to end (last bite taken) within 5 minutes prior to dosing. The subjects will fast for 4 hours thereafter. The following high-fat (approximately 50% of total caloric content of the meal), high-calorie (approximately 1000 calories) breakfast will be ingested 30 minutes prior to administration of the drug:

- 2 eggs fried in butter
- 2 strips of bacon
- 2 slices of toast with butter
- 4 ounces of hash brown potatoes
- 8 ounces of whole milk

This meal contains approximately 150 protein calories, 250 carbohydrate calories, and 500-600 fat calories. An equivalent meal may be substituted with documentation of the menu and caloric contents with Sponsor approval prior to administration of the meal.

Subjects will fast for 4 hours after dosing. Standard meals will be provided at appropriate times after dosing.

Please note that Part 2, Cohort 9 is the same 6 subjects that were in Cohort 8 Arm 4 (IR tablet formulation) under fed conditions. In Cohort 8 Arm 4, subjects fasted.

#### 6.5.2 Beverages

Each dose of TBI-223 oral suspension and placebo for TBI-223 oral suspension will be administered orally followed by approximately 200 mL of room temperature water.

Except for the room temperature water provided with the study treatment, no water may be consumed for 1 hour prior to each dose through 1 hour after each dose.

At other times, subjects will be encouraged to drink water ad libitum.

## 6.6 Drug Administration

### 6.6.1 Administration of oral care strips

Listerine® oral care strips (or similar product) will be used to blind subjects to treatment (TBI-223 Oral Suspension or placebo for TBI-223 oral suspension). One strip will be added to the subject's tongue immediately before administration of the study treatment. Another strip will be placed on the subject's tongue immediately after the subject has swallowed the study treatment and 200 mL of water. Research staff will place the strip on the midsection of the subject's tongue. The subject should keep the strip on the

tongue while it dissolves but may swallow when they feel the need to. A mouth check will be performed, using a flashlight and tongue depressor, after each administration of Listerine oral care strip to ensure that all of the film has been dissolved.

6.6.2 Administration of TBI-223 Oral Suspension or Placebo for TBI-223 Oral Suspension Note: Detailed instructions for preparing and dispensing TBI-223 will be provided in a separate pharmacy manual. Any instructions in the pharmacy manual shall supersede those presented in this protocol.

TBI-223 Oral Suspension or placebo for TBI-223 oral suspension will be transferred and stored in Pyrex glass reagent bottles with a polypropylene (PP) screw cap without a liner. These bottles will be used for mixing, sampling, and storage prior to administration.

The required doses of the drug product will be dispensed using commercially available oral syringes of suitable capacity. The suspension will be dispensed just prior to dosing and not stored in the oral syringes.

Each dose of TBI-223 will be administered orally followed by approximately 200 mL of room temperature water. A mouth check will be performed immediately after dose to ensure that the medication has been appropriately swallowed.

Subjects will remain seated, except as otherwise required for study procedures or personal needs, for the first 4 hours after dosing. Should the need to move about occur during the first 4 hours after dosing on these days, subjects may be escorted to such procedures or activities by research personnel as deemed medically necessary. Subjects will not be allowed to lie down, except as directed by clinical staff secondary to AEs, for the first 4 hours after dosing.

6.6.3 Administration of TBI-223 Sustained Release and Immediate Release Tablets
For Part 2, Cohort 8 and Cohort 9, each subject will receive the oral dose of the
assigned study treatment (TBI-223 SR tablet formulations [Prototypes 1, 2, or 3] or
TBI-223 IR tablet formulation) with approximately 240 mL (8 fl. oz.) of room
temperature water. Subjects must swallow the study medication intact. The medication
should NOT be crushed or chewed. A hand and mouth check will be performed
immediately after dose to ensure that the medication has been appropriately swallowed.

The subjects will remain seated, except as otherwise required for study procedures or personal needs, for the first 4 hours after dosing. Should the need to move about occur during the first 4 hours after each dose, subjects may be escorted to such procedures or activities by research personnel as deemed medically necessary. Subjects will not be allowed to lie down, except as directed by clinical staff secondary to AEs, for the first 4 hours after dosing.

# 6.7 Blood Sampling, Processing and Shipment

Blood samples will be collected as detailed in Appendix 1.

Refer to the Schedule of Events for specific blood collection time points. The Principal Investigator, in conjunction with the Sponsor, may collect additional blood if necessary for repeat laboratory or safety evaluations including AE follow-up.

## 6.7.1 Part 1 fasting cohorts, and Part 2, Cohort 8, Arm 4 only

A total of 80 mL (20 x 4 mL samples) will be collected for pharmacokinetic analysis from each subject. Approximately 51.5 mL of blood will be collected for the clinical laboratory evaluations and coagulation testing. The total volume of blood collected from each subject will not exceed approximately 131.5 mL.

**Table 4** Total Volume of Blood to be Collected for Testing: Fasting Cohorts

| Reason for Collection | Number of<br>Samples | Volume per<br>Sample (mL) | Total Volume (mL) |
|---|---|---|---|
| Clinical labs at screening | 1 | 12.5 | 12.5 |
| Clinical labs during study (check-in, 24 and 72 hours/end-of-study) | 3 | 8.5 | 25.5 |
| Coagulation | 5 | 2.7 | 13.5 |
| Pharmacokinetic analysis | 20 | 4.0 | 80.0 |
| | | Total | 131.5 |

### 6.7.2 Part 1 food-effect cohort, Part 2, Cohort 8, Arms 1-3 only, and Cohort 9

A total of 160 mL (40 x 4 mL samples) will be collected for pharmacokinetic analysis from each subject. Approximately 90.5 mL of blood will be collected for the clinical laboratory evaluations and coagulation testing. The total volume of blood collected from each subject will not exceed approximately 250.5 mL.

Please note that Part 2, Cohort 9 is the same 6 subjects that were in Cohort 8 Arm 4 (IR tablet formulation) under fed conditions. In Cohort 8 Arm 4, subjects fasted.

Table 5 Total Volume of Blood to be Collected for Testing: Food-effect Cohorts

| Reason for Collection | Number of<br>Samples | Volume per<br>Sample (mL) | Total Volume (mL) |
|---|---|---|---|
| Clinical labs at screening | 1 | 12.5 | 12.5 |
| Clinical labs during study (check-in, 24 and 72 hours/end-of-study) | 6 | 8.5 | 51.0 |
| Coagulation | 10 | 2.7 | 27.0 |
| Pharmacokinetic analysis | 40 (20 in each study period) | 4.0 | 160.0 |
| | 1 | Total | 250.5 |

# 6.7.3 Pharmacokinetic Sampling Time Windows

Blood samples collected within the time windows listed below will not be considered deviations. Note: For the food-effect cohort, time windows are relative to dosing in each study period.

Table 6 Acceptable Pharmacokinetic Sampling Time Windows

| | Allowable Time Window | | |
|---|---|---|---|
| Investigation and examination | Postdose* | | |
| CAUMMUTON | ≤24 hours | >24 hours to ≤48 hours | >48 hours |
| Plasma sample collection for pharmacokinetic assessment | ± 2 minutes | ± 5 minutes | ± 10 minutes |

For the food-effect cohort, time windows are relative to dosing in each study period.

# **6.8** End-of-Study Procedures

On the day of study discharge (Day 4), the following procedures will be conducted:

- Physical and neurological examinations
- Vital signs measurements (blood pressure, pulse, temperature, respirations, and pulse oximetry)
- Blood collection for hematology, chemistry, coagulation
- Urine collection for urinalysis
- Concomitant medication review
- AE assessment

Subjects will receive a follow up phone call (Day 11 [+1 day].

For the food-effect cohort, the timing of these assessments is relative to study period 2.

# **6.9** Safety Monitoring and Procedures

#### 6.9.1 Adverse Events

Subjects will be instructed to inform the study physician and/or research personnel of any AEs that occur at any time during the study. Subjects will be monitored for AEs from the first dose through the end-of-study visit.

Refer to Section 7 for details regarding AE reporting.

## 6.9.2 Clinical Laboratory Evaluations

Clinical laboratory evaluations will be performed at the times noted on the appropriate events schedule (Table 9), A Clinical Laboratory Improvement Amendments (CLIA) certified laboratory will perform all clinical laboratory tests for this study. If exclusionary lab criteria are met, values may be confirmed by repeat evaluation.

- Hematology: hemoglobin, hematocrit, total and differential leukocyte count, red blood cell count (RBC), and platelet count.
- Serum Chemistry: albumin, blood urea nitrogen (BUN), creatinine, total bilirubin, alkaline phosphatase (ALP), aspartate transaminase (AST), alanine transaminase (ALT), sodium (Na+), potassium (K+), chloride (Cl-), lactate dehydrogenase (LDH), calcium (Ca), uric acid, glucose, gamma-glutamyltransferase (GGT), and magnesium.
- Serology: hepatitis B surface antigen, hepatitis C antibody, and HIV.
- Coagulation: prothrombin time (PT), partial thromboplastin time (PTT), and international normalized ratio (INR).
- Urinalysis The following will be evaluated by an automated or manual urine "dipstick" method: pH, specific gravity, protein, glucose, ketones, bilirubin, blood, nitrite, leukocyte esterase, and urobilinogen. If protein, occult blood, nitrite, or leukocyte esterase values are out of range, a microscopic examination will be performed.
- Urine Drug, Cotinine, and Alcohol Screens: drugs of abuse (amphetamines, benzodiazepines, barbiturates, cannabinoids, cocaine, opiates), alcohol, and cotinine.
- Pregnancy test (all female subjects).
- Follicle-stimulating hormone (female subjects claiming post-menopausal status).

# 6.9.3 Vital Signs

Vital signs (blood pressure, pulse rate, and respiration rate, pulse oximetry, and temperature) will be measured performed at the times noted on the appropriate events schedule (Table 9).

NOTE: Blood pressure and pulse rate will be noted and collected at the same time.

For purposes of qualifying any given subject for study participation, out-of-range vital signs may be repeated once.

Predose vital signs will be assessed by the Principal Investigator or designee (e.g., a medically qualified Sub-Investigator) prior to each study drug administration. The Principal Investigator or designee will verify the eligibility of each subject with out-of-range vital signs and document approval prior to dosing.

Additional vital signs measurements may be performed as deemed medically necessary by research personnel.

Blood pressure and heart rate should be measured after subjects are in a seated position for at least 2 minutes and then again after standing for at least 1 minute, except when they are supine or semi-reclined because of study procedures and/or AEs, or as deemed necessary by the Investigator.

# 6.9.4 Physical Examinations

Physical examinations, including height and weight measurements, will be conducted at the times noted on the appropriate events schedule (Table 9).

## 6.9.5 Neurological Examinations

Detailed neurological examinations will be conducted at the times noted on the appropriate events schedule (Table 9) and at unscheduled time points as deemed necessary by the Investigator. Each neurological exam will assess the following:

- Mental Status orientation, speech, and memory
- Cranial Nerves excluding fundoscopic examination
- Muscle tone and strength
- Sensory System brief survey for light touch and temperature of the face, neck, arms, trunk, and legs
- Reflexes –deep tendon reflexes and plantar responses (Babinski sign)
- Coordination upper and lower extremities, including tremor
  - Gait tandem gait

# 6.9.6 12-Lead Electrocardiograms

Safety 12-lead ECGs will be recorded and printed for on-site review by the Principal Investigator or designee at the times noted on the appropriate events schedule (Table 9). The interpretation of these ECGs will be noted, but not the ECG intervals, unless as part of an AE (e.g. 1<sup>st</sup> degree AV block with PR interval of 240 msec).

All safety ECGs will be performed after the subject has been in supine position for a minimum of 5 minutes.

## 6.9.7 Cardiac Holter Monitoring, and Cardiodynamic Assessment

In order to detect potential changes in ECG parameters, study subjects will undergo cardiac Holter monitoring. Holter monitoring will begin approximately 24 hours before dosing and continue for at least 48 hours after dosing.

On Day -2 and Day -1, subjects should fast until lunch to avoid circadian fluctuations.

In addition, replicate ECGs will be obtained after dosing, specifically around the estimated  $T_{max}$  (which is estimated to be around 3 hours after dosing; although the timing may be altered based on generated phase 1 pharmacokinetic data). ECG data will be analyzed focusing in particular on changes of the QT segment although other ECG parameters will be analyzed, as specified in the Statistical Analysis Plan (SAP).

Continuous 12-lead ECGs (Holter) will be recorded for 24 hours prior to dose and for at least 48 hours post dose. The ECG waveforms will be stored for analysis as appropriate after the completion of the study. Replicate 12-lead ECGs will be extracted prior to dosing and serially after dosing by the central ECG laboratory at the time points shown in Table 9. At each time point for ECG extraction, subjects should be resting in the supine position for at least 10 minutes.

NOTE: When ECG extractions coincide with safety ECGs, vital signs assessment and blood draws, procedures should be carried out in said order.

Details regarding the equipment and methods to be used for continuous Holter extraction and analysis are provided in Appendix 4.

Part 2 of the study will not have cardiac Holter monitoring.

## 6.9.8 Other Safety Measures

Medical emergency personnel trained in advanced cardiac life support will be on site to monitor subjects during the confinement period in the research center. Emergency medical equipment including but not limited to intubation equipment and pulse oximetry shall be maintained on site to administer appropriate medical care should it be required.

Procedures will be completed as specified in this protocol unless contraindicated due to a reported AE.

#### 7 ADVERSE EVENTS

The Investigator or a suitably medically qualified designee are responsible for eliciting adverse events by observing and questioning the subject and recording all adverse events observed by him/her or reported by the subject during the trial.

#### 7.1 **Definitions**

#### 7.1.1 Adverse Event

Any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a trial treatment whether or not considered related to trial treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a trial treatment, whether or not related to the trial treatment.

#### 7.1.2 Serious Adverse Event

Any untoward medical occurrence that at any dose:

- Results in death;
- Is life threatening (any event in which the participant was at risk of death at the time of the event; it does not refer to an event, which hypothetically might have caused death if it were more severe);
- Requires inpatient hospitalization or prolongation of existing hospitalization; In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious. Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE;
- Results in persistent or significant disability/incapacity; the term disability means a substantial disruption of a person's ability to conduct normal life functions. This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza,
and accidental trauma (e.g., sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption;

- Is a congenital anomaly/birth defect; or
- Is a medically important event.

Note: Medical and scientific judgment should be exercised in deciding which is a medically important event that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the participant or may require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or the development of drug dependency or drug abuse. A "suspected transmission of infectious agent by a medicinal product" is also considered a serious adverse event under the SAE criterion "Other medically important condition".

# 7.2 Attribution/Causality

An adverse reaction, the nature or severity of which is not consistent with the applicable product information (e.g., Investigator's Brochure for an unapproved investigational product).

- The investigator is obligated to assess the relationship between trial treatment and each occurrence of each AE/SAE.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to trial treatment administration will be considered and investigated.
- The investigator will also consult the Investigator's Brochure and/or Product Information, for marketed products, in his/her assessment.
- For each AE/SAE, the investigator must document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred, and the investigator has
  minimal information to include in the initial report to the Sponsor/designee.
  However, it is very important that the investigator always make an assessment of
  causality for every event before the initial transmission of the SAE data to the
  Sponsor/designee.
- The investigator may change his/her opinion of causality in light of follow-up information and send a SAE follow-up report with the updated causality assessment.

 Table 7
 Adverse Event Attribution/Causality Ratings

| Relatedness Rating | Definition |
|---|---|
| Not Related | An adverse event, which is not related to the use of the drug. |
| Unlikely | An adverse event for which an alternative explanation is more likely, e.g., concomitant drug(s) or concomitant disease(s), and/or the relationship in time suggests that a causal relationship is unlikely. |
| Possible | An adverse event, which might be due to the use of the drug. An alternative explanation, e.g., concomitant drug(s) or concomitant disease(s), is inconclusive. The relationship in time is reasonable; therefore, the causal relationship cannot be excluded. |
| Probable | An adverse event, which might be due to the use of the drug. The relationship in time is suggestive, e.g., confirmed by dechallenge. An alternative explanation is less likely, e.g., concomitant drug(s) or concomitant disease(s). |
| Certain | An adverse event, which is listed as a possible adverse reaction and cannot be reasonably explained by an alternative explanation, e.g., concomitant drug(s) or concomitant disease(s). |

**Table 8** Definitions for Adverse Event Severity Gradings

| Grade | Severity Rating | Definition |
|---|---|---|
| GRADE 1 | Mild | Transient or mild discomfort (< 48 hours); no medical intervention/therapy required. |
| GRADE 2 | Moderate | Mild to moderate limitation in activity - some assistance may be needed; no or minimal medical intervention/therapy required. |
| GRADE 3 | Severe | Marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible. |
| GRADE 4 | Potentially Life-<br>Threatening | Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable. |

See Appendix 3 for full DMID Toxicity Tables. The above ratings should be used to estimate the grade for abnormalities NOT found elsewhere in the Toxicity Tables. Lab results within the testing facility's normal range will not be considered AEs when referenced to the DMID assessment/grading scale (Appendix 3).

Laboratory abnormalities and cardiovascular findings of hypertension or hypotension Grade 2 or above on the DMID toxicity tables will be considered AEs.

# 7.3 Reporting

#### 7.3.1 Adverse Event

Adverse Events will be collected by the Investigator or qualified designee(s) from the time a subject signs the Informed Consent Form through the follow-up phone calls (Day 11+1 day). Any AE (serious or non-serious) observed by the Investigator (or a suitably medically qualified designee) or reported by the subject will be recorded on the Adverse Event Case Report Form. The Investigator will review each AE and assess its relationship to drug treatment based on all available information at the time of the completion of the CRF. The following information will be recorded for each Adverse Event reported:

- Diagnosis of the AE, if possible. In the case where an overall diagnosis cannot be made, each specific sign and/or symptom will be recorded as individual AEs;
- Date of onset;
- Stop date (with duration, if applicable);
- Severity;
- Action taken with IMP;
- Other action taken;
- Outcome:
- Relationship to IMP;
- Occurrence:
- Seriousness

### 7.4 Serious Adverse Event Reporting

The Investigator or designee will notify the appropriate Sponsor contact immediately after the SAE detection, observation, or report of occurrence (regardless of the relationship to test article). The Sponsor contact information for SAE reporting is provided below:

PPD PVG (pharmacovigilance service provider for TB Alliance)

Email: rtpsafety@ppdi.com Safety Hotline: +1 888 483 7729 Safety Fax Number +1 888 529 3580

And

Paul Bruinenberg MD, MBA Global Alliance for TB Drug Development 40 Wall Street, 24th Floor New York, NY 10005, United States of America Telephone: +1 646.616.8629 Mobile: +1 201.312.0988 Facsimile: +1 212.227.7541

Email: Paul.Bruinenberg@tballiance.org

These SAE reports must contain the following information:

- A. Study name/number (for EU also the EudraCT number)
- B. Study drug
- C. Investigator details (name, phone, fax, e-mail)
- D. Subject number
- E. Subject demographics
- F. Clinical event:
  - 1) Description
  - 2) Date of onset
  - 3) Treatment (drug, dose, dosage form)
  - 4) Adverse event relationship to study drug
  - 5) Action taken regarding study drug in direct relationship to the AE
- G. If the AE was fatal or life-threatening
- H. If applicable, cause of death (whether or not the death was related to study drug)
- I. If applicable, autopsy findings (if available)

Any new SAE that occurs within one month after the study period and is considered to be possibly related to the Investigational Product (IP) should be recorded and reported immediately to the Sponsor.

The person responsible for the study shall take care that the study has been carried out in accordance with pharmacovigilance local regulations.

All serious event reporting will adhere to U.S. Code of Federal Regulations (21 CFR Part 312.32) for IND drugs and 21 CFR 314.80 for marketed drugs (15-day alerts). The Institutional Review Board (IRB) will be notified of the alert reports per Food and Drug Administration (FDA) regulations.

All AEs, including SAEs, will be followed to resolution when possible. All AEs and treatment administered will be recorded on the case report form (CRF).

The Sponsor will be responsible for processing and reporting any SAEs (and their relevant updates) to the FDA or other applicable regulatory agency.

### 7.5 Follow up of Adverse Events

All AEs will be followed until:

- Satisfactory clinical resolution or stabilization; or
- End of the follow-up period; and
- All gueries on these AEs have been resolved.

Certain long-term AEs cannot be followed until resolution within the setting of this protocol. In these cases, follow-up will be the responsibility of the treating physician. However, this will have to be agreed upon with the Sponsor Medical Monitor.

The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by Sponsor or representative to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals. Investigator should contact Sponsor/designee to discuss appropriate medical follow-up if consultation required.

If a participant dies during participation in the trial or during a recognized follow-up period, the investigator will provide Sponsor/representative with a copy of any post-mortem findings including histopathology.

New or updated information on an SAE will be recorded in the originally completed CRF and submitted to Sponsor within 24 hours of the information becoming known per SAE reporting guidelines.

### 7.6 Post-Trial Serious Adverse Events

Any new SAEs reported by the subject to the Investigator that occur up to 30 days after last contact and are determined by the Principal Investigator to be possible, probable or very likely related to the use of the IMP, will be reported to the Sponsor, IRB and FDA on an expedited basis as required in accordance with local requirements and ICH guidelines for GCP.

# 7.7 Clinical Laboratory Adverse Events

Changes in the results of the Clinical Laboratory assessment results which the Investigator feels are clinically significant will be reported as AEs. It is the Investigators' responsibility to review the results of all laboratory tests as they become available. This review must be documented by the Investigators' dated signature on the laboratory report. For each abnormal laboratory test result, the Investigator needs to ascertain and document if this is a clinically significant change from baseline for that individual participant. This determination, however, does not necessarily need to be made the first time an abnormal value is observed. The Investigator may repeat the laboratory test or request additional tests to verify the results of the original laboratory

tests. If this laboratory value is determined by the Investigator to be a clinically significant change from baseline for that participant, it is considered to be an AE.

# 7.8 **Drug Interaction**

If the Investigator becomes aware that the subject has experienced a drug interaction which has resulted in an adverse event, it will be recorded as an AE.

# 7.9 Pregnancy

The Investigator will immediately notify the Sponsor of any pregnancy that is discovered during the clinical trial. Pregnancy forms will be completed for all pregnancies reported during the study or in the 30 days after completion of the IMP. In addition, the Investigator will report to the Sponsor follow up information regarding the outcome of the pregnancy, including perinatal and neonatal outcome. Infants should be followed for 6 months.

If pregnancy is suspected while the subject is receiving IMP, the IMP will be withheld immediately until the result of the pregnancy test is known. If pregnancy is confirmed, the IMP will be permanently discontinued in an appropriate manner and the subject withdrawn from the trial. Protocol-required procedures for trial discontinuation and follow up will be performed unless contraindicated by the pregnancy.

If the Investigator becomes aware the female partner of a male subject becomes pregnant during the study or in the 30 days after the completion of IMP, consent will be requested from the female partner for collection of information on her pregnancy history and for information on the current pregnancy and birth.

### 7.10 Monitoring and Safety for Specific Toxicities

During preclinical testing, issues with increased heart rate and lowering of blood pressure were detected. Therefore, heart rate and blood pressure changes should be monitored carefully. When abnormalities are detected both blood pressure and pulse rate should be captured simultaneously

#### 8 GENERAL CONSIDERATIONS

### 8.1 Basic Principles

This research will be carried out in accordance with the protocol, the International Council for Harmonisation (ICH), Guideline for Good Clinical Practice: Consolidated Guidance (E6), and applicable regulatory requirements(s) including clinical research guidelines established by the Basic Principles defined in the U.S. 21 CFR Parts 50, 56, and 312 and the principles enunciated in the Declaration of Helsinki (revised version Fortaleza 2013).

### 8.2 Institutional Review Board

This protocol will be reviewed by an appropriate IRB and study enrollment will not commence until the Board has approved the protocol or a modification thereof. The Board is constituted and operates in accordance with the principles and requirements described in 21 CFR Part 56.

#### 8.3 Informed Consent

Written informed consent will be obtained from each subject prior to performing any baseline study-specific evaluations. The ICD is prepared by the Investigator or designee, subject to review and approval by the Sponsor, and forwarded to a qualified IRB for final review and approval. The IRB-approved document must contain, at minimum, the eight basic elements of informed consent. Only the most recently IRB-approved ICD must be used to consent prospective study subjects. One copy of the signed and dated ICD will be given to the subject and the original retained by the Investigator/site.

# 8.4 Indications for Subject Withdrawal

Subjects will be free to withdraw at any time for any reason, or they may be withdrawn if necessary, to protect their health and safety or the integrity of the study data.

The final report will include reasons for withdrawals. In the event of an early termination, subjects will undergo the procedures described in Section 6.8.

Subjects who experience emesis may be replaced if the emesis could potentially impact drug absorption and therefore the pharmacokinetic data. Cases of emesis will be evaluated by the Sponsor and Principal Investigator to determine if subject replacement is needed.

For Part 1, replacement subjects will be numbered 17XX where XX is 10 plus the original subject's last 2 assigned numbers (e.g. if subject 1702 needs to be replaced due to emesis, the replacement subject number would be 1712). Replacement subjects will receive the same dose allocation of study drug (active or placebo) and they will all be blinded aside from the pharmacist assigning the drug.

# 8.5 Termination of the Study

The Principal Investigator reserves the right to terminate the study in the interest of subject safety and welfare. The Sponsor reserves the right to terminate the study at any time for administrative reasons.

### 8.6 Documentation

All documents pertaining to the study, including a copy of the approved protocol, copy of the ICD and Health Insurance Portability and Accountability Act (HIPAA) documents, completed CRFs (where applicable), drug accountability and retention records, and other study related documents will be retained in the permanent archives of the study site. These will be available for inspection at any time by the Sponsor or the FDA. Per 21 CFR 312, record retention for this study is required for a period of two years following the date on which this study agent is approved by the FDA for the marketing purposes that were the subject of this investigation; or, if no application is to be filed or if the application is not approved for such indication, until two years following the date on which the entire study is completed, terminated, or discontinued, and the FDA is notified.

Subject records will be kept private except when ordered by law. The following individuals will have access to study subject records: Principal Investigator and designees, study Sponsor, monitors, and auditors, the FDA, other government offices, and the IRB.

### 8.7 Trial Monitoring

Sponsor personnel (or designees) will be responsible for monitoring the study to ensure compliance with the protocol and GCP. Compliance may be verified by one or more of the following methods: on-site visits, frequent communication with the Investigator, and/or review of CRFs and source documents. The Investigator agrees to permit such monitoring as well as audits or reviews by regulatory authorities and the IRB.

### 8.8 Reimbursement, Indemnity, and Insurance

Reimbursement, indemnity, and insurance shall be addressed in a separate agreement on terms agreed upon by the parties.

#### 9 PHARMACOKINETIC ANALYSIS

### 9.1 Analytical Methodology

Plasma samples will be analyzed for TBI-223 and M2 using validated assays. Plasma samples from subjects who receive placebo for TBI-223 oral suspension will not be analyzed.

### 9.2 Pharmacokinetic Analysis

Final pharmacokinetic calculations will be performed using appropriate software, e.g. Phoenix<sup>TM</sup> WinNonlin<sup>®</sup> (Version 8.1 or higher, Certara, L.P. in conjunction with the internet-accessible implementation of Pharsight<sup>®</sup> Knowledgebase Server<sup>TM</sup> [PKSO;

Version 4.0.4 or higher, Certara, L.P.]) and/or SAS® (Version 9.4 or higher, SAS Institute Inc.).

Pharmacokinetic parameters will be calculated using non-compartmental analysis. The following pharmacokinetic parameters will be determined as appropriate as detailed below.

| AUC <sub>Extrap</sub> (%) | The percentage of AUC <sub>inf</sub> based on extrapolation |
|---|---|
| | Area under the concentration-time curve from time-zero extrapolated to infinity; calculated as: $AUC_{inf} = AUC_{last} + \frac{C_{last}}{\lambda_z}$ |
| AUC <sub>last</sub> | Area under the concentration-time curve from time-zero to the time of the last quantifiable concentration; calculated using the linear trapezoidal rule |
| $C_{last}$ | The last quantifiable concentration determined directly from individual concentration-time data |
| CL/F | Apparent total clearance after single administration (TBI-223 only) |
| C <sub>max</sub> | Maximum concentration, determined directly from individual concentration-time data |
| T <sub>last</sub> | Time of the last quantifiable concentration |
| T <sub>max</sub> | Time of the maximum concentration |
| T <sub>1/2</sub> | The observed terminal half-life, calculated as: $T_{1/2} = \frac{\ln(2)}{\lambda_z}$ |
| Vz/F | Apparent volume of distribution in the terminal phase (TBI-223 only) |
| $\lambda_{\mathrm{z}}$ | The observed terminal rate constant; estimated by linear regression through at least 3 data points in the terminal phase of the log concentration-time profile |

Additional pharmacokinetic parameters may be calculated if deemed appropriate.

Pharmacokinetic parameters will be summarized by cohort using descriptive statistics. Dose proportionality will be assessed using the power model approach.

Food Effect: The effect of food will be assessed comparing pharmacokinetic parameters ( $C_{max}$ , AUCs) under fed versus fasting conditions using an analysis of variance (ANOVA) approach.

# 9.3 Statistical Analysis

Final statistical analyses will be performed using appropriate software, e.g. Phoenix<sup>™</sup> WinNonlin<sup>®</sup> (Version 8.1 or higher, Certara, L.P. in conjunction with the internet-accessible implementation of Pharsight<sup>®</sup> Knowledgebase Server<sup>™</sup> [PKSO; Version 4.0.4 or higher, Certara, L.P.]) and SAS<sup>®</sup> (Version 9.4 or higher, SAS Institute Inc.).

Pharmacokinetic parameters will be summarized by cohort using descriptive statistics. Summary statistics will also be presented by gender within each cohort. Dose proportionality for exposure parameters ( $C_{max}$ , AUCs) will be assessed using a power model approach.

Food-effect cohort: The effect of food will be assessed comparing pharmacokinetic parameters (C<sub>max</sub>, AUCs) under fed versus fasting conditions using an analysis of variance (ANOVA) approach.<sup>3</sup>

### 10 FACILITIES

### **CLINICAL TRIAL SITE**

Worldwide Clinical Trials Early Phase Services, LLC 2455 N.E. Loop 410, Suite 150 San Antonio, Texas 78217 Telephone: 210.635.1500

Fax: 210.635.1646

### CLINICAL LABORATORIES

Worldwide Clinical Trials Early Phase Services, LLC 2455 N.E. Loop 410, Suite 150 San Antonio, Texas 78217 Telephone: 210.635.1500

Fax: 210.635.1646

### ANALYTICAL LABORATORY

Alliance Pharma, Inc.

Project Manager: Michelle Black

Contact for Sample Shipment: Anna Cucinotta

17 Lee Boulevard Malvern, PA 19355 Phone: 610.296.3152 Fax: 610.296.3153

Email: samples@alliancepharmaco.com Web: www.alliancepharmaco.com

### **CARDIAC VENDOR**

iCardiac Technologies, Inc. 150 Allens Creek Road Rochester, New York 14618

Phone: 585.295.7610 Fax: 585.285.4130

### 11 DRUG SUPPLIES

Global Alliance for TB Drug Development will supply sufficient a quantity of the study drug, TBI-223 for preparation of TBI-223 oral suspension. Study drug will be shipped to Worldwide Clinical Trials Early Phase Services, LLC pursuant to site standard operating procedures. Upon receipt of the study drug, the study drug will be inventoried and stored in an environmentally controlled and secure, limited access area. The suspending vehicle and other supplies will be procured, inventoried, and stored appropriately by Worldwide Clinical Trials Early Phase Services, LLC pursuant to site standard operating procedures.

The lot numbers of the study drug, vehicle, and other supplies along with the expiration dates (where available) will be recorded and copies of the Certificate of Analysis (where available) will be maintained on file. Records will be maintained of the receipt and dispensation of the drugs supplied.

Samples will be collected from each batch of test product (TBI-223 Oral Suspension) and stored frozen until the clinical study report is issued. At the conclusion of the study, any unused study drug will be returned to the Sponsor or destroyed by the site pursuant to written authorization by the Sponsor and applicable federal and state regulations.

Global Alliance for TB Drug Development will supply sufficient quantity of the study drug, TBI-223 SR tablet formulations (Prototypes 1, 2, and 3) and TBI-223 IR tablet formulation for Part 2 of the study.

Study drug formulations will be shipped to Worldwide Clinical Trials Early Phase Services, LLC pursuant to site standard operating procedures. Upon receipt of the study drug products, the supplies will be inventoried and stored in an environmentally controlled and secure, limited access area. The lot numbers of the drugs along with the expiration dates (where available) will be recorded and copies of the Certificate of Analysis (where available) will be maintained on file. Records will be maintained of the receipt and dispensation of the drugs supplied. At the conclusion of the study, any unused study drug will be returned to the sponsor or destroyed by the site pursuant to written authorization by the sponsor and applicable federal and state regulations.

### 12 ADMINISTRATIVE ISSUES

The Investigator is referred to the Investigator Brochure, or information provided during the study initiation visit, information provided by the study monitor, and ICH Guidelines for Good Clinical Practice for information regarding the study drug, details, or general considerations to be followed during the course of this study.

# 13 EVENTS SCHEDULE

 Table 9
 Schedule of Assessments, Part 1

| Table 7 Sell | SCR | 011 | 1000 | 3311101 | 165, 1 | | | | | | CON | IFINI | EMI | ENT | | | | | | | | | 1 | FU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| STUDY DAY | -28 | -2 | -1 | | | | | | | DAY | | 12.11 | | 51 1 1 | | | | Т | DAY: | 2. | | 3 | 4 | 11 |
| 510212111 | to | CI | • | | | | | | | | - | | STU | DY I | HOUR | | | | | | | | | $(+1)^{a}$ |
| EVENT | -2 | | | 0 | 0.5 | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 12 | 16 <sup>b</sup> | 20 | 24 | 30 | 36 | 42 | 48 | 72 | N/A |
| Informed consent and medical history | X | | | | | | | | | | | | | | | | | | | | | | | |
| Height | X | X | | | | - | | | | | | | | | | | | | | | | | | |
| Weight Physical and neurological examinations <sup>c</sup> | X | X | | X | | | | | X | | | | | | X | | | X | | | | X | X | |
| Vital signs<br>(blood pressure,<br>pulse,<br>temperature,<br>respiration rate,<br>and pulse<br>oximetry) d | X | X | X | | X | X | X | X | X | X | | X | | X | X | X | X | X | X | X | X | X | X | |
| 12-lead safety<br>ECGs <sup>e</sup> | X | X | Xf | X | | X | | X | X | X | | X | | X | X | X | X | X | X | X | | X | | |
| HIV/hepatitis B, | X | | | | | | | | | | | | | | | | | | | | | | | |
| Clinical<br>laboratory tests<br>(hematology,<br>chemistry, and<br>urinalysis) | X | X | | | | | | | | | | | | | | | | X | | | | | X | |
| Coagulation tests | X | X | | | | | | | | | | | | | X | | | X | | | | | X | |

| | SCR | | | | | | | | | | CON | IFIN | EMI | ENT | | | | | | | | | | FU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| STUDY DAY | -28 | -2 | -1 | | | | | | | DAY | 1 | | | | | | | I | DAY | 2 | | 3 | 4 | 11 |
| | to | CI | | | STUDY HOUR | | | | | | | | | | | | | | (+1)a | | | | | |
| EVENT | -2 | | | 0 | 0.5 | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 12 | 16 <sup>b</sup> | 20 | 24 | 30 | 36 | 42 | 48 | 72 | N/A |
| Urine drug, | X | X | | | | | | | | | | | | | | | | | | | | | | |
| alcohol, cotinine | | | | | | | | | | | | | | | | | | | | | | | | |
| screen | | | | | | | | | | | | | | | | | | | | | | | | |
| Serum | X | X | | | | | | | | | | | | | | | | | | | | | | |
| pregnancy<br>(females only) | | | | | | | | | | | | | | | | | | | | | | | | |
| FSH (post- | X | | | | | | | | | | | | | | | | | | | | | | | |
| menopausal | | | | | | | | | | | | | | | | | | | | | | | | |
| females only) | | | | | | | | | | | | | | | | | | | | | | | | |
| Concomitant | X | | | | | | | | | | | | | | | | | | | | | | | |
| medication | | < | < | | | | | | | | | X | | | | | | | | | | | > | |
| review | | | | 1 | 1 | | | | | | | | | | | 1 | | | | | 1 | 1 | 1 | |
| Check-in | | X | | | | | | | | | | | | | | | | | | | | | | |
| questions | | | | | | | | | | | | | | | | | | | | | | | | |
| Adverse events <sup>g</sup> | X | X | | X | | X | | X | X | X | | X | | X | X | X | X | X | X | X | X | X | X | X |
| High-fat, high- | | | | X | | | | | | | | | | | | | | | | | | | | |
| calorie breakfast | | | | | | | | | | | | | | | | | | | | | | | | |
| (food-effect | | | | | | | | | | | | | | | | | | | | | | | | |
| cohort only)h | | | | 37 | | | | | | | | | | | | | | | | | | | | |
| Breath strip | | | | X | | | | | | | | | | | | | | | | | | | | |
| application <sup>i</sup> | | | | X | | | | | | | | | | | | | | | | | | | | |
| Dose <sup>j</sup> | | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| PK blood collection <sup>k</sup> | | | | X | X | X | X | X | X | X | X | X | Х | X | X | X | X | X | X | X | X | X | X | |
| Cardiac | | | | l. | | | | | | | | | | | | | | | | | | | | |
| telemetry | | | | | | | | | | | | | , | 5.7 | | | | | | | | | | |
| 12-lead Holter | | | < | | X> | | | | | | | | | | | | | | | | | | | |
| monitoring <sup>l</sup> | | | | | | | | | | | | | | | | | | | | | | | | |
| ECG extractions | | | X | X* | X | X | | X | X | X | X | X | | X | X | X | X | X | X | X | | X | | |
| from Holter | | | | | | | | | | | | | | | | | | | | | | | | |
| recording <sup>m</sup> | | | | | | | | | | | | | | | | | | | | | | | | |

CI = check-in; ECG = electrocardiogram; FSH = follicle-stimulating hormone; FU = follow up; HIV = human immunodeficiency virus; N/A = not applicable; PK = pharmacokinetic; SCR = screening; T and R = temperature and respirations

- a. For the food-effect cohort, the timing of the Day 11 (+1) follow up phone call will be relative to Period 2 dosing.
- b. The 16-hour time point following dosing on Day 1 will either be on Day 1 or Day 2, depending upon time of dosing on Day 1.
- c. A detailed neurological exam will be conducted by a licensed physician or suitably medically qualified designee at both scheduled and unscheduled time points as deemed necessary by the Investigator. The neurological examination is planned to be performed around the estimated T<sub>max</sub> (currently estimated at 3 hours post dosing; this time could change based on data generated during the study). Timepoints can be altered based on generated PK data
- d. Vitals signs will be measured at screening, check-in, and while subjects are in confinement. Vitals signs will be measured within 90 minutes prior to dosing and within 15 minutes of the remaining defined time points in flowchart. Both blood pressure and heart rate (pulse) should be captured simultaneously. Blood pressure and heart rate should be measured after subjects are in a seated position for at least 2 minutes and then again after standing for 1 minute, except when they are supine or semi-reclined because of study procedures and/or AEs, or as deemed necessary by the Investigator.
- e. 12-lead safety ECGs will be printed and reviewed on-site by the Principal Investigator or designee. Triplicate ECGs will be completed at screening, Day -2, Day -1, and at 48 hours only. All other time points will be single ECG readings within 15 minutes at time points within flowchart. The predose ECG should be performed prior to the pre-dose blood draw. If a subject experiences a post-dosing QTcF >500 msec or a change-from-baseline QTcF >60 msec, after repeat testing, additional ECGs should be recorded until normalization or return to baseline.
- f. The first ECG may be done within 2 hours prior to dosing and must be completed 20 minutes prior to the pre-dose blood draw. All safety ECGs on Day 1 and Day 2 will be extracted from a continuous 12 lead Holter recording at discrete timepoints as noted in above flow chart and Day -1 will be extracted at the same time as vital sign measurements.
- g. Subjects will be monitored for treatment-emergent AEs from the time of dosing and throughout the study via safety assessments, observation, and subject reporting. A specific inquiry regarding AEs will be conducted prior to dosing and at time points determined by the Investigator postdose and upon return to clinic for subsequent visits. The inquiry to collect AEs using non-leading questions on Day 11 (±1 day) will be done via a phone call.
- h. In the fed treatment period of the food-effect cohort, a high-fat, high-calorie breakfast meal will be given 30 minutes before treatment administration.
- i. A breath strip will be added to the subject's tongue before and after dose administration in order to blind the subject to treatment.
- j. TBI-223 oral suspension and placebo for TBI-223 oral suspension will be administered orally followed by approximately 200 mL of water.
- k. Samples collected for plasma pharmacokinetic analysis will be processed per the instructions in Appendix 1.
- 1. Cardiac telemetry will begin at least 24 hours before and end at least 48 hours after dosing.
- m. Replicate 12-lead ECGs will be extracted from a continuous Holter recording at discrete timepoints as noted on Day 1 in above flow chart for cardiodynamic assessment.
- \*Three timepoints before dosing: -45, -30, and -15 minutes.
- NOTE: When ECG extractions coincide with safety ECGs, vital signs assessments, and/or blood draws, then procedures should be carried out in said order.

### 14 REFERENCES

- 1. Prescription Monograph for Linezolid
- 2. FDA Guidance for Industry, Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers
- 3. FDA Food-Effect Guidance [https://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/ucm070241.pdf].

### APPENDIX 1 PHARMACOKINETIC SAMPLE PROCESSING

### A. Collection and Processing

A more detailed description of plasma sample preparation requirements may be provided by the analytical laboratory. If such a description is provided, the method of sample preparation provided by the laboratory shall supersede those provided in this protocol and appropriate documentation shall be placed in the Investigator Site File (ISF).

| | Processing Instructions |
|---|---|
| 1 | Samples will be collected via direct venipuncture at the time points delineated in the appropriate Events Schedule (Section 13). |
| 2 | Blood will be drawn into pre-chilled 4 mL evacuated tubes containing K <sub>3</sub> -EDTA and immediately placed on wet ice and then processed to plasma within 60 minutes. |
| 3 | Samples will be centrifuged at 1500 g at approximately 4°C (± 10 degrees) for 10 minutes. After centrifugation, two aliquots of plasma (the first containing at least 0.5 mL and the second containing the remainder of the plasma) will be removed and placed in appropriately labeled 5 mL polypropylene vials. |
| 4 | The aliquots will be immediately placed on dry ice. Within 90 minutes of collection, the aliquots will be stored in a freezer set at $-20^{\circ}\text{C} \pm 10^{\circ}\text{C}$ and remain in the freezer until transferred for analysis. |
| 5 | Samples will be transferred at the agreed upon intervals. |
| 6 | The aliquots will be transferred on dry ice to the Alliance Pharma, Inc. bioanalytical laboratory for the determination of plasma concentrations of TBI-223 and TBI-223 M2, using a validated procedure at Alliance Pharma. |
| 7 | Blood sampling, plasma processing, and storage time will be documented in the study records. |

# Labeling of aliquot tubes

Labels will contain at least the following information:

- a) Study number
- b)Subject number
- c) Period or dosing phase; sampling time (relative to dosing)
- d)Aliquot letter (A or B)

# **Shipment**

- 1. The samples will be transferred to the analytical laboratory after completion of the study or at mutually agreed upon time points during the clinical conduct of the study. The second set of samples will be shipped after the bioanalytical laboratory confirms receipt of the first set of samples.
- 2. Samples will be packaged into cryoboxes and sorted by subject and time point.
- 3. Prior to shipment, the samples will be appropriately packed in a cooler containing dry ice. Sufficient dry ice will be added to ensure that the samples will remain frozen for at least 72 hours.
- 4. An electronic manifest will be provided in advance. The shipment will be accompanied by documentation containing the following information: name of the study drug product, protocol number, number of subjects, and number of samples included in the shipment. Expected samples that are not present will be identified.
- 5. All frozen pharmacokinetic samples will be transferred with accompanying documentation to:

Alliance Pharma, Inc. 17 Lee Blvd Malvern, PA 19355 Telephone: 610.296.3152

Fax: 610.296.3153

Contact name: Anna Cucinotta

Contact e-mail: samplesa@alliancepharmaco.com

### APPENDIX 2 DESCRIPTION AND COMPOSITION OF TEST PRODUCT

### **Oral Suspension**

# **Description of the Dosage Form**

TBI-223 Oral Suspension is a compounded preparation at 25 mg/mL TBI-223 in Ora-Blend<sup>®</sup>. The suspension is compounded at the clinical study site with TBI-223 and Ora-Blend<sup>®</sup>, a commercially available flavored suspending vehicle.

Placebo for TBI-223 Oral Suspension is Ora-Blend<sup>®</sup>, a commercially available flavored suspending vehicle (without TBI-223). The placebo suspension, 100% Ora-Blend<sup>®</sup>, is purchased commercially by the clinical study site.

The required doses of the drug product are dispensed using commercially available oral syringes of suitable capacity.

# **Composition of the Drug Product**

The quantitative composition, function and quality of each ingredient in the drug product (TBI-223 Oral Suspension, 25 mg/mL) is described in the table below.

Qualitative and Quantitative Composition of the TBI-223 Oral Suspension, 25 mg/mL

| Ingredient | Function | Quality<br>Standard | Quantity per<br>Dose (50 mg) | Quantity<br>per Dose<br>(100 mg) | Quantity<br>per Dose<br>(300 mg) | Quantity<br>per Dose<br>(600 mg) | Quantity<br>per Dose<br>(1200 mg) | Quantity<br>per Dose<br>(1400 mg) |
|---|---|---|---|---|---|---|---|---|
| TBI-223 | Drug<br>Substance | In-house | 50 mg | 100 mg | 300 mg | 600 mg | 1200 mg | 1400 mg |
| Ora-Blend <sup>®1</sup> | Flavored<br>Oral<br>Suspending<br>Vehicle | Commercially available | q.s. to 2 mL | q.s to<br>4 mL | q.s to<br>12 mL | q.s. to<br>24 mL | q.s. to<br>48 mL | q.s to<br>56 mL |
| Total Volume | | | 2 mL | 4 mL | 12 mL | 24 mL | 48 mL | 56 mL |

<sup>&</sup>lt;sup>1</sup>Purified water, sucrose, glycerin, sorbitol, flavoring, microcrystalline cellulose, carboxymethylcellulose sodium, xanthan gum, carrageenan, calcium sulfate, trisodium phosphate, citric acid and sodium phosphate as buffers, dimethicone antifoam emulsion. Preserved with methylparaben and potassium sorbate.

### **Container and Closure System**

TBI-223 drug substance is shipped to the clinical study site in amber colored wide mouth glass bottles with a polypropylene screw cap without a liner.

TBI-223 Oral Suspension is transferred and stored in Pyrex glass reagent bottles with a polypropylene (PP) screw cap without a liner. These bottles are used for mixing, sampling and storage prior to administration.

### Enteric Capsules

# **Description of the Dosage Form**

TBI-223 Oral Enteric Capsules contain 150 mg TBI-223 in Vcaps<sup>®</sup> Enteric capsules. The capsules are filled at the clinical study site by manually filling TBI-223 into Vcaps<sup>®</sup> Enteric capsules which are commercially available empty capsule shells.

### **Composition of the Drug Product**

The quantitative composition, function and quality of each ingredient in the drug product (TBI-223 Oral Enteric Capsules, 150 mg) is provided in Table 10.

Table 10 Qualitative and Quantitative Composition of the TBI-223 Oral Enteric Capsules, 150 mg

| Ingredient | Function | Quality Standard | Quantity per 300 mg Dose |
|---|---|---|---|
| TBI-223 | Drug Substance | In-house | 300 mg |
| Vcaps® Enteric Capsules¹, Off-<br>white, Opaque, Size 00 | Capsule shell | Commercially available | 2 capsules |
| | Total Quantity | | 300 mg in 2 capsules |

<sup>&</sup>lt;sup>1</sup>Capsule shell composition: titanium dioxide 2% in Hypromellose-Hypromellose AS.

# **Container and Closure System**

TBI-223 Oral Enteric Capsules are stored in white HDPE bottles with PP CRC with a liner. These bottles are used for storage prior to administration.

#### **Tablets**

# **Description of the Dosage Form**

TBI-223 tablets are supplied as immediate release (IR) or sustained release (SR). The description of the tablets and strengths are presented in Table 11.

Table 11 Strength, Tablet Weight and Appearance of TBI-223 IR and SR Tablets

| Tablet Strength | Tablet Weight | Tablet Appearance |
|---|---|---|
| TB | I-223 Immediate Release (IR) Tal | olets |
| 600 mg | 750 mg | White to off-white, capsule shaped tablets, debossed with "TBA" on one side and "22" on the other |
| 1000 mg | 1250 mg | White to off-white, oval shaped tablets, debossed with "TBA" on one side and "23" on the other |
| TB | TBI-223 Sustained Release (SR) Tablets | |
| 600 mg (Prototype 1) | 1000 mg | White to off-white, capsule shaped tablets, debossed with "TBA" on one side and "11" on the other |
| 600 mg (Prototype 2) | 1000 mg | White to off-white, capsule shaped tablets, debossed with "TBA" on one side and "SR" on the other |
| 900 mg (Prototype 3) | 1200 mg | White to off-white, oval shaped tablets, debossed with "TBA" on one side and "900" on the other |

# **Composition of the Drug Product**

The composition of TBI-223 IR tablets, 600 mg and 1000 mg is presented in Table 12. The composition of TBI-223 SR Tablets, 600 mg (Prototype 1), 600 mg (Prototype 2) and 900 mg (prototype 3) is presented in Table 13, Table 14 and Table 15, respectively.

Table 12 Composition of TBI-223 IR Tablets, 600 mg and 1000 mg

| C | E | Percentage | 600 mg | 1000 mg | Reference to |
|---|---|---|---|---|---|
| Component | Function | (% w/w) | mg/t | mg/tablet | |
| | | I | ntragranular | | |
| TBI-223 a | Active | 80.00 | 600.00 | 1000.00 | In-House |
| Microcrystalline cellulose<br>(Avicel PH 302) <sup>b</sup> | Diluent | 10.00 | 75.00 | 125.00 | USP-NF,<br>Ph.Eur. |
| Hypromellose<br>(Methocel E5 Premium LV) | Binder | 3.00 | 22.50 | 37.50 | USP-NF,<br>Ph.Eur. |
| Crospovidone<br>(Kollidon CL) | Disintegrant | 3.00 | 22.50 | 37.50 | USP-NF,<br>Ph.Eur. |
| Purified water <sup>c</sup> | Granulating solvent | q.s | q.s | q.s | USP, Ph.Eur. |
| | | Е | xtragranular | | |
| Crospovidone<br>(Kollidon CL) | Disintegrant | 2.00 | 15.00 | 25.00 | USP-NF,<br>Ph.Eur. |
| Colloidal silicon dioxide<br>(Aerosil 200 Pharma) | Glidant | 1.00 | 7.50 | 12.50 | USP-NF,<br>Ph.Eur. |
| Magnesium stearate<br>(Ligamed MF-2-V) | Lubricant | 1.00 | 7.50 | 12.50 | USP-NF,<br>Ph.Eur. |
| Total unit dose | | 100.00 | 750.0 | 1250.0 | |

The molecular weight of TBI-223 is 365.4 g/mol. The actual quantity may be adjusted based on the assay value (anhydrous basis) and water content of the drug substance lot used.

Table 13 Composition of TBI-223 SR Tablets, 600 mg (Prototype 1)

| Component | Function | Percentage<br>(% w/w) | mg/tablet | Reference to<br>Standard |
|---|---|---|---|---|
| | | Intragi | ranular | _ |
| TBI-223 a | Active | 60.00 | 600.00 | In-House |
| Lactose monohydrate <sup>b</sup> (Pharmatose 200M) | Diluent | 9.90 | 99.00 | USP-NF, Ph.Eur. |
| Microcrystalline cellulose<br>(Avicel PH 200) | Diluent | 6.60 | 66.00 | USP-NF, Ph.Eur. |
| Hypromellose<br>(Methocel E5 Premium LV) | Binder | 5.00 | 50.00 | USP-NF, Ph.Eur. |
| Purified water <sup>c</sup> | Granulating solvent | q.s | q.s | USP, Ph.Eur. |

The quantity of microcrystalline cellulose may be adjusted to compensate for the actual amount of TBI-223 and to maintain a constant tablet weight.

<sup>&</sup>lt;sup>c</sup> Removed during processing.

| Component | Function | Percentage<br>(% w/w) | mg/tablet | Reference to<br>Standard |
|---|---|---|---|---|
| | | Intrag | ranular | |
| | | Extrag | ranular | - |
| Hypromellose (Methocel K100M Premium DC2) | Control Release<br>Polymer | 16.00 | 160.00 | USP-NF, Ph.Eur. |
| Colloidal silicon dioxide<br>(Aerosil 200 Pharma) | Glidant | 1.50 | 15.00 | USP-NF, Ph.Eur. |
| Magnesium stearate<br>(Ligamed MF-2-V) | Lubricant | 1.00 | 10.00 | USP-NF, Ph.Eur. |
| Total unit dose | | 100.00 | 1000.0 | |

The molecular weight of TBI-223 is 365.4 g/mol. The actual quantity may be adjusted based on the assay value (anhydrous basis) and water content of the drug substance lot used.

Table 14 Composition of TBI-223 SR Tablets, 600 mg (Prototype 2)

| Component | Function | Percentage<br>(% w/w) | mg/tablet | Reference to<br>Standard |
|---|---|---|---|---|
| | _ | Intragra | anular | |
| TBI-223 <sup>a</sup> | Active | 60.00 | 600.00 | In-House |
| Lactose monohydrate <sup>b</sup> (Pharmatose 200M) | Diluent | 12.90 | 129.00 | USP-NF, Ph.Eur. |
| Microcrystalline cellulose<br>(Avicel PH 200) | Diluent | 8.60 | 86.00 | USP-NF, Ph.Eur. |
| Hypromellose<br>(Methocel K4M Premium CR) | Control Release<br>Polymer | 5.00 | 50.00 | USP-NF, Ph.Eur. |
| Purified water <sup>c</sup> | Granulating solvent | q.s | q.s | USP, Ph.Eur. |
| | | Extragr | anular | |
| Hypromellose (Methocel K100<br>Premium LV) | Control Release<br>Polymer | 11.00 | 110.00 | USP-NF, Ph.Eur. |
| Colloidal silicon dioxide<br>(Aerosil 200 Pharma) | Glidant | 1.50 | 15.00 | USP-NF, Ph.Eur. |
| Magnesium stearate<br>(Ligamed MF-2-V) | Lubricant | 1.00 | 10.00 | USP-NF, Ph.Eur. |
| Total unit dose | | 100.00 | 1000.0 | |

The quantity of lactose monohydrate may be adjusted to compensate for the actual amount of TBI-223 and to maintain a constant tablet weight.

<sup>&</sup>lt;sup>c</sup> Removed during processing.

| Component | Function | Percentage<br>(% w/w) | mg/tablet | Reference to<br>Standard |
|---|---|---|---|---|
| | Intragranular | | | |

The molecular weight of TBI-223 is 365.4 g/mol. The actual quantity may be adjusted based on the assay value (anhydrous basis) and water content of the drug substance lot used.

Table 15 Composition of TBI-223 SR Tablets, 900 mg (Prototype 3)

| Component | Function | Percentage<br>(% w/w) | mg/tablet | Reference to<br>Standard |
|---|---|---|---|---|
| | | Intragi | ranular | |
| TBI-223 a | Active | 75.00 | 900.00 | In-House |
| Lactose monohydrate <sup>b</sup> (Pharmatose 200M) | Diluent | 3.90 | 46.80 | USP-NF, Ph.Eur. |
| Microcrystalline cellulose<br>(Avicel PH 200) | Diluent | 2.60 | 31.20 | USP-NF, Ph.Eur. |
| Hypromellose<br>(Methocel E5 Premium LV) | Binder | 5.00 | 60.00 | USP-NF, Ph.Eur. |
| Purified water <sup>c</sup> | Granulating solvent | q.s | q.s | USP. Ph.Eur. |
| | | Extrag | ranular | |
| Hypromellose (Methocel<br>K100M Premium DC2) | Control Release<br>Polymer | 11.00 | 132.00 | USP-NF, Ph.Eur. |
| Colloidal silicon dioxide<br>(Aerosil 200 Pharma) | Glidant | 1.50 | 18.00 | USP-NF, Ph.Eur. |
| Magnesium stearate<br>(Ligamed MF-2-V) | Lubricant | 1.00 | 12.00 | USP-NF, Ph.Eur. |
| Total unit dose | | 100.00 | 1200.0 | |

The molecular weight of TBI-223 is 365.4 g/mol. The actual quantity may be adjusted based on the assay value (anhydrous basis) and water content of the drug substance lot used.

### **Container and Closure System**

TBI-223 IR and SR Tablets are packaged as 30-count in 100 cc round high-density polyethylene (HDPE) bottles and closed with aluminum foil lined heat induction seals and 38 mm polypropylene (PP) child resistant closures (CRC).

The quantity of lactose monohydrate may be adjusted to compensate for the actual amount of TBI-223 and to maintain a constant tablet weight.

c Removed during processing.

The quantity of lactose monohydrate may be adjusted to compensate for the actual amount of TBI-223 and to maintain a constant tablet weight.

c Removed during processing.

# APPENDIX 3 DIVISION OF MICROBIOLOGY AND INFECTIOUS DISEASE TOXICITY TABLE

### Division of Microbiology and Infectious Disease (DMID) Toxicity Table

Source: U.S. National Institute of Allergy and Infectious Diseases, DMID, November 2007 (Draft)

### **ABBREVIATIONS**: Abbreviations utilized in the Table:

| ULN = Upper Limit of Normal | LLN = Lower Limit of Normal |
|----------------------------------|-----------------------------|
| $R_x$ = Therapy | Req = Required |
| Mod = Moderate | IV = Intravenous |
| ADL = Activities of Daily Living | Dec = Decreased |

### **ESTIMATING SEVERITY GRADE**

For abnormalities NOT found elsewhere in the Toxicity Tables use the scale below to estimate grade of severity:

| Grade | Severity Rating | Definition |
|---|---|---|
| GRADE 1 | Mild | Transient or mild discomfort (< 48 hours); no medical intervention/therapy required. |
| GRADE 2 | Moderate | Mild to moderate limitation in activity - some assistance may be needed; no or minimal medical intervention/therapy required. |
| GRADE 3 | Severe | Marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible. |
| GRADE 4 | Potentially Life-<br>threatening | Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable. |

### **SERIOUS OR LIFE-THREATENING AES**

ANY clinical event deemed by the clinician to be serious or life-threatening should be considered a grade 4 event. Clinical events considered to be serious or life-threatening include, but are not limited to: seizures, coma, tetany, diabetic ketoacidosis, disseminated intravascular coagulation, diffuse petechiae, paralysis, acute psychosis, severe depression.

### COMMENTS REGARDING THE USE OF THESE TABLES

- Standardized and commonly used toxicity tables (Division of AIDS, NCI's Common Toxicity Criteria (CTC), and World Health Organization (WHO)) have been adapted for use by the Division of Microbiology and Infectious Diseases (DMID) and modified to better meet the needs of Patients in DMID trials.
- For parameters not included in the following Toxicity Tables, sites should refer to the "Guide For Estimating Severity Grade" located above.

- Criteria are generally grouped by body system.
- Some protocols may have additional protocol specific grading criteria, which will supersede the use of these tables for specified criteria.

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin | 9.5 - 10.5 gm/dL | 8.0 - 9.4gm/dL | 6.5 - 7.9 gm/dL | < 6.5 gm/dL |
| Absolute Neutrophil<br>Count | 1000-1500/mm <sup>3</sup> | 750-999/mm <sup>3</sup> | 500-749/mm <sup>3</sup> | <500/mm <sup>3</sup> |
| Platelets | 75,000-99,999/mm <sup>3</sup> | 50,000-74,999/mm <sup>3</sup> | 20,000-49,999/mm <sup>3</sup> | <20,000/mm <sup>3</sup> |
| WBCs | 11,000-13,000/<br>mm <sup>3</sup> | 13,000-15,000<br>/mm <sup>3</sup> | 15,000-30,000/mm <sup>3</sup> | >30,000 or <1,000<br>/mm <sup>3</sup> |
| % Polymorphonuclear<br>Leucocytes + Band<br>Cells | > 80% | 90 – 95% | >95% | |
| Abnormal Fibrinogen | Low:<br>100-200 mg/dL<br>High:<br>400-600 mg/dL | Low:<br><100 mg/dL<br>High:<br>>600 mg/dL | Low:<br>< 50 mg/dL<br> | Fibrinogen associated with gross bleeding or with disseminated coagulation |
| Fibrin Split Product | 20-40 mcg/ml | 41-50 mcg/ml | 51-60 mcg/ml | > 60 mcg/ml |
| Prothrombin Time (PT) | 1.01 - 1.25 x ULN | 1.26-1.5 x ULN | 1.51 -3.0 x ULN | >3 x ULN |
| Activated Partial<br>Thromboplastin (APPT) | 1.01 -1.66 x ULN | 1.67 - 2.33 x ULN | 2.34 - 3 x ULN | > 3 x ULN |
| Methemoglobin | 5.0 - 9.9 % | 10.0 - 14.9 % | 15.0 - 19.9% | > 20.0 % |

| CHEMISTRIES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130-135 mEq/L | 123-129 mEq/L | 116-122 mEq/L | < 116 mEq/L or abnormal<br>sodium with mental status<br>changes or seizures |
| Hypernatremia | 146-150 mEq/L | 151-157 mEq/L | 158-165 mEq/L | > 165 mEq/L or abnormal<br>sodium <i>with</i> mental status<br>changes or seizures |
| Hypokalemia | 3.0 - 3.4 mEq/L | 2.5 - 2.9 mEq/L | 2.0 - 2.4 mEq/L or intensive replacement therapy or hospitalization required | < 2.0 mEq/L or abnormal potassium <i>with</i> paresis, ileus or life-threatening arrhythmia |

| CHEMISTRIES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyperkalemia | 5.6 - 6.0 mEq/L | 6.1 - 6.5 mEq/L | 6.6 - 7.0 mEq/l | > 7.0 mEq/L or abnormal<br>potassium with life-<br>threatening arrhythmia |
| Hypoglycemia | 55-64 mg/dL | 40-54 mg/dL | 30-39 mg/dL | <30 mg/dL or abnormal<br>glucose <i>with</i> mental status<br>changes or coma |
| Hyperglycemia<br>(non-fasting and no<br>prior diabetes) | 116 - 160 mg/dL | 161- 250 mg/dL | 251 - 500 mg/dL | > 500 mg/dL or abnormal glucose <i>with</i> ketoacidosis or seizures |
| Hypocalcemia<br>(corrected for<br>albumin) | 8.4 - 7.8 mg/dL | 7.7 - 7.0 mg/dL | 6.9 - 6.1 mg/dL | < 6.1 mg/dL or abnormal calcium with life threatening arrhythmia or tetany |
| Hypercalcemia<br>(correct for albumin) | 10.6 - 11.5 mg/dL | 11.6 - 12.5<br>mg/dL | 12.6 - 13.5 mg/dL | > 13.5 mg/dL or abnormal calcium with life threatening arrhythmia |
| Hypomagnesemia | 1.4 - 1.2 mEq/L | 1.1 - 0.9 mEq/L | 0.8 - 0.6 mEq/L | < 0.6 mEq/L or abnormal magnesium with life-<br>threatening arrhythmia |
| Hypophosphatemia | 2.0 - 2.4 mg/dL | 1.5 -1.9 mg/dL<br>or replacement<br>Rx required | 1.0 -1.4 mg/dL<br>intensive therapy or<br>hospitalization<br>required | < 1.0 mg/dL or abnormal<br>phosphate <i>with</i> life-<br>threatening arrhythmia |
| Hyperbilirubinemia (when accompanied by any increase in other liver function test) | 1.1 - <1.25 x ULN | 1.25 - <1.5 x<br>ULN | 1.5 – 1.75 x ULN | > 1.75 x ULN |
| Hyperbilirubinemia<br>(when other liver<br>function are in the<br>normal range) | 1.1 - <1.5 x ULN | 1.5 - <2.0 x ULN | 2.0 – 3.0 x ULN | > 3.0 x ULN |
| BUN | 1.25 - 2.5 x ULN | 2.6 - 5 x ULN | 5.1 - 10 x ULN | > 10 x ULN |
| Hyperuricemia (uric acid) | 7.5 – 10.0 mg/dL | 10.1 – 12.0<br>mg/dL | 12.1 – 15.0 mg/dL | >15.0 mg/dL |
| Creatinine | 1.1 - 1.5 x ULN | 1.6 - 3.0 x ULN | 3.1 - 6 x ULN | > 6 x ULN or dialysis required |

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| AST (SGOT) | 1.1 - <2.0 x ULN | 2.0 – <3.0 x ULN | 3.0 – 8.0 x ULN | > 8 x ULN |
| ALT (SGPT) | 1.1 - <2.0 x ULN | 2.0 – <3.0 x ULN | 3.0 – 8.0 x ULN | > 8 x ULN |

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| GGT | 1.1 - <2.0 x ULN | 2.0 – <3.0 x ULN | 3.0 – 8.0 x ULN | > 8 x ULN |
| Alkaline Phosphatase | 1.1 - <2.0 x ULN | 2.0 – <3.0 x ULN | 3.0 – 8.0 x ULN | > 8 x ULN |
| Amylase | 1.1 - 1.5 x ULN | 1.6 - 2.0 x ULN | 2.1 - 5.0 x ULN | > 5.1 x ULN |
| Lipase | 1.1 - 1.5 x ULN | 1.6 - 2.0 x ULN | 2.1 - 5.0 x ULN | > 5.1 x ULN |

| URINALYSIS | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Proteinuria | 1+ or 200 mg - 1<br>gm loss/day | 2-3+ or 1- 2 gm<br>loss/day | 4+ or 2-3.5 gm<br>loss/day | nephrotic syndrome<br>or > 3.5 gm<br>loss/day |
| Hematuria* | microscopic only<br><10 rbc/hpf | gross, no clots >10<br>rbc/hpf | gross, with or<br>without clots, OR<br>red blood cell casts | obstructive or required transfusion |

<sup>\*</sup>Assessment does not apply if a subject is on menses.

| CARDIOVASCULAR | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cardiac Rhythm | | asymptomatic,<br>transient signs, no<br>Rx required | recurrent/persistent;<br>symptomatic Rx<br>required | unstable<br>dysrythmia;<br>hospitalization and<br>treatment required |
| Hypertension | transient increase<br>> 20 mm/Hg; no<br>treatment <sup>1</sup> | recurrent, chronic<br>increase ><br>20mm/Hg.<br>/treatment required | acute treatment required; outpatient treatment or hospitalization possible | end organ damage<br>or hospitalization<br>required |
| Hypotension | transient orthostatic hypotension with heart rate increased by <20 beat/min or decreased by <10 mm Hg systolic BP, No treatment required <sup>1</sup> | symptoms due to<br>orthostatic<br>hypotension or BP<br>decreased by <20<br>mm Hg systolic;<br>correctable with oral<br>fluid treatment | requires IV fluids; no hospitalization required | mean arterial pressure <60mm/ Hg or end organ damage or shock; requires hospitalization and vasopressor treatment |

| CARDIOVASCULAR | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Pericarditis | minimal effusion | mild/moderate<br>asymptomatic<br>effusion, no<br>treatment | symptomatic<br>effusion; pain; EKG<br>changes | tamponade;<br>pericardiocentesis<br>or surgery required |
| Hemorrhage, Blood<br>Loss | microscopic/occult | mild, no transfusion | gross blood loss; 1-2<br>units transfused | massive blood<br>loss; > 3 units<br>transfused |

<sup>1)</sup> For protocol TBI-223-CL-001, defined as increase from baseline in predose vital signs.

| RESPIRATORY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cough | Transient - no<br>treatment | persistent cough;<br>treatment responsive | Paroxysmal cough;<br>uncontrolled with<br>treatment | |
| Bronchospasm,<br>Acute | transient; no<br>treatment; 70% -<br>80% FEV <sub>1</sub> of peak<br>flow | requires treatment;<br>normalizes with<br>bronchodilator; FEV <sub>1</sub><br>50% - 70% (of peak<br>flow) | no normalization with<br>bronchodilator;FEV <sub>1</sub><br>25% - 50% of peak<br>flow; or retractions<br>present | cyanosis: FEV <sub>1</sub> < 25% of peak flow or intubation necessary |
| Dyspnea | dyspnea on exertion | dyspnea with normal activity | dyspnea at rest | dyspnea requiring Oxygen therapy |

| GASTROINTESTINA | L | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Nausea | mild or transient;<br>maintains<br>reasonable intake | moderate discomfort; intake decreased significantly; some activity limited | no significant<br>intake; requires IV<br>fluids | hospitalization<br>required; |
| Vomiting | 1 episode in 24<br>hours | 2-5 episodes in 24 hours | >6 episodes in 24<br>hours or needing IV<br>fluids | physiologic<br>consequences<br>requiring<br>hospitalization or<br>requiring parenteral<br>nutrition |
| Constipation | requiring stool<br>softener or dietary<br>modification | requiring laxatives | obstipation<br>requiring manual<br>evacuation or<br>enema | obstruction or toxic megacolon |
| Diarrhea | mild or transient; 3-<br>4 loose stools/day<br>or mild diarrhea | moderate or<br>persistent; 5-7 loose<br>stools/day or | >7 loose stools/day<br>or bloody diarrhea;<br>or orthostatic | hypotensive shock<br>or physiologic<br>consequences |

| GASTROINTESTINAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| | last < 1 week | diarrhea lasting >1<br>week | hypotension or<br>electrolyte<br>imbalance or >2L<br>IV fluids required | requiring<br>hospitalization |
| Oral<br>Discomfort/Dysphagia | mild discomfort; no difficulty swallowing | some limits on eating/drinking | eating/talking very<br>limited; unable to<br>swallow solid foods | unable to drink<br>fluids; requires IV<br>fluids |

| NEUROLOGICAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Neuro-Cerebellar | slight<br>incoordination<br>dysdiadochokinesis | intention tremor,<br>dysmetria, slurred<br>speech; nystagmus | locomotor ataxia | incapacitated |
| Psychiatric | mild anxiety or<br>depression | moderate anxiety or<br>depression; therapy<br>required; change in<br>normal routine | severe mood<br>changes requiring<br>therapy; or suicidal<br>ideation; or<br>aggressive ideation | acute psychosis requiring hospitalization; or suicidal gesture/attempt or hallucinations |
| Muscle Strength | Subjective<br>weakness no<br>objective<br>symptoms/ signs | mild objective<br>signs/symptoms no<br>decrease in function | objective weakness function limited | paralysis |
| Paresthesia (burning, tingling, etc.) | mild discomfort; no treatment required | moderate<br>discomfort; non-<br>narcotic analgesia<br>required | severe discomfort;<br>or narcotic<br>analgesia required<br>with symptomatic<br>improvement | incapacitating; or<br>not responsive to<br>narcotic analgesia |
| Neuro-sensory | mild impairment in sensation (decreased sensation, e.g., vibratory, pinprick, hot/cold in great toes) in focal area or symmetrical distribution; or change in taste, smell, vision and/or hearing | moderate impairment (mod decreased sensation, e.g., vibratory, pinprick, hot/cold to ankles) and/or joint position or mild impairment that is not symmetrical | severe impairment (decreased or loss of sensation to knees or wrists) or loss of sensation of at least mod degree in multiple different body areas (i.e., upper and lower extremities) | sensory loss<br>involves limbs and<br>trunk; paralysis; or<br>seizures |

| MUSCULOSKELETAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Arthralgia (joint pain) | mild pain not<br>interfering with<br>function | moderate pain,<br>analgesics and/or<br>pain interfering with<br>function but not with<br>activities of daily<br>living | severe pain; pain<br>and/or analgesics<br>interfering with<br>activities of daily<br>living | disabling pain |
| Arthritis | mild pain with inflammation, erythema or joint swelling – but not interfering with function | moderate pain with inflammation, erythema or joint swelling – interfering with function, but not with activities of daily living | severe pain with inflammation, erythema or joint swelling –and interfering with activities of daily living | permanent and/or<br>disabling joint<br>destruction |
| Myalgia | myalgia with no limitation of activity | muscle tenderness (at other than injection site) or with moderate impairment of activity | severe muscle<br>tenderness with<br>marked impairment<br>of activity | frank<br>myonecrosis |

| SKIN | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Mucocutaneous | erythema; pruritus | diffuse, maculo<br>papular rash, dry<br>desquamation | vesiculation or moist desquamation or ulceration | exfoliative dermatitis, mucous membrane involvement or erythema, multiforme or suspected Stevens-Johnson or necrosis requiring surgery |
| Induration | < 15mm | 15-30 mm | >30mm | |
| Erythema | < 15mm | 15-30 mm | >30mm | |
| Edema | < 15mm | 15-30 mm | >30mm | |
| Rash at Injection<br>Site | < 15mm | 15-30 mm | >30mm | |
| Pruritus | slight itching at injection site | moderate itching at injection extremity | itching over entire body | |

| SYSTEMIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Allergic Reaction | pruritus without rash | localized urticaria | generalized urticaria;<br>angioedema | anaphylaxis |
| Headache | mild, no treatment required | transient, moderate;<br>treatment required | severe; responds to initial narcotic therapy | intractable; requires<br>repeated narcotic<br>therapy |
| Fever: oral | 37.7 - 38.5 C or<br>100.0 - 101.5 F | 38.6 - 39.5 C or<br>101.6 - 102.9 F | 39.6 - 40.5 C or 103<br>- 105 F | > 40 C or > 105 F |
| Fatigue | normal activity reduced < 48 hours | normal activity<br>decreased 25- 50%<br>> 48 hours | normal activity<br>decreased > 50%<br>can't work | unable to care for self |

### APPENDIX 4 HOLTER RECORDING AND ANALYSIS

Continuous 12-lead ECGs (Holters) will be recorded using the Mortara Surveyor system.

The continuous 12-lead digital ECG data will be stored and transmitted to iCardiac using the appropriate medium (e.g., file transfer protocol [FTP], disc, or flash drive). ECGs to be used in the analyses will be selected by pre-determined time points as defined in the Schedule of Assessments and Procedures, and will be read centrally by iCardiac Technologies, Inc.

The following principals will be followed in iCardiac's core laboratory:

- ECG analysts are blinded to the subject, visit and treatment allocation
- Baseline and on-treatment ECGs for a particular subject will be over-read on the same lead and will be analyzed by the same reader.
- The primary analysis lead is lead II. If lead II is not analyzable, then primary lead of analysis will be changed to another lead for the entire subject data set.

The following is a brief description of ECG analysis methods utilized by iCardiac' core laboratory.

### **TQT Plus ECG Extraction Technique**

Ten 14-second digital 12-lead ECG tracings will be extracted from the continuous Holter recordings using the "TQT Plus method", a computer-assisted and statistical process utilized by iCardiac Technologies. The method enables extraction of ECGs with the lowest HR variability and noise within the protocol-specified extraction time window (e.g., the HR and QT changes from beat-to-beat in the range of <10%). At each protocol-specified timepoint, 10 ECG replicates will be extracted from a 5-minute "ECG window" (typically, the last 5 minutes of the 15-minute period when the subject is maintained in a supine or semi-recumbent quiet position).

# **High-Precision QT Analysis**

High-precision QT analysis will be performed on all analyzable (non-artifact) beats in the 10 ECG replicates. Statistical quality control procedures are used to review and assess all beats and identify "high" and "low" confidence beats using several criteria, including:

- QT or QTc values exceeding or below certain thresholds (biologically unlikely).
- RR values exceeding or below certain thresholds (biologically unlikely).
- Rapid changes in QT, QTc or RR from beat to beat.

Measurements of all primary ECG parameters (QT, QTc, RR) in all recorded beats of all replicates that are deemed "high confidence" is performed using COMPAS software. All low confidence beats are reviewed manually and adjudicated using pass-fail criteria. The final QC assessment is performed by a cardiologist. The beats found acceptable by manual review are included in the analysis. The median QT, QTc, and RR value from each extracted replicate is

calculated, and then the mean of all available medians from a nominal timepoint is used as the subject's reportable value at that timepoint.

Categorical T-wave morphology analysis and the measurement of PR and QRS intervals will be performed manually in 3 of the 10 ECG replicates at each timepoint. Each fiducial point (onset of P-wave, onset of Q-wave, offset of S-wave, and offset of T-wave) is electronically marked.

# T-wave morphology categories (assessed manually)

| Category | Description |
|---|---|
| Normal T-wave | Any T-wave not meeting any criterion below |
| Flat T-waves | T amplitude < 1 mm (either positive or negative) including flat isoelectric line |
| Notched T-wave (+) | Presence of notch(es) of at least 0.05 mV amplitude on ascending or descending arm of the positive T-wave |
| Biphasic | T-wave that contains a second component with an opposite phase that is at least 0.1 mV deep (both positive and negative/positive and polyphasic T-waves included) |
| Normal T-wave (-) | T amplitude that is negative, without biphasic T-wave or notches |
| Notched T-wave (-) | Presence of notch(es) of at least 0.05 mV amplitude on descending or ascending arm of the negative T-wave |

In addition to the T-wave categorical analysis, the presence of abnormal U-waves is noted.

### APPENDIX 5 REPEAT COHORT USING DIFFERENT DOSAGE FORMULATION

Procedures and analyses as outlined in this protocol will be the same, with the following exceptions:

- The dose of TBI-223 will be delivered in enteric capsules.
- All subjects will receive active treatment.
- A minimum of 6 subjects is needed. Ideally, all 8 subjects who participated in the original cohort will participate in the re-dose cohort. If less than 6 subjects from the original cohort agree to participate, additional subjects will be screened as needed in order to dose a minimum of 6 subjects.
- Repeat subjects will be assigned a new subject number so as not to break the blinding of the original cohort.
- The repeat cohort will not be blinded (blinding is not necessary because all subjects will receive the same treatment).
- Cardiac telemetry and Holter recording will not be performed during the re-dose cohort.
- Subjects will check-in on Day -1 instead of Day -2. With the exception of cardiac telemetry and Holter monitoring, the procedures that were previously scheduled for Day -2 will be performed on Day -1. The Day -1 results will be used to qualify repeat subjects for study participation. If additional subjects are needed, they will undergo screening to qualify for the study.
- Neurological examinations will be performed at Screening, Day -1, and at 3 and 48 hours postdose.

### **APPENDIX 6 PART 2 OF THE STUDY**

Procedures and analyses as outlined in this protocol will be the same, with the following exceptions:

The dose of TBI-223 will be delivered as follows in Cohort 8:

- Arm 1 TBI-223 SR Tablets (Prototype 1) 1800 mg dose (3 x 600 mg tablets), under fed conditions
- Arm 2 TBI-223 SR Tablets (Prototype 2) 1800 mg dose (3 x 600 mg tablets), under fed conditions
- Arm 3 TBI-223 SR Tablets (Prototype 3) 1800 mg dose (2 x 900 mg tablets), under fed conditions
- Arm 4 TBI-223 IR Tablets 2000 mg dose (2 x 1000 mg tablets), under fasting conditions

In Cohort 9, the subjects from Cohort 8, Arm 4, who received the IR tablet formulation will be brought back following a 7-day washout and administered TBI-223 IR tablets, 2000 mg dose (2 x 1000 mg tablets), under fed conditions.

- A minimum of 6 subjects per treatment arm in Part 2.
- Part 2 will not be blinded (blinding is not necessary because all subjects will receive the same treatment).
- Cardiac telemetry and Holter recording will not be performed during Part 2. Subjects will check-in on Day -1 instead of Day -2. With the exception of cardiac telemetry and Holter monitoring, the procedures that were previously scheduled for Day -2 will be performed on Day -1. The Day -1 results will be used to qualify repeat subjects for study participation. If additional subjects are needed, they will undergo screening to qualify for the study.
- Neurological examinations will be performed at Screening, Day -1, and at 3 and 48 hours postdose.

Table 16 Schedule of Assessments, Part 2

| Table 10 Sch | SCR | 011155 | CONFINEMENT | | | | | | | | | | | | | 1 | FU | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| STUDY DAY | -28 | -1 | | | | | | | DAY | | | | | | | | I | DAY: | 2 | | 3 | 4 | 11 |
| | to | CI | | | | | | | | | S | TUI | DY E | IOUR | | | | | | | (+1) | | |
| EVENT | -2 | | 0 | 0.5 | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 12 | 16 <sup>a</sup> | 20 | 24 | 30 | 36 | 42 | 48 | 72 | N/A |
| Informed consent and medical history | X | | | | | | | | | | | | | | | | | | | | | | |
| Height | X | | | | | | | | | | | | | | | | | | | | | | |
| Weight | X | X | | | | | | | | | | | | | | | | | | | | | |
| Physical and<br>neurological<br>examinations <sup>b</sup> | X | X | X | | | | | X | | | | | | | | | X | | | | X | X | |
| Vital signs<br>(blood pressure,<br>pulse,<br>temperature,<br>respiration rate,<br>and pulse<br>oximetry) c | X | X | | X | X | X | X | X | X | | X | | X | X | X | X | X | X | X | X | X | X | |
| 12-lead safety<br>ECGs <sup>d</sup> | X | X | Xe | | X | | X | X | X | | X | | X | X | X | X | X | X | X | | X | | |
| HIV/hepatitis B, | X | | | | | | | | | | | | | | | | | | | | | | |
| Clinical<br>laboratory tests<br>(hematology,<br>chemistry, and<br>urinalysis) | X | X | | | | | | | | | | | | | | | X | | | | | X | |
| Coagulation tests | X | X | | | | | | | | | | | | X | | | X | | | | | X | |
| Urine drug,<br>alcohol, cotinine<br>screen | X | X | | | | | | | | | | | | | | | | | | | | | |

# Protocol TBI-223-CL-001 Final Version 3.0

| | SCR | | | | | | | | | CO | NFIN | EM | ENT | | | | | | | | | I | FU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| STUDY DAY | -28 | -1 | | | | | | | DAY | 1 | | | | | | | I | DAY: | 2 | | 3 | 4 | 11 |
| | to | CI | | | | | | | | | , | STU | DY E | IOUR | | | | | | | | | (+1) |
| EVENT | -2 | | 0 | 0.5 | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 12 | 16 <sup>a</sup> | 20 | 24 | 30 | 36 | 42 | 48 | 72 | N/A |
| Serum | X | X | | | | | | | | | | | | | | | | | | | | | |
| pregnancy<br>(females only) | | | | | | | | | | | | | | | | | | | | | | | |
| FSH (post-<br>menopausal | X | | | | | | | | | | | | | | | | | | | | | | |
| females only) | | | | | | | | | | | | | | | | | | | | | | | |
| Concomitant medication review | X | < | <> | | | | | | | | | | | | | | | | | | | | |
| Check-in questions | | X | | | | | | | | | | | | | | | | | | | | | |
| Adverse events <sup>f</sup> | X | X | X | | X | | X | X | X | | X | | X | X | X | X | X | X | X | X | X | X | X |
| High-fat, high-<br>calorie<br>breakfast <sup>g</sup> | | | X | | | | | | | | | | | | | | | | | | | | |
| Dose | | | X | | | | | | | | | | | | | | | | | | | | |
| PK blood collection <sup>h</sup> | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |

CI = check-in; ECG = electrocardiogram; FSH = follicle-stimulating hormone; FU = follow up; HIV = human immunodeficiency virus; N/A = not applicable; PK = pharmacokinetic; SCR = screening; T and R = temperature and respirations

- a. The 16-hour time point following dosing on Day 1 will either be on Day 1 or Day 2, depending upon time of dosing on Day 1.
- b. A detailed neurological exam will be conducted by a licensed physician or suitably medically qualified designee at both scheduled and unscheduled time points as deemed necessary by the Investigator. The neurological examination is planned to be performed around the estimated T<sub>max</sub> (currently estimated at 3 hours post dosing; this time could change based on data generated during the study). Timepoints can be altered based on generated PK data.
- c. Vitals signs will be measured at screening, check-in, and while subjects are in confinement. Vitals signs will be measured within 90 minutes prior to dosing and within 15 minutes of the remaining defined time points in flowchart. Both blood pressure and heart rate (pulse) should be captured simultaneously. Blood pressure and heart rate should be measured after subjects are in a seated position for at least 2 minutes and then again after standing for 1 minute, except when they are supine or semi-reclined because of study procedures and/or adverse events, or as deemed necessary by the Investigator.
- d. 12-lead safety ECGs will be printed and reviewed on-site by the Principal Investigator or designee. Triplicate ECGs will be completed at screening, Day -2, Day -1, and at 48 hours only. All other time points will be single ECG readings within 15 minutes at time points within flowchart. The predose ECG should be performed prior to the pre-dose blood draw. If a subject experiences a post-dosing QTcF >500 msec or a change-from-baseline QTcF >60 msec, after repeat testing, additional ECGs should be recorded until normalization or return to baseline.
- e. The first ECG may be done within 2 hours prior to dosing and must be completed 20 minutes prior to the pre-dose blood draw. All safety ECGs on Day 1 and Day 2 will be extracted from a continuous 12 lead Holter recording at discrete timepoints as noted in above flow chart and Day -1 will be extracted at the same time as vital sign measurements.
- f. Subjects will be monitored for treatment-emergent adverse events from the time of dosing and throughout the study via safety assessments, observation, and subject reporting. A specific inquiry regarding adverse events will be conducted prior to dosing and at time points determined by the Investigator postdose and upon return to clinic for subsequent visits. The inquiry to collect adverse events using non-leading questions on Day 11 (±1 day) will be done via a phone call.
- g. In Part 2, Cohort 8, Arms 1-3 and Cohort 9, a high-fat, high-calorie breakfast meal will be given 30 minutes before treatment administration.
- h. Samples collected for plasma pharmacokinetic analysis will be processed per the instructions in Appendix 1. \*Three timepoints before dosing: -45, -30, and -15 minutes.
- NOTE: When ECG extractions coincide with safety ECGs, vital signs assessments, and/or blood draws, then procedures should be carried out in said order.